# **PROTOCOL AS0008 AMENDMENT 2**

PARALLEL-GROUP, DOSE-RANGING STUDY TO EVALUATE THE EFFICACY AND SAFETY OF BIMEKIZUMAR IN SUBJECTS WITH ACTIVE AND

EudraCT Number: 2016-001102-42 IND Number: 128708

UCB BIOPHARMA SPRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

| Protocol/Amendment number | Date | Type of amendment |
|---------------------------|-------------|-------------------|
| Final Protocol | 29 Jul 2016 | Not applicable |
| Protocol Amendment 1 | 15 Mar 2017 | Nonsubstantial |
| Protocol Amendment 2 | 09 Mar 2018 | Substantial |

## **Confidential Material**

# Confidential

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


# STUDY CONTACT INFORMATION

# **Sponsor**

UCB BIOPHARMA SPRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

# **Sponsor Study Physician**

| nsor | | , | |
|----------------|-----------------|----------------------------|---|
| BIOPHARMA | SPRL | , com | * |
| de la Recherch | ne 60 | "He" | |
| Brussels | | *ions | |
| GIUM | | diate | |
| nsor Study | Physician | ions of valiations thereof | |
| Name: | , MD, MSc, PhD | -51 | |
| Address: | UCB Pharma Ltd. | and any exerc | |
| | 208 Bath Road | A <sup>o</sup> | |
| | Slough, SL1 3WE | 80 | |
| | UNITED KINGDOM | alle | |
| Phone: | | Ajio <sup>1</sup> | |

# **Clinical Project Manager**

| Name: | , PharmD, PhD |
|---|---|
| Address: | UCB BIOSCIENCES GmbH Alfred-Nobel-Str. 10 40789 Monheim am Rhein GERMANY |
| Phone: | |

# Clinical Trial Biostatistician

| Name: | , MS |
|----------|---------------------------|
| Address: | UCB BIOSCIENCES Inc. |
| 69 | 8010 Arco Corporate Drive |
| US | Raleigh, NC 27617 |
| 200 | UNITED STATES |
| Phone: | |


# **Clinical Monitoring Contract Research Organization**

| | Name: | PRA Health Sciences | ] |
|---|---|---|---|
| | Address: | 4130 Park Lake Avenue, Suite 400 | , eot. |
| | | Raleigh, NC 27612 | eille. |
| _ | Phone: | ONITED STATES | idions |
| | Fax: | | Ague |
| This document cal | inot be used to si | PRA Health Sciences 4130 Park Lake Avenue, Suite 400 Raleigh, NC 27612 UNITED STATES COPY TO A COPY TO | |


# **SERIOUS ADVERSE EVENT REPORTING**

| Γ | | |
|---|---|---|
| | | Serious adverse event reporting (24h) |
| | Fax | Europe and Rest of the World: +32 2 386 2421 |
| | | USA and Canada: +1 800 880 6949 or +1 866 890 3175 |
| | Email | Global: DS_ICT@ucb.com |
| This document ce | inot be used | Europe and Rest of the World: +32 2 386 2421 USA and Canada: +1 800 880 6949 or +1 866 890 3175 Global: DS_ICT@ucb.com Global: DS_ICT@ucb.com |


# **TABLE OF CONTENTS**

| LIST OF | ABBREVIATIONS | | 11 |
|---|---|---|---|
| 1 SUM | MARY | | 16 |
| 2 INTI | RODUCTION | | 18 |
| 2.1 Axia | l spondyloarthritis | | 18 |
| 2.1.1 | Clinical studies | | 19 |
| 2.1.2 | Nonclinical studies | | 21 |
| 3 STU | DY OBJECTIVES | | 21 |
| 3.1 Prim | DY OBJECTIVES ary objective ondary objectives or objectives DY VARIABLES ary variable(s) Primary efficacy variable ondary variables Secondary efficacy variables Secondary safety variables or variables Other efficacy variables Other safety variables Other PK and PD variables Other immunological variables Other pharmacogenomic, proteomic, and metabolite va | :00 | 21 |
| 3.2 Seco | ondary objectives | | 22 |
| 3.3 Othe | r objectives | o to | 22 |
| 4 STU | DY VARIABLES | kg | 22 |
| 4.1 Prim | ary variable(s) | ······································ | 22 |
| 4.1.1 | Primary efficacy variable | 0 | 22 |
| 4.2 Seco | ndary variables | ` | 22 |
| 4.2.1 | Secondary efficacy variables | | 22 |
| 4.2.2 | Secondary safety variables | | 23 |
| 4.3 Othe | r variables | | 23 |
| 4.3.1 | Other efficacy variables | | 23 |
| 4.3.2 | Other safety variables | | 24 |
| 4.3.3 | Other PK and PD variables | | 24 |
| 4.3.4 | Other immunological variables | | 24 |
| 4.3.5 | Other pharmacogenomic proteomic, and metabolite va | riables | 24 |
| 5 STU | DY DESIGN | | 25 |
| 5.1 Stud | Other pharmacogenomic proteomic, and metabolite va DY DESIGN y description | | 25 |
| 5.1.1 | Screening Period/Baseline | | 25 |
| 5.1.2 | Double-Bland Period | | |
| 5.1.3 | Dose-Blind Period | | 26 |
| 5.1.4 | Resoue therapy | | 27 |
| 5.1.5 | Safety Follow-Up Visit | | 27 |
| 5.1.6 | Safety monitoring strategy | | 27 |
| 5.437<br>5.1.8 | Imaging evaluation | | 28 |
| <b>3</b> .1.8 | Study duration per subject | | 28 |
| 5.1.9 | Planned number of subjects and site(s) | | 28 |
| 5.1.10 | Anticipated regions and countries | | 28 |
| 5.2 Sche | edule of study assessments | | 28 |
| 5.3 Sche | matic diagram | | 34 |
| 5.4 Ratio | onale for study design and selection of dose | | 35 |

| 6 | SELECTION AND WITHDRAWAL OF SUBJECTS | 35 |
|---|---|---|
| 6.1 | 1 Inclusion criteria | 35 |
| 6.2 | 2 Exclusion criteria | 37 |
| 6.3 | 3 Withdrawal criteria | 41 |
| ( | 6.3.1 Potential drug-induced liver injury IMP discontinuation criteria | 43 |
| 7 | STUDY TREATMENTS | 43 |
| 7.1 | Description of investigational medicinal products Treatments to be administered Packaging Labeling Handling and storage requirements Drug accountability Procedures for monitoring subject compliance Concomitant medication(s)/treatment(s) | 43\0 |
| 7.2 | 2 Treatments to be administered | 44 |
| 7.3 | 3 Packaging | 544 |
| 7.4 | 4 Labeling | <u></u> |
| 7.5 | 5 Handling and storage requirements | 44 |
| 7.6 | 5 Drug accountability | 45 |
| 7.7 | 7 Procedures for monitoring subject compliance | 45 |
| 7.8 | 3 Concomitant medication(s)/treatment(s) | 45 |
| | 7.8.1 Permitted concomitant treatments (medications and therapies) | 46 |
| | 7.8.2 Prohibited concomitant treatments (medications and therapies) | 46 |
| 7.9 | 9 Blinding. | 47 |
| | 7.9.1 Procedures for maintaining and breaking the treatment blind | 48 |
| | 7.9.1.1 Maintenance of study treatment blind | 48 |
| | 7.9.1.2 Breaking the treatment blindin an emergency situation | |
| | 10 Randomization and numbering of subjects | 49 |
| 8 | STUDY PROCEDURES BY VISIT | 49 |
| 8.1 | | 49 |
| 8.2 | 2 Baseline (Day 1, first dose of TMP) (Visit 2) | 51 |
| | 3 Double-Blind Period (Week 1 to Week 12) | 52 |
| | 8.3.1 Week 1 (+/-3 days) (Visit 3) | |
| | 8.3.2 Week 2 (+/-3 days) (Visit 4) | |
| | 8.3.3 Week 4.0+/-3 days) (Visit 5) | |
| | 8.3.4 Week 8 (+/-3 days) (Visit 6) | |
| | 8.3.5 Week 12 (+/-3 days) (Visit 7) | |
| 8.4 | 4 Dose Blind Period (Week 16 to Week 48) | |
| } | 8.4.1 Week 16 (+/-4 days) (Visit 8) | |
| ~0\ | 8.4.2 Week 20 (+/-4 days) (Visit 9) | |
| * | | |
| | 8.4.4 Week 28 (+/-4 days) (Visit 11) | |
| | 8.4.5 Week 32 (+/-4 days) (Visit 12) | |
| | 8.4.6 Week 36 (+/-4 days) (Visit 13) | |
| 7 | 8.4.7 Week 40 (+/-4 days) (Visit 14) | 60 |

| 8.4 | 4.8 Week 44 (+/-4 days) (Visit 15) | 61 |
|---|---|---|
| 8.4 | 4.9 Week 48 (+/-4 days) (Visit 16) | 61 |
| 8.5 | Early Termination Visit | 62 |
| 8.6 | Safety Follow-Up Visit (20 weeks [-3 days/+7 days] after the final dose) | 64 |
| 8.7 | Unscheduled Visit | 65 |
| 9 | ASSESSMENT OF EFFICACY | 65 |
| 9.1 | ASAS20, 40, ASAS 5/6 response, and ASAS partial remission | 65 |
| 9.2 | Patient global assessment | 66 |
| 9.3 | Total and nocturnal spinal pain | 66 |
| 9.4 | Function – BASFI | 66 |
| 9.5 | Inflammation – BASDAI (mean of questions 5 and 6) | 66 |
| 9.6 | CRP 66 | |
| 9.7 | ASDAS-CRP | 67 |
| 9.8 | BASDAI | 67 |
| 9.9 | BASMI | 67 |
| 9.10 | MASES | 68 |
| 9.11 | PhGADA | 68 |
| 9.12 | ASAS20, 40, ASAS 5/6 response, and ASAS partial remission Patient global assessment Total and nocturnal spinal pain Function – BASFI Inflammation – BASDAI (mean of questions 5 and 6) CRP 66 ASDAS-CRP BASDAI BASMI MASES PhGADA SF-3668 MOS-12 ASQoL MRI Assessment (SPARCC and ASspiMRI) Hospital Anxiety and Depression Scale | |
| 9.13 | MOS-12 | 68 |
| 9.14 | ASQoL C 150 | 69 |
| 9.15 | MRI Assessment (SPARCC and ASspiMRI) | 69 |
| 9.16 | Hospital Anxiety and Depression Scale | 70 |
| | ASSESSMENT OF PHARMACOKINETIC, PHARMACODYNAMIC, | |
| | PHARMACOGENOMIC, AND PROTEOMIC VARIABLES | |
| | ASSESSMENT OF IMMUNOLOGICAL VARIABLES | |
| 12 | ASSESSMENT OF SAFETY | 71 |
| 12.1 | Adverse events | 71 |
| 12 | .1.1 Definition of adverse event | |
| 12 | .1.2 Adverse events of special interest | |
| 12 | .1.3 Adverse events for special monitoring | 71 |
| 12 | .1.4 Procedures for reporting and recording adverse events | 72 |
| 12 | .1.4 Procedures for reporting and recording adverse events Description of adverse events 1.6 Follow-up of adverse events | 72 |
| 12 | 1.6 Follow-up of adverse events | 72 |
| (©12 | .1.7 Rule for repetition of an adverse event | 73 |
| 12 | .1.8 Pregnancy | 73 |
| 12 | .1.9 Suspected transmission of an infectious agent via a medicinal product | 74 |
| 12 | .1.10 Overdose of investigational medicinal product | 74 |
| 12 | 1.11 Safety signal detection | 74 |

| 12.2 Serio | us adv | erse events | 75 |
|---|---|---|---|
| 12.2.1 | Defi | nition of serious adverse event | 75 |
| 12.2.2 | Proc | cedures for reporting serious adverse events | 75 |
| 12.2.3 | | ow-up of serious adverse events | |
| 12.3 Imme | ediate 1 | reporting of adverse events | 76 |
| 12.4 Antic | ipated | serious adverse events | 76 |
| 12.5 Labor | ratory | measurements | 77 |
| 12.5.1 | Eva | luation of PDILI | 78 |
| 12.5 | .1.1 | Consultation with Medical Monitor and local hepatologist Immediate action: determination of IMP discontinuation IMP restart/rechallenge Testing: identification/exclusion of alternative etiology | §82 |
| 12.5 | .1.2 | Immediate action: determination of IMP discontinuation | 82 |
| 12.5 | .1.3 | IMP restart/rechallenge | 82 |
| 12.5 | .1.4 | Testing: identification/exclusion of alternative etiology | 82 |
| 12.5 | .1.5 | Follow-up evaluation | 84 |
| 12.6 Other | safety | Follow-up evaluation measurements l signs y weight and height sical examination ead electrocardiogram erculosis and TB risk factor assessment and management | 84 |
| 12.6.1 | Vita | l signs | 84 |
| 12.6.2 | Bod | y weight and height | 85 |
| 12.6.3 | Phys | sical examination | 85 |
| 12.6.4 | 12-1 | ead electrocardiogram | 85 |
| 12.6.5 | Tub | erculosis and TB risk factor assessment and management | 85 |
| 12.6 | 0.5.1 | Tuberculosis assessment by to RA | 8/ |
| | 5.5.2 | Chest x-ray for tuberculosis | |
| | 5.5.3 | Tuberculosis questionnaire | |
| | 5.5.4 | Tuberculosis management | |
| 12.6.6 | | gnancy testing | |
| 12.6.7 | | essment of suicidal ideation and behavior | |
| | | UDY MEASUREMENTS | |
| | | yzu | |
| 13.2 Medi | cal his | toryO | 89 |
| | | spondylitis history | |
| | V 1- | oncomitant medications. | |
| 1/- | | ANAGEMENT AND ADMINISTRATION | |
| | | to protocol | |
| 14.2 Moni<br>14.2.1 | | | |
| )· | | inition of source data | |
| 14.2.2 | | rce data verification | |
| | | ng | |
| 14.3.1 | | e Report Form completion | |
| 14.3.2 | Dala | abase entry and reconciliation | 91 |

| 14.3.3 Subject Screening and Enrollment log/Subject Identification Code list | 92 |
|---|---|
| 14.4 Termination of the study | 92 |
| 14.5 Archiving and data retention | 92 |
| 14.6 Audit and inspection | 92 |
| 14.7 Good Clinical Practice | 93 |
| 15 STATISTICS | 93 |
| 15.1 Definition of analysis sets | 93 |
| 15.2 General statistical considerations | 94 |
| 15.3 Planned efficacy analyses | 94 |
| 15.3.1 Analysis of the primary efficacy variable | 94 |
| 15.3.1.1 Supportive analyses | 95 |
| 15.3.2 Other efficacy analyses | 95 |
| 15.3.2.1 Analysis of the secondary efficacy variables | 95 |
| 15.3.2.2 Analysis of the other efficacy variables | 96 |
| 15.4 Subgroup analyses | 96 |
| 15.5 Planned safety and other analyses | 96 |
| 15.5.1 Safety analyses | 96 |
| 15.5.2 Other analyses. | 97 |
| 15.3.2.2 Analysis of the other efficacy variables 15.4 Subgroup analyses 15.5 Planned safety and other analyses 15.5.1 Safety analyses 15.5.2 Other analyses 15.6 Handling of protocol deviations 15.7 Handling of dropouts or missing data | 97 |
| 15.7 Handling of dropouts or missing data | 97 |
| 13.8 Planned interim analysis and data monitoring | 99 |
| 15.9 Determination of sample size. | 99 |
| 16 ETHICS AND REGULATORY REQUIREMENTS | . 100 |
| 16.1 Informed consent | . 100 |
| 16.2 Subject identification cards | . 100 |
| 16.3 Institutional Review Boards and Independent Ethics Committees | . 100 |
| 16.4 Subject privacy | .101 |
| 16.5 Protocol amendments | .101 |
| 17 FINANCE INSURANCE, AND PUBLICATION | . 102 |
| 18 REFERENCES | . 102 |
| 19 APPENDICES | . 106 |
| 19.1 Modified New York (mNY) Classification Criteria for AS | . 106 |
| 19.2 Markedly abnormal laboratory values | |
| 9.3 Protocol Amendment 1 | |
| 20 DECLARATION AND SIGNATURE OF INVESTIGATOR | . 142 |
| 21 SPONSOR DECLARATION | 143 |

# LIST OF TABLES

| | LIST OF TABLES | |
|---|---|---|
| Table 5–1: | Schedule of study assessments | 29 |
| Table 7–1: | Prohibited or restricted medications and required wash-out periods prior to Baseline | 46 |
| Table 7–2: | Preparation of placebo and bimekizumab injections | 48 |
| Table 12–1: | Anticipated serious adverse events for the population of subjects with ankylosing spondylitis Laboratory measurements Required investigations and follow-up for PDILI PDILI laboratory measurements PDILI information to be collected Modified New York (mNY) Classification Criteria for AS | |
| Table 12–2: | Laboratory measurements. | 78 |
| Table 12–3: | Required investigations and follow-up for PDILI | 80 |
| Table 12–4: | PDILI laboratory measurements | 83 |
| Table 12–5: | PDILI information to be collected | 84 |
| Table 19–1: | Modified New York (mNY) Classification Criteria for AS | 106 |
| Table 19–2: | Definitions of markedly abnormal hematology values | 107 |
| Table 19–3: | Definitions of markedly abnormal biochemistry values | 107 |
| Figure 5–1: | Definitions of markedly abnormal hematology values Definitions of markedly abnormal biochemistry values LIST OF FIGURES Schematic diagram LIST OF FIGURES Schematic diagram | 34 |


**UCB** Clinical Study Protocol 09 Mar 2018 AS0008

# LIST OF ABBREVIATIONS

AE adverse event

**AESI** adverse event of special interest

**AESM** adverse event for special monitoring

**ALP** alkaline phosphatase

**ALT** alanine aminotransferase **ANCOVA** analysis of covariance

AS ankylosing spondylitis

ASAS Assessment of SpondyloArthritis International Society

Assessment in SpondyloArthritis International Society 20%, 40%, 5 out ASAS20, 40, 5/6

of 6 response criteria

Ankylosing Spondylitis Disease Activity Score-C-reactive protein **ASDAS-CRP ASDAS-MI** Ankylosing Spondylitis Disease Activity Score major improvement Ankylosing Spondylitis spine Magnetic Resonance Imagine-activity ASspiMRI-a

Ankylosing Spondylitis Quality of Life **ASQoL** 

aspartate aminotransferase **AST** 

axSpA axial spondyloarthritis

Bath Ankylosing Spondylitis Disease Activity Index **BASDAI** 

Bath Ankylosing Spondylitis Functional Index **BASFI** 

**BASMI** Bath Ankylosing Spondylitis Metrology Index

**BSA** body surface area

**CDC** Centers for Disease Control

**CDMS** clinical data management system

**CHO** Chinese Hamster Ovarian

CL/F total body clearance

COX-2 inhibitor cyclooxygenase 2 inhibitor Clinical Project Manager

**CPMP** Committee for Proprietary Medicinal Products

his docurero contract research organization

C-reactive protein

C-SSRS/eC-SSRS Columbia-Suicide Severity Rating Scale/electronic C-SSRS

**CZP** certolizumab pegol

Dose-Blind Responder Set **DBRS** 

DBS Dose-Blind Set

**DMARD** disease-modifying antirheumatic drug

**Data Monitoring Committee DMC** 

disco-vertebral unit **DVU ECG** electrocardiogram

eCRF electronic Case Report Form

**EDC** electronic data capture

ES Enrolled Set

**ESS Escape Subject Set FAS** Full Analysis Set

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice **GFR** glomerular filtration rate

GI gastrointestinal

on application and any extensions of variations thereof. Hospital Anxiety and Depression Scale **HADS** 

Hospital Anxiety and Depression Scale—Anxiety HADS-A

Hospital Anxiety and Depression Scale—Depression HADS-D

HbcAg hepatitis B core antibody HbsAg hepatitis B surface antigen

**HBV** hepatitis B virus hepatitis C virus **HCV** 

human immunodeficiency virus HIV

human leukocyte antigen HLA HRQoL health-related quality of life

hs-CRP high sensitivity C-reactive protein

IB Investigator's Brochure

IBD inflammatory bowel disease

International Council for Harmonisation

Informed Consent Form

**Independent Ethics Committee** 

**IGRA** Interferon-Gamma Release Assay IIV interindividual variability

ILinterleukin im intramuscular

**IMP** investigational medicinal product

Institutional Review Board **IRB** 

**IUD** intrauterine device

**IUS** intrauterine hormone-releasing system

iv intravenous

**IXRS** interactive voice or web response system

latent tuberculosis LTB

latent tuberculosis infection LTBI

MAR missing at random

and any extensions of variations thereoff. Maastricht Ankylosing Spondylitis Enthesitis Index **MASES** 

minimal clinically important difference **MCID** 

multiple comparison procedure - modeling MCP-Mod

**MCS** mental component summary

MedDRA<sup>®</sup> Medical Dictionary for Regulatory Activities

multiple imputation MI measles-mumps-rubella **MMR** 

mNY Modified New York (criteria)

MOS Medical Outcomes Study

magnetic resonance imaging MRI mycobacterium tuberculosis **MTB** 

methotrexate **MTX** 

nonradiographic-axial spondyloarthritis nr-axSpA

**NRI** nonresponder imputation Numeric Rating Scale **NRS** 

**NSAID** nonsteroidal anti-inflammatory drug

NY NY nontuberculous mycobacteria New York Heart Association

**OMERACT** Outcome Measures in Rheumatology Clinical Trials

**OPV** oral polio vaccine

physical component summary PCS

PD pharmacodynamics

**PDILI** potential drug-induced liver injury PD-PPS Pharmacodynamics Per-Protocol Set

**PGADA** Patient's Global Assessment of Disease Activity

**PhGADA** Physician's Global Assessment of Disease Activity

PK pharmacokinetics

**PK-PPS** Pharmacokinetic Per-Protocol Set

**PPS** Per-Protocol Set PS **Patient Safety PsA** psoriatic arthritis

Q4W every 4 weeks (monthly)

and any extensions of variations thereof. QT interval corrected for heart rate using Bazett's formula **QTcB** 

QT interval corrected for heart rate using Fridericia's formula QTcF

RA rheumatoid arthritis

**RIF** mycobacterium tuberculosis rifampicin

RS Randomized Set

Rheumatology Common Toxicity Criteria **RCTC** 

residual unexplained variability RUV

SAE serious adverse event SAP Statistical Analysis Plan

subcutaneous(ly) SC standard deviation SD

SF-36 Short-Form 36-item Health Survey

**SFU** Safety Follow-up

SI sacroiliac

spondyloarthritis

**SPARCC** Spondyloarthritis Research Consortium of Canada

standard operating procedure

his docursop Safety Set sulfasalazine

> **STIR** short-tau-inversion recovery

The document control be used to support any materials as the control of the contr

# SUMMARY

This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group,

Eligible subjects will have active AS, determined by documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984), including symptoms for  $\geq 3$  months age of onset <45. Furthermore, subjects will have moderate to several Ankylosing Spondylitis Disease Activity In 1900 Question 21) Subjects will be subjected by Subjects will have moderate to several Ankylosing Spondylitis Disease Activity In 1900 Question 210 Subjects will have moderate to several Ankylosing Spondylitis Disease Activity In 1900 Question 21 Question 2]). Subjects must have at least 1 of the following: 1) inadequate response to nonsteroidal anti-inflammatory drug (NSAID) therapy, 2) intolerance to administration of at least 1 NSAID, or 3) contraindication(s) to NSAID therapy. Inadequate response to an NSAID is defined as lack of response for at least 4 weeks of continuous NSAID therapy at the highest tolerated dose of the administered NSAID or the lack of response to treatment with at least 2 NSAIDs at the maximum tolerated dose for at least 4 weeks total duration. Subjects may be TNF inhibitor-naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:

- experienced an inadequate response to previous treatment given for at least 3 months
- been intolerant to administration (eg, had a side effect/AE that led to discontinuation)
- lost access to TNF inhibitor for other reasons

The primary objective is to assess the dose-response based on the efficacy of bimekizumab administered subcutaneously (sc) Q4W for 12 weeks in the treatment of subjects with active AS. The primary efficacy variable is the Assessment in Axial SpondyloArthritis International Society 40% response criteria (ASAS40) response at Week 12. An ASAS40 response is defined as an improvement of  $\ge 40\%$  and  $\ge 2$  units in at least 3 out of the following 4 domains on a scale of 0 to 10 and no worsening at all in the remaining domain and includes the following assessments:

- Patient global assessment: numeric rating scale (NRS) (global disease activity last week)
- Pain assessment: NRS (last week/spine/at night due to AS)
- Function: Bath Ankylosing Spondylitis Functional Index (BASFI)
- Inflammation: mean of BASDAI Questions 5 and 6

The secondary objectives of the study are to assess the efficacy of the individual dose regimens of bimekizumab compared to placebo, safety and tolerability, PK, PD, immunogenicity, and the exposure:response relationship of bimekizumab as it relates to efficacy and safety. The secondary efficacy variables include: Change from Baseline in Ankylosing Spondylitis Disease Activity Score- C-reactive protein (ASDAS-CRP), Assessment in Axial SpondyloArthritis International Society 20% response criteria (ASAS20) response, Assessment in Axial SpondyloArthritis International Society 5 out of 6 response criteria (ASAS5/6) response, Change from Baseline in BASDAI, and Change from Baseline in BASFI, all at Week 12. Safety variables include incidence of adverse events (AEs), serious adverse events (SAEs), and withdrawal due to AEs as secondary safety variables and change from Baseline in vital signs,


09 Mar 2018 AS0008

body weight, physical examination, ECG, and clinical laboratory variables as other safety variables.

Other objectives are to assess the impact on patient-reported quality of life (fatigue, sleep, and Proteomic analysis of subject samples and evaluation of the potential for subject stratification approaches, and to assess the impact of bimekizumab on inflammatory changes in the spine and sacroiliac (SI) joint using magnetic resonance imaging (MRI) in a subset of subjects.

An estimated 100 sites in Europe and North American per treatment arm) Ti

per treatment arm). The enrollment of TNF inhibitor-experienced subjects will be limited to 30% of the total study population.

The study consists of a Screening Period (up to 28 days), Double-Blind Period (12 weeks), Dose-Blind Period (36 weeks) and Safety Follow-up (SFU) Period (20 weeks; only for subjects who do not enter the extension study). Therefore, the maximum duration of the study is 68 weeks.

# Screening Period/Baseline

The Screening Period will be up to 28 days. During the Screening Period, the Investigator will assess the eligibility of subjects according to the inclusion and exclusion criteria. The Screening Period will also enable washout of any medications not permitted for use during the study and allow initiation of latent TB treatment where necessary and appropriate.

# **Double-Blind Period**

At Baseline/Day 1 subjects will be randomized in a 1:1:1:1:1 ratio (stratified by region and prior TNF inhibitor exposure) to receive the following blinded study treatment regimens during the Double-Blind Period:

- Placebo
- Bimekizumab 16mg administered sc every 4 weeks (Q4W)
- Bimekizumab 64mg administered sc Q4W
- Bimekizumab 160mg administered sc Q4W
- Bimekizumab 320mg administered sc Q4W

The investigational medicinal product (IMP) will be administered sc in the clinic at Baseline, Week 4, Week 8, and Week 12. Additional study visits in the Double-Blind Period (without dosing) will occur at Week 1 and Week 2. At Week 12, subjects will transition from the Double-Blind Period into the 36-week Dose-Blind Period.

09 Mar 2018 AS0008

# Dose-Blind Period

The Dose-Blind Period lasts from Week 12 to Week 48. Subjects randomized to bimekizumab 160mg Q4W or bimekizumab 320mg Q4W will remain on their randomized dose and subjects randomized to placebo, bimekizumab 16mg Q4W, and bimekizumab 64mg Q4W, will be rerandomized in a 1:1 fashion to bimekizumab 160mg Q4W or bimekizumab 320mg Q4W. The total duration of treatment is 48 weeks.

During the 36-week Dose-Blind Period, subjects will be evaluated for eligibility to rescue treatment at defined time points. Subjects who do not show an improvement in both PGADA and spinal pain compared to Baseline will be eligible to receive rescue therapy as defined in Section 5.1.4.

# Safety Follow-Up (SFU) Visit/Extension study

At the completion of the Dose-Blind Period, subjects will be given the opportunity to enter an extension study at Week 48. All subjects who complete the study and do not enter the extension study or who discontinue early, including those withdrawn from study treatment, will have a SFU Visit at 20 weeks after their last dose of IMP.

# 2 INTRODUCTION

# 2.1 Axial spondyloarthritis

Spondyloarthritis (SpA) is an umbrella term applied to a family of rheumatic diseases (including axial spondyloarthritis [axSpA], psoriatic arthritis [PsA], reactive arthritis, the arthritis of inflammatory bowel disease [IBD], and undifferentiated spondyloarthritis) that have features in common with each other and distinct from other inflammatory arthritides, particularly rheumatoid arthritis (RA).

Axial SpA is a chronic inflammatory disease that impacts a substantial proportion of the population. Limited evidence exists regarding the exact prevalence of axSpA; however, recent data suggest that the prevalence is similar to that of RA in the US (axSpA: 0.7% to 1.4%; RA: 0.5% to 1.0%) (Reveille et al, 2012; Myasoedova et al, 2010; Helmick et al, 2008).

The ASAS working group established classification criteria to distinguish 2 broad categories of SpA: peripheral SpA and axSpA (Rudwaleit et al, 2011; Rudwaleit, 2010; Rudwaleit et al, 2009b). This division is based on the body part predominantly involved in the inflammatory process. Therefore, peripheral SpA includes diseases affecting mainly peripheral joints, such as reactive arthritis and PsA, whereas axSpA comprises those diseases with mainly axial involvement (SI joints and spine), including AS diagnosed with radiographic involvement and nonradiographic axSpA (nr-axSpA).

Patients with axSpA have inflammatory back pain. The disease typically originates in the sacroiliac joints, then progresses to the spine. In the sacroiliac joints and the spine, active inflammation results in erosions, sclerosis, and fatty lesions seen on MRI. However, the most characteristic feature is new bone formation leading to ankylosis of the SI joints and syndesmophytes attached to the vertebral bodies. As a result of extended syndesmophyte formation, over time the spine may become fused. Objective signs of inflammation (such as enthesitis, dactylitis, peripheral arthritis, or uveitis), genetic features (such as the presence of human leukocyte antigen [HLA] B27), and laboratory parameters (such as elevated C-reactive

protein [CRP]) may also be present (Braun, 2012; Rudwaleit et al. 2009a; Braun and Sieper, 2007). Disability in axSpA is related to both the degree of inflammatory activity, causing pain, stiffness, fatigue, and poor quality of sleep, and to the degree of bony ankylosis, causing loss of

Nonsteroidal anti-inflammatory drugs are often rapidly effective for the symptoms (pain and stiffness) of axSpA (Poddubnyy, 2013; Poddubnyy et al, 2012), but many patients lose or make the clinically meaningful response and structural damage often processor of the fibrous ring of the symptoms (pain and stiffness) of axSpA (Poddubnyy, 2013; Poddubnyy et al, 2012), but many patients lose or make the clinically meaningful response and structural damage often processor of the fibrous ring of the symptoms (pain and stiffness) of axSpA (Poddubnyy, 2013; Poddubnyy et al, 2012), but many patients lose or make the symptoms (pain and stiffness) of axSpA (Poddubnyy, 2013; Poddubnyy et al, 2012), but many patients lose or make the symptoms (pain and stiffness) and stiffness) of axSpA (Poddubnyy, 2013; Poddubnyy et al, 2012), but many patients lose or make the symptoms (pain and stiffness) and stiffness (pain and stiffness) are stiffness (pain and stiffness). sulfasalazine [SSZ]) have no proven efficacy in axial disease, but may benefit patients with peripheral joint disease (Haibel et al, 2007; Braun et al, 2006; Haibel et al, 2005). Therefore, DMARDs are recommended only in patients with predominantly peripheral manifestations (Braun et al, 2011). Patients who are intolerant of or have inadequately responded to NSAIDs, or those in whom NSAIDs are contraindicated, have approved treatment options such as TNF inhibitors.

Recently, the interleukin (IL)-17 cytokine family has been identified as a therapeutic target in axSpA and secukinumab, an IL-17A monoclonal antibody, has recently been approved as a treatment option in active AS.

Bimekizumab (UCB4940) is an engineered, humanized full-length monoclonal antibody of IgG1 subclass of approximately 150,000 Dalton, which is expressed in a genetically engineered Chinese Hamster Ovarian (CHO) cell line, Bimekizumab has high affinity for human IL-17A and human IL-17F and selectively and potently inhibits the activity of both isoforms in vitro. Interleukin-17A and IL-17F are key proinflammatory cytokines believed to play important roles in autoimmune and inflammatory diseases. Therefore, bimekizumab permits an evaluation of the potential for additional efficacy, which may be conferred by dual inhibition of both cytokines, in patients suffering from diseases in which both cytokines are active. Bimekizumab is being developed for the treatment of patients with inflammatory diseases such as PsA, PsO, and AxSpA.

As a consequence, a Phase 2b dose-ranging study (AS0008) was designed to investigate the efficacy and safety of various bimekizumab dose regimens in subjects with active AS.

#### 2.1.1 **Clinical studies**

Four clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque psoriasis, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, and UP0031 in 12 healthy volunteers.

WP0008 was a Phase 1, single ascending dose study in adults with mild to moderate psoriasis affecting ≤5% body surface area (BSA). In this blinded study, single doses of bimekizumab up to 640mg (approximately 8mg/kg in an 80kg adult) were evaluated. There were no clinically relevant safety findings identified at any dose and all doses were well tolerated. The prespecified exploratory assessment of disease activity showed clinically relevant and statistically significant improvements at the higher doses studied.

RA0124 was a Phase 1, open-label, parallel-group, single-dose study in healthy subjects. The primary objective of this study was to determine the absolute bioavailability of single sc doses of bimekizumab (80mg and 160mg). The secondary objectives were to evaluate the dose proportionality of bimekizumab 80mg and 160mg sc, and to evaluate the safety and tolerability of these sc doses and 160mg given by intravenous (iv) infusion. In RA0124, the absolute bioavailability was similar for the 2 doses tested (0.656 and 0.631 for the bimekizumab 80mg and 160mg sc doses, respectively). The median half-life (t<sub>1/2</sub>) following sc administration was similar to that following iv administration (27.81 days and 28.25 days for bimekizumab 160mg sc and bimekizumab 160mg iv, respectively).

Bimekizumab has also been investigated in a Phase 1b, proof of concent randomic in placebo-controlled, multiple-dose study (PA0007).

Bimekizumab has also been investigated in a Phase 1b, proof of concept, randomized, placebo-controlled, multiple-dose study (PA0007). The primary objective of PA0007 was to assess the safety and PK of multiple dose administration of iv bimekizumab in subjects with PsA. Four active doses and a placebo were tested. Drug was administered as a loading dose of bimekizumab 80mg, 160mg, 240mg, or 560mg at Week 1, and 2 additional doses of bimekizumab 40mg, 80mg, 160mg, or 320mg at Week 4 and Week 7. In each treatment group, subjects received a total of 3 doses of bimekizumab, administered every 3 weeks. There were no unexpected clinically relevant safety findings and all doses were well tolerated. The PK was linear across the tested dose range and no change in PK was observed following multiple doses. Observed changes in inflammatory biomarkers were consistent with expectations based on the IL-17A and IL-17F mechanism of action. The exploratory analysis showed clinically relevant improvement in activity of PsA and in skin involvement in those subjects with concomitant active psoriatic lesions. Data from the top 3 bimekizumab dose groups pooled showed that by Week 9 80% [95% CI: 62.7, 90.5] of subjects achieved an ACR20 response (vs 16.7% [95% CI: 4.7, 44.8] in the placebo group) and 100% [95% CI: 79.6, 100.0] of subjects with active psoriatic lesions had achieved a PASI75 response (vs 0% [95% CI: 0.0, 43.4] in the placebo group).

Infections (mostly nasopharyngitis) were the most commonly reported events in both the active (36.8% of subjects) treatment and the placebo group (35.7% of subjects). None of the infections were considered serious or required treatment with antibiotics. Two subjects in the active treatment group experienced 1 local candida infection each (oropharyngitis and vulvovaginitis, respectively) that were nonserious and resolved with topical therapy. There was a reduction in mean neutrophil count in the active treatment group, although this drop was not clinically relevant and a clear relationship with dose or time was not evident. IL-17 plays a significant role in regulating neutrophil recruitment and granulopoiesis and thus, receipt of an anti-IL-17 antibody may be associated with effects on neutrophil count. Previous clinical experience with administration of anti-IL-17 antibodies in humans indicates that this potential risk is low and reversible. Some increases in liver function tests were reported, but none had a convincing relationship to exposure to IMP.

In the bimekizumab clinical studies to date, the most commonly reported GI AEs were abdominal distension, abdominal pain, diarrhea, flatulence, nausea, and vomiting. All of these events, except 1 event of vomiting, were mild or moderate in intensity. T helper-17 and other IL-17-producing cell types are present in a high frequency in the physiologic, healthy state of the intestinal mucosa. Interleukin-17 is recognized as an important player in the pathophysiology of infectious and immune-mediated GI diseases, and has been shown to contribute to the gut barrier function (Ivanov et al. 2008). Clinical data with secukinumab suggest that the drug may worsen

symptoms of co-existing Crohn's disease in patients with psoriasis and ankylosing spondylitis (Baeten et al 2015).

UP0031 was a Phase 1, open-label, parallel-group, randomized, single-dose study to evaluate the BA, PK, and tolerability of 2 different formulations of bimekizumab in healthy subjects. There were no treatment-emergent adverse events (TEAEs) leading to discontinuation, and no SAEs or fatalities were reported.

One additional study of bimekizumab is ongoing. RA0123 is a Phase 2a, double-blind, randomized, placebo-controlled, multiple dose study to evaluate the safety, PK, PD, and efficacy of multiple doses of bimekizumab administered as add-on therapy to stable certolizumab pegol (CZP; Cimzia<sup>®</sup>) therapy in subjects with moderate to severe RA.

Additional information on the clinical data for bimekizumab is available in the current version of the Investigator's Brochure (IB).

## 2.1.2 Nonclinical studies

Parallel inhibition of IL-17A and IL-17F has shown potent effects in a variety of animal models of inflammatory disease. Intravenously administered bimekizumab was well tolerated in repeat dose toxicology studies in Cynomolgus monkeys with a no adverse effect level of 200mg/kg/week. The findings of note in toxicity studies were diarrhea related to infectious enteritis (observed in the single dose study) and asymptomatic mild colonic ulceration in a proportion of animals (in the repeat-dose study); this latter finding was not associated with hematology abnormalities. Data suggest that bimekizumab has induced primary lesions to the mucosa-associated lymphoid tissue via a pharmacologically-related mechanism. In a second repeat-dose study, none of the minor apoptosis/necrosis findings observed in gut associated lymph nodes were seen. In animals given the highest dose of bimekizumab in the study (20mg/kg/week), a slightly higher number of protozoa (*Balantidium coli*) was observed in the cecum and colon as compared to the control animals and low dose animals. Therefore, the gut-associated lymph node lesions observed in the first study are considered to be accidental and/or linked to exaggerated pharmacology and proliferation of *Balantidium coli* and are considered to be the result of a change in local mucosal immunity.

Additional information on the nonclinical data for bimekizumab is available in the current version of the IB.

# 3 STUDY OBJECTIVES

This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group dose-ranging study to evaluate the efficacy and safety of bimekizumab in subjects with active AS.

# 3.1 Primary objective

The primary objective is to assess the dose-response based on the efficacy of bimekizumab administered sc Q4W for 12 weeks in the treatment of subjects with active AS.

#### 3.2 Secondary objectives

The secondary objectives of the study are as follows:

- , or variations thereof. To assess the efficacy of the individual dose regimens of bimekizumab compared to placebo
- To assess the safety and tolerability of bimekizumab
- To assess the PK of bimekizumab
- To assess the PD of bimekizumab
- To assess the immunogenicity of bimekizumab
- To assess the exposure:response relationship of bimekizumab as it relates to efficacy and safety

#### 3.3 Other objectives

- To assess disease activity
- To assess the impact on patient-reported quality of life (function, fatigue, sleep, and pain)
- To assess the impact on enthesitis
- To assess the impact of administration of bimekizumab on biological pathways relating to disease biology, progression, and response to therapy via biomarker analysis, and to enable genomic and related approaches for analysis of subject samples and evaluation of the potential for subject stratification approaches
- To assess the impact of bimekizumab on inflammatory changes in the spine and SI joint using MRI in a subset of subjects.

#### 4 STUDY VARIABLES

#### Primary variable(s) 4.1

#### Primary efficacy variable 4.1.1

The primary efficacy variable for this study is as follows:

ASAS40 response at Week 12

#### 4.2 Secondary variables

#### 4.2.1 Secondary efficacy variables

The secondary efficacy variables for this study are as follows:

- Change from Baseline in ASDAS-CRP at Week 12
- ASAS20 response at Week 12
- ASAS5/6 response at Week 12
- Change from Baseline in BASDAI at Week 12
- Change from Baseline in BASFI at Week 12

#### 4.2.2 Secondary safety variables

Assessment time points for safety variables are specified in Table 5–1. Variables are as follows:

- Incidence of AEs and SAEs
- Withdrawal due to AEs

#### 4.3 Other variables

#### 4.3.1 Other efficacy variables

Assessment time points for the other efficacy variables are specified in Table 5–1 (analyses at all time points not specified in Section 4.1.1 or Section 4.2.1 are exploratory). Variables are as and any extensic follows:

- ASAS40 response
- Time to ASAS40 response
- Change from Baseline in ASDAS-CRP
- ASDAS status (eg, inactive disease, moderate, high and very high disease activity)

- ASAS20 response
  Time to ASAS20 response
  ASAS5/6 response
  Ankylosing Spondylitis Disease Activity Score major improvement (ASDAS-MI)
- ASAS partial remission
- Change from Baseline in BASD
- Change from Baseline in BASFI?
- Change from Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
- Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index
- Physician's Global Assessment of Disease Activity (PhGADA)
- Change from Baseline in Patient's Global Assessment of Disease Activity (PGADA)
- Change from Baseline in total and nocturnal spinal pain (NRS)
- Change from Baseline in the average of Questions 5 and 6 of the BASDAI



- Change from Baseline in Sleep quality (Medical Outcomes Study [MOS]-12 item scale)
- Change from Baseline in Ankylosing Spondylitis Quality of Life (ASQoL)

- Change from Baseline in:
  - Spondyloarthritis Research Consortium of Canada (SPARCC) MRI index for Assessment
- Change from Baseline in Hospital Anxiety and Depression Scale Anxiety (HADS-A) and Hospital Anxiety and Depression (HADS-D) scores

  Percentage of subjects with scores below 8 in HADS scores)

#### 4.3.2 Other safety variables

Assessment time points for other safety variables are specified in Table 5–1. Variables are as follows:

- Change from Baseline in vital signs (blood pressure, pulse rate) and body weight
- Standard 12-lead electrocardiogram (ECG) intervals (RR, PR, QRS, QT, and QT intervals corrected for heart rate using Bazett's and Fridericia's formulas [QTcB and QTcF]), including changes from Baseline Electrocardiogram (ECG) variables
- Change from Baseline in clinical laboratory variables (hematology, biochemistry, and urinalysis)

#### Other PK and PD variables 4.3.3

- The PK variables are plasma concentrations of bimekizumab.
- The PD variables are concentrations of cytokines of relevance to the IL-17A/F signaling pathway and AS biology, and include but are not limited to IL-17A, IL-17F, IL-23, IL-6, and TNFα.

#### Other immunological variables 4.3.4

Immunological variables allow evaluation of immunogenicity as well as immunological biomarkers.

- Anti-bimekizumab antibody detection prior to and following study treatment
- Serum complement concentrations.
- Flow cytometry analysis of key immune cell populations, including but not limited to CD3, CD19, CD4, CD8, and CD69 (using fluorescence activated cell sorting).
- Cytokines and other exploratory markers

# Other pharmacogenomic, proteomic, and metabolite variables

docura.3.5 Where local regulations permit, additional blood samples will be collected from consenting subjects at specific time points and stored at -80°C for up to 20 years to allow for potential, exploratory analyses of genomic, genetic, proteomic, and metabolomic biomarkers relevant to disease biology and progression, response to therapy, and the inflammatory and immune response processes.

#### STUDY DESIGN 5

#### 5.1 Study description

Subject has active AS, determined by documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984) (see Table 19–1), including symptoms for  $\geq$ 3 months and age of onset  $\leq$ 45 years. This is a multicenter, Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study to evaluate the efficacy and safety of bimekizumab in subjects with active AS. To be eligible to participate in this study, subjects must meet the following key inclusion criteria:

- - BASDAI score >4
  - Spinal pain  $\geq$ 4 on a 0 to 10 NRS (from BASDAI item 2)
- Subjects must have at least 1 of the following:
  - inadequate response to NSAID therapy
  - intolerance to administration of at least 1 NSAID
  - contraindication(s) to NSAID therapy

- contraindication(s) to NSAID therapy

Inadequate response to an NSAID is defined as lack of response for at least 4 weeks of continuous NSAID therapy at the highest tolerated dose of the administered NSAID or the lack of response to treatment with at least 2 NSAIDs at the maximum tolerated dose for at least 4 weeks total duration.

- Subjects may be TNF inhibitor-naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:
  - experienced an inadequate response to previous treatment given for at least 3 months
  - been intolerant to administration (eg, had a side effect/AE that led to discontinuation)
  - lost access to TNF inhibitor for other reasons

Approximately 285 eligible subjects will be randomized to 1 of 5 treatment arms to receive treatment according to their randomized placebo or bimekizumab dose regimen (Section 5.1.2) until Week 12. Thereafter, subjects randomized to bimekizumab 160mg Q4W or bimekizumab 320mg Q4W will remain on their randomized dose and subjects randomized to placebo, bimekizumab 16mg Q4W, and bimekizumab 64mg Q4W, will be rerandomized in a 1:1 fashion to birnekizumab 160mg Q4W or birnekizumab 320mg Q4W. The total duration of treatment is 48 weeks.

# Screening Period/Baseline

his docurs.1.1 Assessments of eligibility as described in Section 6 will be initiated during the 28-day Screening Period. The Screening Period will also enable the washout of medications not permitted for use during the study and allow initiation of latent TB treatment where necessary.

The assessments at the Screening Period Visit are presented in Table 5–1.

#### 5.1.2 **Double-Blind Period**

At Baseline/Day 1, subjects will be randomized 1:1:1:1:1 (stratified by region and prior Atensions of variations thereof TNF inhibitor exposure) to receive the following blinded IMP treatment regimens at the clinical site. The enrollment of TNF inhibitor-experienced subjects will be limited to approximately 30% of the total study population.

- Placebo
- Bimekizumab 16mg administered sc Q4W
- Bimekizumab 64mg administered sc Q4W
- Bimekizumab 160mg administered sc Q4W
- Bimekizumab 320mg administered sc Q4W

The IMP will be administered sc in the clinic at Baseline and Q4W thereafter up to Week 12. Additional study visits (without dosing) are scheduled at Week 1 and Week 2. At 12 weeks, subjects will transition from the Double-Blind Period into the 36-week Dose-Blind Period, as discussed in Section 5.1.3

Subjects withdrawing early from the study will undergo the Early Termination Visit assessments and will enter the SFU Period.

The assessments during the Treatment Period are presented in Table 5–1.

#### 5.1.3 **Dose-Blind Period**

After the 12-week Double-Blind Period, subjects will enter the 36-week Dose-Blind Period. At the Week 12 Visit, subjects will be allocated to bimekizumab treatment regimens as follows:

- Subjects in the placebo group, bimekizumab 16mg Q4W, or bimekizumab 64mg Q4W will be rerandomized in a 1:1 fashion to bimekizumab 160mg or bimekizumab 320mg Q4W.
- Subjects in the bimekizumab 160mg dose group will continue to receive bimekizumab 160mg Q4W.
- Subjects in the bimekizumab 320mg dose group will continue to receive bimekizumab 320mg O4W.

At the completion of the Dose-Blind Period, Investigators should discuss treatment options with the subject. Subjects will be given the opportunity to enter an extension study at Week 48.

The assessments during the Dose-Blind Period are presented in Table 5–1. This document cannot

# 5.1.4 Rescue therapy

At Weeks 16, 24, and 36 of the Dose-Blind Period, subjects will be evaluated for their response to treatment to determine eligibility for rescue therapy.

Subjects with <10% improvement from Baseline in both PGADA and total and nocturnal spinal pain (ASAS domain response criteria) are eligible for rescue treatment. Rescue therapy will be at the Investigator's discretion, with the following options:

NSAIDS and/or joint injections as outlined below. Subjects may receive these add-on rescue
therapies while continuing to receive their randomized dose of bimekizumab.

For subjects taking NSAID/COX-2 inhibitors at Baseline or at Weeks 16, 24, or 36, a change can be made to a different NSAID/COX-2 inhibitor. Changes from an NSAID to a COX-2 inhibitor or from a COX-2 inhibitor to an NSAID are permitted up to the maximum approved or tolerated dose, whichever is lower. Only 1 NSAID/COX-2 inhibitor may be taken at a given time.

- For subjects not taking NSAID/COX-2 inhibitors at Baseline, Weeks 16, 24, or 36, either NSAIDs, or COX-2 inhibitors can be initiated, up to the maximum approved or tolerated dose, whichever is lower. Only 1 NSAID/COX-2 inhibitor may be taken at a given time.
- After the NSAID/COX-2 regimen has been optimized, SI joint injection is permitted, either unilaterally or bilaterally, performed by a qualified physician.
- If the subject does not achieve sufficient response to the above options and/or the Investigator feels that a biologic other than bimekizumab is warranted, the subject must discontinue from study treatment (bimekizumab) and follow the withdrawal criteria and follow up as outlined in Section 6.3.

A decrease in dose or dosing frequency of any agent for the treatment of AS is permitted for reasons of intolerance/AEs/side effects at any time.

Rescue therapy will be determined by the Investigator taking into account the half-life of bimekizumab (27.8 days).

Subjects may be withdrawn from the study or from study medication at any time and continue treatment per the Investigator's discretion, as described in the Withdrawal Section (Section 6.3).

# 5.1.5 Safety Follow-Up Visit

All subjects who complete the study and do not enter the extension study or who discontinue from the study early, including those withdrawn from IMP treatment, will have a SFU Visit at 20 weeks after their final dose of IMP.

The assessments at the SFU Visit are presented in Table 5–1.

# 51.6 Safety monitoring strategy

An independent Data Monitoring Committee (DMC) will review study safety data on an ongoing basis. Details will be available in the DMC charter. A cardiovascular adjudication committee will review cardiovascular events. Further details are provided in Section 12.1.11.

09 Mar 2018 AS0008

#### 5.1.7 Imaging evaluation

In a subpopulation of AS0008, MRIs of the spine and SI joints will be performed in approximately 20 subjects per treatment arm at Baseline. Magnetic resonance imaging at Week 12 and Week 48 will be performed only for subjects who are MRI-positive at Baseline based on an ASAS-Outcome Measures in Rheumatology Clinical Trials (OMERACT) assessment. The Baseline MRI should be performed after confirmation of eligibility for the study based on screening assessments and before the first bimekizumab injection. Magnetic resonance imaging at Week 12 and Week 48 should be performed as close to the Week 12/Week 48 Visit as possible. Further details are provided in Section 9.15. Analyses will be exploratory in nature and For each subject, the study will last a maximum of up to 68 weeks, as follows:

Screening Period: up to 28 days

Double Blinks will be performed at selected sites.

Double-Blind Period: 12 weeks

Dose-Blind Period: 36 weeks

A SFU Visit: 20 weeks after the final dose of IMP for subjects not entering the extension study or discontinuing from the study early, including those withdrawn from study treatment.

The end of the study is defined as the date of the last visit of the last subject in the study.

#### Planned number of subjects and site(s) 5.1.9

The planned number of randomized subjects is 285; there will be 57 subjects per treatment arm. The planned number of study sites is approximately 100. The enrollment of TNF inhibitor-experienced subjects will be limited to 30% of the total study population.

#### 5.1.10 Anticipated regions and countries

The study sites will be located in Europe and North America.

#### 5.2 Schedule of study assessments

.udy

This document cannot be used to The schedule of study assessments is presented in Table 5–1.

Table 5-1: Schedule of study assessments

| Table 5-1: Schedule of study assessments | assessm | ents | | | | | | | | | | | | *°!, | 2/2 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | gning<br>of qu) (<br>(syr | enile<br>(2 tisiV<br>(9sob | Dool (wee | uble-<br>ks af | Blind<br>ter fil | Double-Blind Period<br>(weeks after first dose) | d (es | | | Dose-Blind Period (weeks after first dose) | Dose-Blind Period<br>eeks after first dos | d Per<br>first | iod (dose) | 6, | | ET | $\mathbf{SFU}^{\mathbf{b}}$ |
| Visit <sup>a</sup> | Seree<br>Seree<br>Seree | , I yr | 3 | 4 | w | 9 | 7 | ∞ | 9 1 | 10 11 | 22 | 13 | 14 | 15 | 16 | | |
| Week <sup>a</sup> | (A) | | 1 | 7 | 4 | ∞ | 12 1 | 16 2 | 20 2 | 24 28 | 30,32 | 36 | 40 | 44 | 48 | | |
| Protocol activity | | | | | | | | | | 40 | | | | | | | |
| Written informed consent | × | | | | | | | | 40 | <b>5.</b> | | | | | | | |
| Demographic data | × | | | | | | | 0/ | 40 | | | | | | | | |
| AS history | × | | | | | - | -1/ | 0 | | | | | | | | | |
| Significant past medical history and concomitant diseases | × | × | | | 5 | (V) | 0/6 / | | | | | | | | | | |
| Inclusion/exclusion criteria | × | × | | A) | (). | (b) | | | | | | | | | | | |
| Prior medication | × | | <i>D</i> | (a). | 04 | | | | | | | | | | | | |
| Concomitant medication | × | × | <b>*</b> | \&_{\( \) | × | × | × | × | X | X | X | X | × | × | × | × | × |
| Adverse events | | X | K | × | × | × | × | × | X | X X | X | X | × | × | × | X | X |
| eC-SSRS | × | × | × | × | × | × | × | × | × | X | × | × | × | × | × | × | × |
| HADS | × | × | | × | × | × | × | × | X | X | X | × | × | × | × | × | × |
| AsQoL | | X | | | × | × | × | × | F 7 | × | | × | | | × | × | × |
| BASDAI | 9/1/ | × | × | × | × | × | × | × | - 1 | × | | × | | | × | × | × |
| BASFI | S <sub>O</sub> | X | × | × | × | × | × | × | - 1 | X | | X | | | × | X | × |
| SF-36 | , | × | | | × | | × | × | ۲٦ | × | | × | | | × | × | × |
| MOS Short Sleep Scale (12 items) | | × | | | × | | × | × | F 4 | × | | × | | | × | × | × |
| PGADA | | × | × | × | × | × | × | × | 7 4 | × | | × | | | × | × | × |
| Total and nocturnal spinal pain (NRS) | | × | × | × | × | × | × | × | FY | × | | × | | | × | × | × |
| Tuberculosis questionnaire | × | × | | | | | × | | FY | × | | × | | | × | × | × |

Schedule of study assessments Table 5-1:

| Visit** Double-Blind Period (weeks after first dose) (weeks after first dose) Visit** Serie after first dose) (weeks after first dose) (weeks after first dose) Visit** X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Dose-Blind Period (weeks after first do | ts | assessment | Table 5-1: Schedule of study assessments |
|---|---|---|---|---|
| Screen S | 6 7 8 9 10 11 12 13 14 15<br>8 17 16 20 24 28 37 36 40 44 | (S tisit Z) (Secondary) | əuile | |
| igns (BP, pulse, temperature) <sup>d</sup> X X X X X X X X X X X X X | 8 17 16 20 24 28 32 36 40 44 | ,l ya<br>tani)<br>w | Base | /isit <sup>a</sup> |
| igns (BP, pulse, temperature) <sup>d</sup> | 11 01 00 10 01 11 0 | ) | | Veek <sup>a</sup> |
| igns (BP, pulse, temperature) <sup>d</sup> | | | × | leight |
| A | X X X X X X X X | X | | 'ital signs (BP, pulse, temperature) <sup>d</sup> |
| ES ES II | × | × | | ody weight |
| S | 5// | | × | hysical examination <sup>e</sup> |
| III X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | 100 | | | AASES |
| DA X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X | Ç | | ASMI |
| Asample for CRP* X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X | × | | hGADA |
| | X X X | | × | CGf |
| | X | X | | ematology/biochemistry/urinalysis |
| X X X X X X X X X X X X X X X X X X X | X | 10 × | | lood sample for CRP <sup>g</sup> |
| × × × × | X | X | | lood sample for hs-CRP <sup>g</sup> |
| × Xs | XXX | 78. | | regnancy testing <sup>h</sup> |
| (A) | | | × | epatitis B and C testing |
| 0, | | | Z, | IV testing |
| | | × | | ollect blood sample for determination of LA-B27 status |
| Blood sample for bimekizumab plasma X X X X X X X X X X X X X X X X X X X | × × × × × | × | | lood sample for bimekizumab plasma<br>oncentrations <sup>8</sup> |
| Bimekizumab antibody detections X X X X X X X X X X X X X X X X X X X | X X X X | | | imekizumab antibody detection <sup>g</sup> |

Schedule of study assessments Table 5-1:

| OCB<br>Clinical Study Protocol | | | 7 | | | 2 | | | | | | | | | 7 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5-1: Schedule of study assessm | assessm | ents | | | | | | | | | | | | 7.4 | 0/1/5 | 10/10/14 | |
| | gninə<br>01 qu) (1<br>(2 gri | eline<br>, Visit 2)<br>(920b.) | Doi<br>(wee | ıble-F<br>ks aft | Double-Blind Period<br>(weeks after first dose) | Perio<br>st do | ф<br>(9) | | | Dose-Blind Period (weeks after first dose) | Dose-Blind Period | d Per | dose | 7 .0 | | ET | $SFU^b$ |
| ${ m Visit}^{ m a}$ | Sere<br>I sit I | l yr | 3 | 4 | v | 9 | 7 | | 9 1 | 10 11 | 1 12 | 13 | 3 14 | 15 | 16 | | |
| $Week^a$ | л) | <b>a</b> ) | 1 | 2 | 4 | ∞ | 12 1 | 16 2 | 20 2 | 24 2 | 280 32 | 36 | 5 40 | 44 | 48 | | |
| Blood samples for cytokines, complement, and biomarker analysis <sup>g</sup> | | × | × | | × | | × | | 1,00 | XO, | r | | | | × | × | |
| Blood sample for genomic, proteomic/metabolomic analyses <sup>g, i</sup> | | × | × | | × | | × | 10/2 | 40/2 | × | | | | | × | × | |
| Blood samples for genetic/epigenetic analysis <sup>g,i</sup> | | × | × | | ( | To | X C | ), | | × | | | | | | | |
| For participating centers:<br>Blood samples for flow cytometry <sup>g,</sup> | | × | × | | | 0/20. | × | | | × | | | | | × | × | |
| IGRA tuberculosis test <sup>j</sup> | × | | | (). | O. | | | | | | | | | × | | × | × |
| Evaluation for rescue therapy <sup>k</sup> | | C | ()) | 0 | | | , , | × | | × | | × | | | | | |
| Chest x-ray <sup>1</sup> | × | | 1/20 | 2 | | | | | | | | | | | | | |
| Sacroiliac joint x-ray | X <sub>m</sub> | YO' | L. | | | | | | | | | | | | | | |
| Spine and sacroiliac MRI <sup>n</sup> | | × | | | | | × | | | | | | | | × | | |
| Enter IXRS° | × | X | × | × | × | × | × | × | × | X | × | × | × | × | × | × | × |
| Bimekizumah or placeho administration <sup>p, q</sup> | 94 | > | | | > | > | > | > | > | ^ | 4 | > | 7 | * | | | |

AS=ankylosing spondylitis; ASAS=Assessment of SpondyloArthritis International Society; AsQoL=Ankylosing Spondylitis Quality of Life; BASDAI=Bath NRS=numeric rating scale; PGADA=Patient's Global Assessment of Disease Activity; PhGADA=Physician's Global Assessment of Disease, Activity; SF-Ankylosing Spondylitis Disease Activity Index, BASFI=Bath Ankylosing Spondylitis Functional Index; BASMI=Bath Ankylosing Spondylitis Metrology IGRA=interferon gamma release assas; IMP=investigational medicinal product; IMS=International Menopause Society; IXRS= interactive voice or web Index;BP=blood pressure; CRP=C-reactive protein; eC-SSRS=electronic Columbia Suicide Severity Rating Scale; ECG=electrocardiogram; ET=Early response system; MASES=Maastricht Ankylosing Spondylitis Enthesitis Index; MOS=Medical outcomes study; MRI=magnetic resonance imaging; Termination; HADS=Hospital Anxiety and Depression Scale; HIV=human immunodeficiency virus; hs-CRP=high sensitivity C-reactive protein; 36=Short Form-36; SFU=Safety Follow-Up; TB=tuberculosis AS0008

# Table 5-1: Schedule of study assessments

| $\mathbf{SFU}^{\mathbf{b}}$ | | |
|---|---|---|
| ET | | |
| | 16 | 48 |
| 0 | 15 | 44 |
| (986) | 10 11 12 13 14 15 | 4 8 12 16 20 24 28 32 36 40 44 48 |
| nd Period | 13 | 36 |
| lind<br>fter fi | (Z) | 32 |
| Dose-Blind Period<br>(weeks after first dose | 11 | 280 |
| D<br>(wee | 10 | 24 |
| | 9 | 20 |
| | 8 | 91 |
| od<br>ose) | 6 8 2 9 8 | 12 |
| Double-Blind Period<br>weeks after first dose | 9 | 8 |
| Blind<br>fter fi | 5 | 4 |
| uble-<br>eks af | 4 | 2 |
| Do<br>(wed | 3 | 1 |
| eline<br>, Visit 2)<br>( dose) | Bag<br>I ya | a) |
| gnins:<br>ot qu) (1<br>(sysb | 1isi | <b>A</b> ) |
| | Visit <sup>a</sup> | $Week^a$ |

Visit windows of +/-3 days from the first dose at all visits through Week 12 and +/- 4 days for all visits after Week 12 except SFU. The SFU Visit window is -3 and +7 days from last dose.

Safety Follow-Up Visit occurs 20 weeks after the last dose for all subjects who complete the study and do not enter the extension study or who discontinue early, including those withdrawn from study treatment.

Ensure there are no significant changes in medical history that would exclude the subject based on the exclusion criteria.

At Baseline/Day 1 and Week 12, collect pulse and BP prior to drug administration and then at 30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing. All other procedures are done prior to dosing.

<sup>e</sup> Includes evaluation of signs and symptoms of active TB, risk for exposure to TB.

f ECGs will be performed at the study site and read locally.

At dosing visits, all blood samples are taken prior to dosing. Blood samples for binekizumab and anti-bimekizumab anti-bimekizumab anti-bimekizumab antibody detection will be processed as per instructions in the laboratory manual. Both CRP and hs-CRP will be tested. After Screening, both hs-CRP and CRP data will not be sent to the Investigator to protect the blinded nature of the treatment assignments.

potential with infrequent or irregular menstrual cycles and women during menopause. Natural menopause is recognized to have occurred after 12 consecutive A serum pregnancy test will be performed at Screening for all women of childbearing potential. This recommendation also applies to women of childbearing pregnancy test is also required at the Baseline, Week 48, ET, and at SFU visits. A urine pregnancy test will also be performed at any study visit where there has been a delay in menses. This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles. Pregnancy months of amenorrhea, for which there is no other obvious pathological or physiological cause (International Menopause Society [IMS], 2015). A urine test results must be negative prior to administering IMP.

A separate Informed Consent Form will be required for subjects who provide samples for genetic testing. The Informed Consent Form must be signed prior to collecting samples.

It is recommended that Quantiferon TB GOLD test be performed.

Subjects with <10% improvement from Baseline in both PGADA and total and nocturnal spinal pain (ASAS domain response criteria) are eligible for rescue At Weeks 16, 24, and 36 of the Dose-Blind Period, subjects will be evaluated for their response to treatment to determine eligibility for rescue therapy. treatment. Rescue therapy will be at the Investigator's discretion as outlined in Section 5.1.4.

<sup>1</sup> If a subject has had a recent radiograph of the chest within 3 months prior to the Screening Visit, it may be used as the Screening chest x-ray.

reading. If no x-ray is available one must be performed at Screening. If the previous x-ray is more than 1 year old, and central read criteria for randomization "If subjects have a previous x-ray documenting AS meeting eligibility criteria, they are eligible for study entry after reconfirming their eligibility by central are not met, another x-ray may be performed if permitted by local guidelines.

# Schedule of study assessments Table 5-1:

| ∞ ∞ ∣ | i l | | ı | |
|---|---|---|---|---|
| Aar 201<br>AS000 | | $ m SFU^b$ | | |
| AS0008 | | ET | | |
| 1. S. | 0, | | 16 | 48 |
| | 190/1/ | | 15 | 44 |
| | | (əsə | 14 | 40 |
| | | nd Period<br>r first dose | 13 | 36 |
| | | lind <br>ter fi | 11 12 13 | 280 32 36 |
| | | ose-B<br>eks af | 11 | |
| | | Dew) | 10 | 24 |
| | | | 6 | 20 |
| | | | ∞ | 16 |
| | | ose) | 7 | 12 |
| nab | | Double-Blind Period<br>(weeks after first dose) | 9 | 8 |
| Bimekizumab | | Blind<br>fter fi | S | 4 |
| Bime | | uble-<br>eks a | 4 | 7 |
| | | Do<br>(we | 3 | 1 |
| | ents | Baseline<br>(Day 1, Visit 2)<br>(first dose) | | |
| | assessm | gning<br>ot qu) (1<br>(8ys) | isi | ۸) |
| rotocol | Table 5–1: Schedule of study assessments | | | |
| UCB<br>Clinical Study Protocol | Table 5–1: | | $Visit^a$ | Week <sup>a</sup> |

of eligibility based on screening assessments for the study and before the first bimekizumab injection. Magnetic resonance imaging at Week 12 and Week 48 at Week 12 and Week 48 will be performed for those subjects who were MRI-positive at Baseline. The Baseline MRI should be performed after confirmation An MRI of the spine and sacroiliac joints will be performed in a substudy with approximately 20 subjects perfreatment arm at Baseline. A central reader will assess Baseline MRIs to identify MRI-positive subjects as per the ASAS-Outcome Measures in Rheumatology Clinical Trials (OMERACT) criteria. An MRI should be performed as close to the Week12/Week 48 Visit as possible. For logistical reasons, it may not be possible to schedule the MRIs at the actual visit date and an additional visit for the MRI may be required.

IXRS is used to register the Subject at Screening, randomize the Subject at Baseline/Day 1, rerandomize the Subject at Week 12 (Subject in the placebo,

bimekizumab 16mg, and bimekizumab 64mg treatment groups), and to register all visits.

P The minimum time between doese during the Double-Ellind Period double and the prodest than 31 days and during the Dose-Blind Period should be no less than 24 days and no more than 32 days.

4 At Week 12, the Dose-Blind Period dosing will start, as detailed in Section 31.34

At Week 12, the Dose-Blind Period dosing will start, as detailed in Section 31.34

At Week 12, the Dose-Blind Period dosing will be proved the Section 31.34

At Week

5.3

# Schematic diagram

The study schematic diagram for AS0008 is presented in Figure 5–1.

Figure 5-1: Schematic diagram



ASAS=Assessment of SpondyloArthritis International Society; DMARD=disease-modifying antirheumatic drug; NSAID=nonsteroidal anti-inflammatory drug; PGADA=Patient's Global Assessment of Disease Activity; Q4W=every 4 weeks; SFU=Safety Follow-Up

Subjects with <10% improvement from Baseline in both PGADA and total and nocturnal spinal pain (ASAS domain response criteria) are eligible for rescue treatment. Rescue therapy will be at the Investigator's discretion as outlined in Section 5.1.4.

This document cannot be

<sup>&</sup>lt;sup>a</sup> After 12 weeks of double-blind treatment, subjects randomized to placebo, bimekizumab 16mg Q4W, or bimekizumab 64mg Q4W doses will be rerandomized 1:1 to receive either bimekizumab 160mg Q4W or bimekizumab 320mg Q4W. Subjects randomized to bimekizumab 160mg Q4W or 320mg Q4W will continue to receive their originally randomized dose (Section 5.1.3).

<sup>&</sup>lt;sup>b</sup> At Weeks 16, 24, and 36 of the Dose-Blind Period, subjects will be evaluated for their response to treatment to determine eligibility for rescue therapy.

09 Mar 2018

AS0008

#### 5.4 Rationale for study design and selection of dose

The following doses of bimekizumab are proposed in the Phase 2b study: 16mg, 64mg, 160mg, and 320mg administered sc Q4W. The proposed dose range has been selected based on a dose

Doses greater than 320mg have been previously studied in the development of bimekizumab. In the single ascending dose study UP0008, a single dose of bimekizumab 640mg was tested. In the multiple dose study PA0007, a bimekizumab 560mg loading. 320mg doses every 3 weeks was tested. At exposure levels achieved at these doses, the compound had no significant safety concerns. In the previous clinical studies, bimekizumab was administered iv and the current study proposes to administer the compound sc. Due to lower bioavailability, bimekizumab exposure is expected to be lower with sc administration compared to after iv administration, therefore, the dose regimens are expected to be safe?

Simulations were performed using the developed model to predict the dose response of ASAS40 at Week 12, which indicated that increasing doses above bimekizumab 320mg may not provide additional benefit in terms of efficacy. Therefore, bimekizumab 320mg has been selected as the maximum dose in the current study. Three dose levels below bimekizumab 320mg were selected to characterize the dose-exposure response curve at the end of current study. The lowest dose level of bimekizumab 16mg Q4W was selected because this dose is expected to provide an ASAS40 response rate close to placebo, while still delivering some benefit to patients. The bimekizumab 64mg and 160mg O4W doses were selected in order to precisely characterize the dose-exposure response curves. The proposed doses will provide adequate information to study the dose-exposure response of bimekizumab in AS. This information will be used to determine the right dose and dosage regimen for future studies of bimekizumab in this indication.

#### SELECTION AND WITHDRAWAL OF SUBJECTS 6

#### Inclusion criteria 6.1

To be eligible to participate in this study, all of the following criteria must be met:

- 1. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent Form is signed and dated by the subject or legal representative.
- 2. Subject or legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, or medication intake according to the judgment of the Investigator.
- 3. Subject is male or female and at least 18 years of age. This document can

- 4. **Female** subjects must be postmenopausal (at least 1 year; to be confirmed hormonally as part of the screening process, if less than 2 years since last menstrual period), permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception up till 20 weeks after last administration of IMP, and have a negative pregnancy test at Visit 1 (Screening) and immediately prior to first dose. The following methods are considered highly effective when used consistently and correctly.
  - combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
  - progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  - intrauterine device (IUD)
  - intrauterine hormone-releasing system (IUS)
  - bilateral tubal occlusion
  - vasectomized partner
  - sexual abstinence if it is in accordance with a subject's preferred and common lifestyle. Subjects who use abstinence as a form of birth control must agree to abstain from heterosexual intercourse until 20 weeks after the last dose of IMP. Study personnel must confirm the continued use of abstinence is still in accordance with the subject's lifestyle at regular intervals during the study.

Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up till 20 weeks after the last administration of IMP (anticipated 5 half-lives).

- 5. Subject has active AS, determined by documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984) (see Table 19–1), including symptoms for ≥3 months and age of onset <45 years.
- 6. Subject has moderate to severe active disease as defined by each of the following:
  - BASDAI score ≥4
  - Spinal pain ≥4 on a 0 to 10 NRS (from BASDAI item 2)
- 7. Subjects must have at least 1 of the following:
  - inadequate response to NSAID therapy

intolerance to administration of at least 1 NSAID

- contraindication(s) to NSAID therapy

Inadequate response to an NSAID is defined as lack of response for at least 4 weeks of continuous NSAID therapy at the highest tolerated dose of the administered NSAID or the lack of response to treatment with at least 2 NSAIDs at the maximum tolerated dose for at least 4 weeks total duration.
- 8. Subjects who are regularly taking NSAIDs/COX-2 inhibitors as part of their AS therapy are required to be on a stable dose for at least 14 days before Baseline and should remain on a stable dose up to Week 16.
- 10. Subjects taking MTX (≤25mg/week) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomizated by the least 12 weeks prior to Baseline, which is the least 12 weeks by the least 12 weeks before randomizated by the least 12 weeks 12 weeks by the least 12 weeks 12 weeks 12 weeks 12 weeks folic acid supplementation.
- 11. Subjects taking sulfasalazine (up to 3g/day) or hydroxychloroquine (up to 400mg per day total) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomization. Dose and dosing schedule should remain stable up to Week 16.
- 12. Subjects may be TNF inhibitor-naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:
  - experienced an inadequate response to previous treatment given for at least 12 weeks
  - been intolerant to administration (eg, had a side effect/AE that led to discontinuation)
  - lost access to TNF inhibitor for other reasons

### **Exclusion criteria** 6.2

Subjects are not permitted to enroll in the study if any of the following criteria are met:

- 1. Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 20 weeks following last dose of IMP. Male subjects who are planning a partner pregnancy during the study or within 20 weeks following the last dose.
- 2. Subjects previously participating in a bimekizumab clinical study and receiving at least 1 dose of IMP.
- 3. Subjects participating in another study of a medication or a medical device under investigation within the last 12 weeks or at least 5 half-lives whichever is greater.
- 4. Subjects with a known hypersensitivity to any excipients of bimekizumab.
- 5. Subjects with a total ankylosis of the spine, or a diagnosis of any other inflammatory arthritis eg, RA, sarcoidosis, systemic lupus erythematosus, or reactive arthritis.
- 6. Subjects with use of any medication listed in Table 7–1 meeting the exclusionary criteria for the specific medication(s) including wash-out described in the table.
- Subject has any current sign or symptom that may indicate an active infection (except for the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of Baseline.

- 8. Subjects with a history of chronic or recurrent infections, or a serious or life-threatening infection within the 6 months prior to the Baseline Visit (including herpes zoster). Subjects with a high risk of infection in the Investigator's opinion (eg, subjects with leg ulcers, 9. Subjects with concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection. Subjects who have evidence of, or tested positive for hepatitis P or hepatitis C are excluded.

  A positive test for the subjects who have evidence of the patitic P or hepatitis P or hepatit

A positive test for the hepatitis B virus (HBV) is defined as:

- positive for hepatitis B surface antigen (HbsAg+); or,
- positive for anti-hepatitis B core antibody (HbcAb+)

A positive test for the hepatitis C virus (HCV) is defined as:

- positive for hepatitis C antibody (anti-HCV Ab), and
- positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction)
- 10. Subjects with known history of or current clinically active infection with Histoplasma, Coccidioides, Paracoccidioides, Pneumocystis, nontuberculous mycobacteria (NTMB), Blastomyces, or Aspergillus or current active Candidiasis (local or systemic).
- 11. Subjects receiving any live (includes attenuated) vaccination within the 8 weeks prior to Baseline (eg. inactivated influenza and pheumococcal vaccines are allowed but nasal influenza vaccination is not permitted). Live vaccines are not allowed during the study or for 20 weeks after the last dose of IMP.

Live vaccines include, but are not limited to the following:

- Anthrax vaccine
- Intranasal influenza vaccine
- Measles-mumps-rubella (MMR) vaccine
- Polio live orabvaccine (OPV)
- Smallpox vaccine
- Tuberculosis BCG vaccine
- Typhoid live oral vaccine

Varicella vaccine

- Yellow fever vaccine
- 12. Subjects receiving Bacillus Calmette-Guerin (BCG) vaccinations within 1 year prior to IMP administration.
- 13. Subjects with a history of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease.

- 14. Subjects with primary immunosuppressive conditions, including subjects who are taking immunosuppressive therapy following organ transplants.
- 15. Subjects with known TB infection, at high risk of acquiring TB infection, with latent TB infection (LTBI)\* or current or history of NTMB infection (refer to Section 12.6.5 for details on determining full TB exclusion criteria).
  \*Subjects with LTBI may enter the study only after they have completed at least 8 weeks of appropriate prophylactic therapy and thereafter, will continue and complete the entire regimen.
- 16. Subjects who have had a splenectomy.
- 17. Subjects with concurrent malignancy or a history of malignancy (including surgically resected uterine/cervical carcinoma-in-situ) during the past 5 years will be excluded, with the following exceptions that may be included:
  - a)  $\leq 3$  excised or ablated basal cell carcinomas of the skin
  - b) One squamous cell carcinoma of the skin (stage T1 maximum) successfully excised, or ablated only (other treatments, ie, chemotherapy, do not apply), with no signs of recurrence or metastases for more than 2 years prior to Screening
  - c) Actinic keratosis (-es)
  - d) Squamous cell carcinoma-in-situ of the skin successfully excised, or ablated, more than 6 months prior to Screening
- 18. Subjects having had major surgery (including joint surgery) within the 6 months prior to Screening, or planned surgery within 6 months after entering the study.
- 19. Subjects with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac (eg, congestive heart failure New York Heart Association [NYHA] Grade 3 and 4), gastrointestinal (GI) (note: subjects with active peptic ulcer disease are excluded; subjects with a history of peptic ulcer disease are allowed), or neurological disease.
- 20. Subjects with a history of uncompensated heart failure, fluid overload, or myocardial infarction, or evidence of new-onset ischemic heart disease or in the opinion of the Investigator other serious cardiac disease, within 12 weeks prior to Baseline.
- 21. Subjects with clinically significant laboratory abnormalities (eg, glomerular filtration rate [GFR] <60 mL/min/1.73m<sup>2</sup>, neutropenia <1.5x10<sup>9</sup>/L, hemoglobin <8.5g/dL, lymphocytes <1.0 x10<sup>9</sup>/L, platelets <100x10<sup>9</sup>/L). Individual screening tests, for which the results are in error, borderline, or indeterminate for inclusion in the study, can be repeated once for confirmation during the Screening Period if they are within 25% of the exclusion limit. Upon retesting, subjects whose results remain outside this threshold should not be randomized.

- 22. Subject has >2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase\* (ALP), or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%).
  - \*An isolated elevation between 2xULN and <3xULN of ALP is acceptable in the absence of an identified exclusionary medical condition.

Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit may be repeated once for confirmation during the Screening Period. Upon retesting, subjects whose ALT, AST, or ALP remain above the thresholds defined above, should not be randomized.

For randomized subjects with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin, a baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report Form (eCRF).

If subject has >ULN ALT, AST, or ALP that does not meet the exclusion limit at screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the Medical Monitor.

- 23. Subjects with any other condition which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study.
- 24. Subjects with erythrodermic, guttate, pustular form of PSO or drug-induced PSO.
- 25. Subjects with a diagnosis of inflammatory conditions other than AS, including but not limited to rheumatoid arthritis or systemic lupus erythematosus. Subjects with a diagnosis of Crohn's disease or ulcerative colitis (whether primary or as an extra-articular manifestation of AS) are allowed provided they have no active and/or symptomatic disease at Screening and Baseline.
- 26. Subjects with fibromyalgia or osteoarthritis symptoms that in the Investigator's judgement would have potential to interfere with efficacy assessments
- 27. Subject has a history of chronic alcohol or drug abuse within the previous year.
- 28. Subject has 12-lead ECG with changes considered to be clinically significant upon medical review by the Investigator or designee.
- 29. Subject has presence of significant uncontrolled neuropsychiatric disorder, active suicidal ideation, or positive suicide behavior using the "Baseline" version of the electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) and the Hospital Anxiety and Depression Scale (HADS) with either of the following criteria:
  - Subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the eC-SSRS at screening.
  - Any subject who develops a HADS-D Depression Score >10 or Anxiety (HADS-A) score ≥15.

- 30. Subject is Investigator site personnel directly affiliated with this study and/or immediate families of Investigator site personnel. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
- vithdrawal criteria

  Subjects are free to withdraw from the study at any time, without prejudice to their continued in the care.

  Subjects should be withdrawn from the study if any of the following.

- 2. There is confirmation of a pregnancy during the study, as evidenced by a positive pregnancy
- 3. The Sponsor or a regulatory agency requests withdrawal of the subject.

# Subjects withdrawn from study treatment:

Subjects should be withdrawn from all study treatment if any of the following events occur:

- 4. Subject develops an illness that would interfere with his/her continued participation.
- 5. Subject considered as having either a suspected new LTBI or who develops active TB or NTMB infection during the study (including but not limited to, conversion demonstrated by interferon-gamma release assay [IGRA] or other diagnostic means) must be immediately discontinued from IMP, and an unscheduled visit must be conducted as soon as possible, but not later than the next regular visit.

The subject must be permanently withdrawn if further examinations result in a diagnosis of active TB, or if the subject is diagnosed with LTBI with no initiation of prophylactic treatment, prematurely discontinues prophylactic treatment, or, in the opinion of the Investigator or Sponsor, is noncompliant with prophylactic TB therapy.

Confirmed active TB is a serious adverse event (SAE) and must be captured on an SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements. As with all SAEs, periodic follow-up reports should be completed as per protocol requirements until such time as the TB infection resolves. Additional information on TB policies are provided in Section 12.6.5.

- 6. Subject is noncompliant with the study procedures or medications which may present a risk
- that may present a risk to the safety of the subject in the opinion of the Investigator and the Medical Monitor. This includes subjects who start a biologic other than bimekizumah as described in Section 5.1.4.

- 8. Subject develops laboratory abnormalities (with or without clinical symptoms) of ALT or AST as defined in Section 6.3.1; neutropenia <0.5x10<sup>9</sup>/L; lymphopenia <0.5x10<sup>9</sup>/L. Any laboratory value or change judged to be clinically significant by the Investigator should prompt consideration of whether the subject should continue on IMP. For clarification, laboratory values that are markedly abnormal as per Table 19–2 and Table 19–3 will be flagged to the Investigator and to the medical monitor but do not trigger mandatory withdrawal unless listed above (Refer to Section 6.3.1 for withdrawal criteria in relation to potential drug-induced liver injury [PDILI].)
- 9. Subject has active suicidal ideation as indicated by a positive response ("Yes") to Questions 4 or 5 or to the suicidal behavior questions of the "Since Last Visit" version of the self-rated eC-SSRS. The subject should be referred immediately to a Mental Healthcare Professional and must be withdrawn from the study.
- 10. Subjects with a HADS-D score ≥15 must be withdrawn. Any subject who develops a HADS-D score of >10 during the study should be referred immediately to a Mental Healthcare Professional for further evaluation and potential withdrawal by the Investigator.
- 11. Subjects with newly diagnosed IBD or with IBD flares during the study must:
  - Be referred, as appropriate, to a health care professional treating IBD, such as a gastroenterologist
  - Discontinue IMP and be followed-up until resolution of active IBD symptoms

If IBD flares increase in severity or frequency during the study, the Investigator should use clinical judgment in deciding whether the subject should continue in the study and contact the Medical Monitor and UCB study physician to confirm the subject's suitability for continued participation in the study.

In an attempt to prevent missing data during the study, efforts will be made to collect data from subjects that withdraw early from the study (NRC, 2010). If a subject withdraws from study treatment for any of the above criteria (#4 through #10) prior to Week 12, they will be asked to return for the study assessments 12 weeks after the first dose (ie, Week 12 Visit) and for the SFU Visit (20 weeks after last dose administration). These data will be used in a sensitivity analysis which is described in Section 15.7. If any of these criteria occur after Week 12, subjects will complete an Early Termination (ET) Visit and the SFU Visit. All subjects who withdraw from the study due to an AE must be followed until resolution of the event or until the event is considered stable. All subjects who withdraw from the study due to development of a laboratory abnormality specified in Criterion #8 must be closely monitored, with additional monitoring of hepatic markers every week or every 2 weeks until resolution of the event, the event is considered stable, or they have reached the end of the SFU Period for those who at any time have an ALT and/or AST >5X but <8X ULN.

Investigators should attempt to obtain information on subjects in the case of withdrawal or discontinuation. For subjects considered as lost to follow-up, the Investigator should make an effort (at least 1 phone call and 1 written message to the subject), and document his/her effort (date and summary of the phone call and copy of the written message in the source documents), to complete the final evaluation. All results of these evaluations and observations, together with a narrative description of the reason(s) for removing the subject, must be recorded in the source documents. The eCRF must document the primary reason for withdrawal or discontinuation.

Investigators should contact the Medical Monitor, whenever possible, to discuss the withdrawal of a subject in advance.

#### 6.3.1 Potential drug-induced liver injury IMP discontinuation criteria

tensions or variations thereof. Subjects with potential drug-induced liver injury (PDILI) must be assessed to determine if IMP must be discontinued. In addition, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued.

The PDILI criteria below require immediate and permanent discontinuation of IMP:

- Subjects with either of the following:
  - ALT or AST >5xULN
  - ALT or AST  $\geq 3xULN$  and coexisting total bilirubin  $\geq 2xULN$
- Subjects with ALT or AST ≥3xULN who exhibit temporally associated symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, right upper quadrant pain or tenderness. Hypersensitivity symptoms include fever (without clear alternative cause), rash, or eosinophilia (ie, >5%).

The PDILI criterion below allows for subjects to continue on IMP at the discretion of the investigator.

Subjects with ALT or AST ≥3xULN (and ≥2x-Baseline) and <5xULN, total bilirubin <2xULN, and no eosinophilia (ie, ≤5%), with no fever, rash, or symptoms of hepatitis (eg, fatigue, nausea, vomiting, right upper quadrant pain or tenderness).

Evaluation of PDILI must be initiated as described in Section 12.5.1. If subjects are unable to comply with the applicable monitoring schedule, IMP must be discontinued immediately.

Investigators should attempt to obtain information on subjects in the case of IMP discontinuation to complete the final evaluation. Subjects with PDILI should not be withdrawn from the study until investigation and monitoring are complete. All results of these evaluations and observations, as well as the reason(s) for IMP discontinuation and subject withdrawal (if applicable), must be recorded in the source documents. The eCRF must document the primary reason for IMP discontinuation.

### STUDY TREATMENTS 7

## Description of investigational medicinal products 7.1

The IMPs used in this study are bimekizumab and placebo.

Bimekizumab will be supplied as a clear to opalescent, colorless to slightly brown, sterile, preservative-free solution in 2mL Type I, colorless glass vials (1.0mL extractable volume) closed with a rubber stopper and sealed with an aluminum cap overseal.

Placebo will be supplied as 0.9% sodium chloride aqueous solution (physiological saline, preservative free) of pharmacopoeia (United States Pharmacopoeia/European Pharmacopoeia) quality appropriate for injection.

09 Mar 2018 AS0008

Further details of the IMPs and their specifications are provided in the Investigational Medicinal Product Handling Manual.

# 7.2 Treatments to be administered

The IMP is to be administered in the clinic by study site staff as 2 sc injections. Suitable areas for sc injections are the lateral abdominal wall and upper outer thigh. During each dosing visit, each of the 2 injections should be administered at a separate injection site. Injection sites should be rotated and injections should not be given into areas where the skin is tender, bruised, red or hard.

The IMP (bimekizumab and placebo) will be administered at the times indicated in Table 5–1. The minimum time between doses during the Double-Blind Period should be no less than 25 days and no more than 31 days and during the Dose-Blind Period should be no less than 24 days and no more than 32 days.

An IMP Handling Manual will be provided to each site containing instructions regarding drug preparation and dosing.

# 7.3 Packaging

Bimekizumab and placebo will be manufactured, packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. They will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

# 7.4 Labeling

Clinical drug supplies will be labeled in accordance with the current International Council for Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and Good Manufacturing Practice and will include any locally required statements. If necessary, labels will be translated into the local language.

# 7.5 Handling and storage requirements

Investigational Medicinal Product must be stored under refrigerated conditions (2°C to 8°C) protected from light. The IMP must not be frozen.

The Investigator (or designee) is responsible for the safe and proper storage of IMP at the site. Investigational medicinal product stored by the Investigator is to be kept in a secured area with limited access.

Appropriate storage conditions must be ensured either by controlled room temperature or by completion of a temperature log in accordance with local requirements on a regular basis (eg, once a week), showing minimum and maximum temperatures reached over the time interval.

In case an out-of-range temperature is noted, it must be immediately communicated to the Clinical Project Manager (CPM) (or designee) before further use of the IMP.

Investigational Medicinal Product will be shipped to the study sites in temperature controlled containers. Out-of-range shipping or storage conditions must be brought to the attention of the Sponsor or designee, immediately. Authorization to use any out-of-range IMP must be documented and received prior to dispensing or administering the IMP at the study site.


# 7.6 Drug accountability

A Drug Accountability Form will be used to record IMP dispensing and return information on a by-subject basis and will serve as source documentation during the course of the study. Details of any IMP lost (due to breakage or wastage), not used, disposed of at the study site, or returned to the Sponsor or designee must also be recorded on the appropriate forms. All supplies and pharmacy documentation must be made available throughout the study for UCB (or designee) to review.

In order to maintain the blind, all IMP documentation (eg, shipping receipts, drug accountability logs, and interactive voice or web response system [IXRS] randomization materials) must be maintained and accessed by unblinded, trained site personnel only. Designated, unblinded site personnel must be appropriately trained and licensed (per country guidelines) to administer injections.

The packaging identifies each kit by a unique number that does not correlate to the contents and therefore, does not unblind study site staff. Unblinded study staff will be responsible for preparation (breaking tamper proof sticker on kit, etc) of the clinical trial material, including recording the administration information on source document.

The Investigator (or designee) is responsible for retaining all used, unused, and partially used containers of IMP until returned or destroyed.

The Investigator may assign some of the Investigator's duties for drug accountability at the study site to an appropriate pharmacist/designee.

The Investigator must ensure that the IMP is used only in accordance with the protocol.

Periodically, and/or after completion of the clinical phase of the study, all used (including empty containers) and unused IMP containers must be reconciled and returned to UCB (or designee), preferably in their original package. Onsite destruction of used kits only may be allowed with prior approval from the Sponsor or designee after reconciliation. Investigational medicinal product intended for the study cannot be used for any other purpose than that described in this protocol.

# 7.7 Procedures for monitoring subject compliance

During the Double-Blind and Dose-Blind Periods, IMP will be administered in the clinic and compliance will be determined at the visit by study personnel. Drug accountability must be recorded on the Drug Accountability Form.

# 7.8 Concomitant medication(s)/treatment(s)

All concomitant medications, including over-the-counter products, herbal, traditional remedies, vitamin/mineral supplements, other dietary supplements, "nutraceuticals," and hormones must be recorded in the subject's source documentation (eg, clinical chart) and on the eCRF. This record should include the name of the drug, the dose, the route and date(s) of administration, and the indication for use.

# 7.8.1 Permitted concomitant treatments (medications and therapies)

The following AS medications/treatments are allowed during this study from Baseline onward, with the following restrictions (if any):

Nonsteroidal anti-inflammatory drugs and/or joint injections as outlined below. For subjects taking NSAID/COX-2 inhibitors at Baseline or at Weeks 16, 24, or 36, a change can be made to a different NSAID/COX-2 inhibitor. Changes from an NSAID to a COX-2 inhibitor or from a COX-2 inhibitor to an NSAID are permitted up to the maximum approved or tolerated dose whichever is lower. Only 1 NSAID/COX-2 inhibitor may be taken at a given time.

- For subjects not taking NSAID/COX-2 inhibitors at Baseline, Weeks 16, 24, or 36, either can be initiated, up to the maximum approved or tolerated dose, whichever is lower. Only 1 NSAID/COX-2 inhibitor may be taken at a given time.
- After the NSAID/COX-2 regimen has been optimized, SI joint injection is permitted, either unilaterally or bilaterally, performed by a qualified physician.
- If the subject does not achieve sufficient response to the above options and/or the Investigator feels that a biologic other than bimekizumab is warranted, the subject must discontinue from study treatment (bimekizumab) and follow the withdrawal criteria and follow up as outlined in Section 6.3.

A decrease in dose or dosing frequency of any agent is permitted for reasons of intolerance/AEs/side effects at any time.

Subjects may be withdrawn from the study or from study medication at any time and continue treatment per the Investigator's discretion, as described in the Withdrawal Section 6.3.

# 7.8.2 Prohibited concomitant treatments (medications and therapies)

Medications listed in Table 7–1 are prohibited or restricted as follows:

Table 7–1: Prohibited or restricted medications and required wash-out periods prior to Baseline

| Drug class | Dose | Exclusion criteria |
|---|---|---|
| Analgesics, including opioid analgesics (acetaminophen/paracetamol, etc) | Any dose | Any ad hoc use in the 24 hours prior to any study visit. |
| JS . | | Stable doses of analgesics permitted. |
| NSAIDs/COX-2 inhibitors | Any dose regimen | Any change in dose/dose regimen in the 14 days prior to the Baseline Visit |
| Oral corticosteroids | Any dose regimen | Any change in dose/dose regimen in the 14 days prior to the Baseline Visit |
| Intramuscular (im)/intravenous (iv)/<br>intra-articular (ia) corticosteroids/bursal<br>corticosteroids | Any dose | Use in the 28 days prior to the Baseline Visit. |
| Intra-articular hyaluronic acid | Any dose | Any use in the 6 months prior to the Baseline Visit. |


Table 7–1: Prohibited or restricted medications and required wash-out periods prior to Baseline

| Drug class | Dose | Exclusion criteria |
|---|---|---|
| DMARDs: -azathioprine -cyclosporine, -cyclophosphamide, -mycophenolic acid, -mycophenylate mofetil -any other small molecule DMARDs (eg tofacitinib, apremilast) | Any dose | Use within 12 weeks prior to the Baseline Visit. |
| MTX | Any dose regimen | Use within 12 weeks prior to the Baseline Visit unless Inclusion Criterion #10 is met |
| SSZ | Any dose | Use within 12 weeks prior to the Baseline<br>Visit unless Inclusion Criterion #11 is met |
| HCQ | Any dose | Use within 12 weeks prior to the Baseline<br>Visit unless Inclusion Criterion #11 is met |
| DMARDs:<br>-leflunomide | Any dose Any dose Any dose Any dose | Use in the 6 months prior to the Baseline Visit unless a cholestyramine washout has been performed; in which case, use up to 28 days prior to the Baseline Visit is acceptable. |
| TNF inhibitors -infliximab (IFX) -adalimumab (ADA) -etanercept (ETN) -golimumab (GOL) | Any dose | For IFX, ADA, GOL, and CZP, any use within the 12 weeks prior to the Baseline Visit For ETN, use within the 28 days prior to |
| -certolizumab pegol (CZP) | Rain | the Baseline Visit. This applies to biosimilar versions of any TNF inhibitors. |
| Any non-TNF biologic medications | Any dose | Any exposure history. |

ADA=adalimumab; COX-2=cyclooxygenase 2; CZP=certolizumab pegol; DMARD=disease modifying antirheumatic drug; ETN=etanercept; GOL=golimumab; HCQ=hydroxychloroquine; IFX=infliximab; ia=intra-articular; im=intramuscular; iv=intravenous; MTX=methotrexate; NSAID=nonsteroidal anti-inflammatory drug; sc=subcutaneous; SSZ=sulfasalazine; TNF=tumor necrosis factor

Subjects who are receiving an established anti-depressant regimen should be on a stable dose of anti-depressant for 12 weeks prior to Baseline.

# 7.9 Blinding

Due to differences in presentation of the IMPs (bimekizumab and placebo), special precautions will be taken to ensure study blinding and study sites will have blinded and unblinded personnel.

Bimekizumab and placebo injections will be prepared and administered at the investigational sites by unblinded, dedicated study personnel according to Table 7–2. The unblinded personnel will not be involved in the study in any way other than assuring the medication is taken from the correct kit and prepared according to the pharmacy manual instructions, and administering the

drug to the subjects. Preparation will be made from either vials (bimekizumab) or Ampoule (placebo) and will be in identical syringe and needle for all arms of the study. Provisions will be made to ensure that volume of injection is not revealed to the subject. The number of injections will be kept identical for all patients by adding placebo injection when the bimekizumab dose requires only 1 injection.

Table 7–2: Preparation of placebo and bimekizumab injections

| Treatment Arm | Number/volume Placebo injections | Number/volume bimekizumab injections |
|---|---|---|
| Placebo | 2 x 1.0mL | 0 |
| Bimekizumab 16mg | 1 x 0.1mL | 1 x 0.1mL |
| Bimekizumab 64mg | 1 x 0.4mL | 1 x 0.4mL |
| Bimekizumab 160mg | 1 x 1.0mL | 1 x 1.0mL |
| Bimekizumab 320mg | 0 | 2 x 1.0mL |

Study sites will be required to have a written blinding plan in place, signed by the Principal Investigator, which will detail the site's steps for ensuring that the double-blind nature of the study is maintained.

During the study the Sponsor will provide blinded and unblinded site monitors for the purposes of verifying safety, efficacy, and drug administration and documentation records. Blinded study monitors and study site personnel, blinded to treatment assignment, will not discuss or have access to any drug-related information.

Bioanalytical staff analyzing blood samples for bimekizumab and anti-bimekizumab antibody detection will be unblinded.

Further details are provided in the study manuals and site blinding plan.

# 7.9.1 Procedures for maintaining and breaking the treatment blind

# 7.9.1.1 Maintenance of study treatment blind

All subject treatment details (bimekizumab or placebo) will be allocated and maintained by the IXRS.

# 7.9.1.2 Breaking the treatment blind in an emergency situation

The integrity of this clinical study must be maintained by observing the treatment blind. In the event of an emergency for which the appropriate treatment for a subject cannot be made without knowing the treatment assignment, it will be possible to determine to which treatment arm and dose the subject has been allocated by contacting the IXRS. All sites will be provided with details of how to contact the system for code breaking at the start of the study. The Medical Monitor or equivalent should be consulted prior to unblinding, whenever possible.

The CPM will be informed immediately via the IXRS when a code is broken, but will remain blinded to specific treatment information. Any unblinding of the IMP performed by the Investigator must be recorded in the source documents and on the Study Termination eCRF page.

# 7.10 Randomization and numbering of subjects

An IXRS will be used for assigning eligible subjects to a treatment regimen based on a predetermined production randomization and/or packaging schedule provided by the Sponsor. The randomization schedule will be produced by an independent biostatistician with the Contract Research Organization (CRO) who is otherwise not involved in this study. Subject treatment assignment will be stratified by region and prior TNF inhibitor exposure (yes/no). The IXRS will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Enrollment of TNF inhibitor experienced subjects will be limited to 30% of the total study population.

At Screening, each subject will be assigned a 5-digit number that serves as the subject identifier throughout the study. The subject number will be required in all communication between the Investigator or designee and the IXRS regarding a particular subject.

At the Baseline Visit (Day 1), a subject will be randomized into the study. The Investigator or designee will use the IXRS for randomization. The IXRS will automatically inform the Investigator or designee of the subject's ID number. The IXRS will allocate kit numbers to the subject based on the subject number during the course of the study.

Subject numbers and kit numbers will be tracked via the IXRS.

# 8 STUDY PROCEDURES BY VISIT

The Schedule of Study Assessments (Table 5–1) provides a general overview of study assessments. A list of procedures to be completed at each visit is described below.

Visit windows are +/-3 days from Baseline (Day1, first dose of IMP) at all visits through the Week 12 Visit and +/-4 days for all visits after Week 12 except the SFU Visit. For the SFU Visit (20 weeks after the last dose), the visit should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date (-3 days/+7 days). The minimum of time between doses should be no less than 24 days and no more than 32 days. Changes to the dosing schedule outside of the allowed windows must be discussed with the Medical Monitor and may result in subject withdrawal.

# 8.1 Screening (Visit 1)

The Screening Period will last up to 28 days.

Prior to any study specific activities, subjects will be asked to read, sign, and date an Informed Consent Form (ICF) that has been approved by the Sponsor and an IEC/IRB, and that complies with regulatory requirements. Subjects will be given adequate time to consider any information concerning the study given to them by the Investigator or designee. As part of the informed consent procedure, subjects will be given the opportunity to ask the Investigator any questions regarding potential risks and benefits of participation in the study.

Subjects will also be given the option to participate in the genomic, genetic/epigenetic, and proteomic substudy. Subjects who decide to participate in the substudy will need to complete a separate ICF following the same procedure and given the same considerations as the main ICF. Their willingness to participate in the substudy will be independent from their consent to participate in the main study.

Subjects who initially fail to meet selected eligibility criteria (including but not limited to OPY application and any extensions of variations thereof. documented completion of LTBI prophylactic therapy) or for whom eligibility assessments could not be completed as planned may be rescreened once after discussion with the Medical Monitor.

The following procedures or assessments will be performed at the Screening Visit:

- Obtain written informed consent for main study.
- Collect demographic data.
- Collect AS history.
- Collect significant past medical history and concomitant diseases.
- Assess inclusion and no exclusion criteria.
- Record prior medications.
- Record concomitant medications.
- eC-SSRS
- HADS
- Administer the tuberculosis questionnaire.
- Measure height.
- Measure temperature, pulse, and blood pressure
- Measure weight.

  Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB.
- Perform an ECG.
- Collect samples for hematology/biochemistry/urinalysis.
- Perform a serum pregnancy test if the subject is a woman of childbearing potential. This requirement also applies to women of childbearing potential with infrequent or irregular menstrual cycles and women during menopause. Natural menopause is recognized to have occurred after 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause (International Menopause Society, 2015).
- Collect samples for Hepatitis B and C tests.
- Collect samples for an HIV test.
- Perform an IGRA tuberculosis test.

Obtain a chest radiograph, unless one has been obtained 3 months prior to the Screening Visit.

- Obtain a radiograph of the SI joint. Note: If subject has a previous x-ray documenting AS meeting eligibility criteria, he/she is eligible for study entry after reconfirming his/her eligibility by central reading. If no x-ray is available one must be performed at Screening. If

The MRI (done at selected sites) can be performed prior to the Baseline (Day 1, first dose of IMP, Visit 2) if eligibility is confirmed based on screening assessments, and before the first of IMP.

8.2 Baseline (Day 1, first dose of IMP).

The following procedures of assessments will be completed prior to administration of IMP:

- Review significant past medical history and concomitant diseases to ensure there are no significant changes in medical history that would exclude the subject based on the exclusion criteria.
- Confirm that the subject meets all inclusion and no exclusion criteria.
- Record concomitant medications.
- Record AEs.
- eC-SSRS
- **HADS**
- Administer the AsQoL.
- Determine the BASDAI.
- Determine the BASFI.
- Administer the SF-36.
- Administer the MOS Short Sleep Scale.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.
- Administer the tuberculosis questionnaire.
- Measure temperature, pulse, and BP.
- Measure weight.

Determine the MASES.

- Determine the BASMI.
- Administer the PhGADA.
- Collect samples for hematology/biochemistry/urinalysis.
- Collect blood sample for CRP.

- Collect blood sample for hs-CRP.
- Perform a urine pregnancy test if the subject is a woman of childbearing. This requirement The is no other obvious pathological or independent of HLA-B27 status.

  Collect blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.

  Collect blood samples for cytokines, complement, and biomarker analysis.

  If subject provides consent (separate from 4).

  Collect blood. also applies to women of childbearing potential with infrequent or irregular menstrual cycles

- - Collect blood samples for genomic and proteomic/metabolomic analyses
  - Collect blood samples for genetic/epigenetic analysis
- For participating centers, collect blood sample for flow cytometry.
- Obtain MRI of spine and the SI joint if the subject is participating in the MRI substudy. The Baseline MRI should be performed after confirmation of eligibility based on screening assessments for the study and before the first bimekizumab injection.
- Randomize the subject using the IXRS.
- Administer IMP (bimekizumab or placebo)

Collect pulse and BP 30 minutes and 1 hour after dosing.

### 8.3 Double-Blind Period (Week 1 to Week 12)

### Week 1 (+/-3 days) (Visit 3) 8.3.1

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- Determine the BASDAI.
- Determine the BASFI.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.
- Measure temperature, pulse, and BP.
- Collect samples for hematology/biochemistry/urinalysis.
- Collect blood sample for hs-CRP.
- If there has been a delay in menses, perform a urine pregnancy test.

- Collect blood sample for bimekizumab plasma concentrations.
- Collect blood samples for cytokines, complement, and biomarker analyses.
- the BASDAI.

  ctermine the BASFI.

  Perform the PGADA.

  Administer the total and nocturnal spinar pain NRS.

  Measure temperature, pulse, and BP

  Collect samples for hematology/blochemistr

  ollect blood sample for hs-CRP

  here has been a delay in re

  ect blood sample

  rd visit ir

# 8.3.2

- Record visit in the IXRS.

### Week 4 (+/-3 days) (Visit 5) 8.3.3

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.
- eČ-SSRS
- **HADS**
- Administer the AsQoL.
- Determine the BASDAI.
- Determine the BASFI.
- Administer the SF-36.

- Administer the MOS Short Sleep Scale.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.
- Measure temperature, pulse, and BP.
- Determine the MASES.
- Determine the BASMI.
- Administer the PhGADA.
- Collect samples for hematology/biochemistry/urinalysis.
- Collect a blood sample for CRP.
- Collect blood sample for hs-CRP.
- If there has been a delay in menses, perform a urine pregnancy test.
- Collect blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.
- Collect blood samples for cytokines, complement, and biomarker analyses.
- For consenting subjects, collect blood samples for genomic, and proteomic/metabolomic analyses.
- For participating centers, collect blood sample for flow cytometry.
- Record visit in the IXRS.
- Administer IMP (bimekizumab or placebo).

Collect pulse and BP once after dosing.

# 8.3.4 Week 8 (+/-3 days) (Visit 6)

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- HADS

Administer the AsQoL.

- Determine the BASDAI.
- Determine the BASFI.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.

- Measure temperature, pulse, and BP.
- Determine the BASMI.
- Administer the PhGADA.
- Collect samples for hematology/biochemistry/urinalysis.
- Collect blood sample for hs-CRP.
- If there has been a delay in menses, perform a urine pregnancy test.
- Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.
- Record visit in the IXRS.
- Administer IMP (bimekizumab or placebo).

• Collect pulse and BP once after dosing.

# 8.3.5 Week 12 (+/-3 days) (Visit 7)

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- HADS
- Administer the AsQoL.
- Determine the BASDAI.
- Determine the BASFI.
- Administer the SF-36.
- Administer the MOS Short Sleep Scale.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.
- Administer the tuberculosis questionnaire.
- Measure temperature, pulse, and BP.
- Measure weight.
- Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB.
- Determine the MASES.
- Determine the BASMI.

- Administer the PhGADA.
- Perform an ECG.

- Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.

  Collect blood samples for cytokines, complement, and biomarks.

  For consenting subjects:

  Collect blood.
- - Collect blood samples for genomic and proteomic/metabolomics analyses.
  - Collect blood sample for genetic/epigenetic analysis.
- For participating centers, collect blood sample for flow cytometry.
- Obtain MRI of spine and the sacroiliac joint if the subject is participating in the MRI substudy and is MRI-positive at Baseline. Magnetic resonance imaging at Week 12 should be performed as close to the Week 12 Visit as possible.
- Record visit in the IXRS.
- Administer IMP (bimekizumab).

Collect pulse and BP once after dosing (pulse and BP to be collected 30 minutes and 1 hour after dosing).

### 8.4 Dose-Blind Period (Week 16 to Week 48)

### Week 16 (+/-4 days) (Visit 8) 8.4.1

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- HADS
- Administer the AsQoL.
- Determine the BASDAI.
- Determine the BASFI.
- Administer the SF-36.
- Administer the MOS Short Sleep Scale.

- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.

- asymple for hs-CRP.

  If there has been a delay in menses, perform a urine pregnancy test.

  Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.

  Evaluation for rescue treatment eligibility (Section 5.1.4).

  Record visit in the IXRS.

  Administer IMP (bimekizumab).

  Following procedures of ollects.

Collect pulse and BP once after dosing.

### Week 20 (+/-4 days) (Visit 9) 8.4.2

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications
- Record adverse events.
- eC-SSRS
- HADS
- Measure temperature pulse, and BP.
- Collect samples for hematology/biochemistry/urinalysis.
- If there has been a delay in menses, perform a urine pregnancy test.
- Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.
- Record visit in the IXRS.

Administer IMP (bimekizumab).

The following procedures of assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing.

### 8.4.3 Week 24 (+/-4 days) (Visit 10)

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- **HADS**
- Administer the AsQoL.
- Determine the BASDAI.
- Determine the BASFI.
- Administer the SF-36.
- Administer the MOS Short Sleep Scale.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.
- Administer the tuberculosis questionnaire.
- Measure temperature, pulse, and BP.
- Measure weight.

  Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB.
- Determine the BASMI.
- Administer the PhGADA.
- Collect samples for hematology/biochemistry/urinalysis.
- Collect a blood sample for CRP.
- Collect blood sample for hs-CRP.
- If there has been a delay in menses, perform a urine pregnancy test.
- Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.
- Collect blood samples for cytokines, complement, and biomarker analyses.
- For consenting subjects:
  - Collect blood samples for genomic and proteomic/metabolomic analyses.
    - Collect blood sample for genetic/epigenetic analysis.
- For participating centers, collect blood sample for flow cytometry.
- Evaluation for rescue treatment eligibility (Section 5.1.4).
- Record visit in the IXRS.
- Administer IMP (bimekizumab).

application and any extensions of variations thereof.

Collect pulse and BP once after dosing.

# 8.4.4

The following procedures of assessments will be completed prior to administration of IMP:

Record visit in the IXRS.
Administer IMP (bimekizumab).
The following procedures of assessments will be completed following administration of IMP:

# 8.4.5

....stration of IMP:

...stration of IMP:

....stration of IMP:

...stration of IMP:

... The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- **HADS**
- Measure temperature, pulse, and BP.
- Collect samples for hematology/biochemistry/urinalysis.
- If there has been a delay in menses, perform a urine pregnancy test.
- Record visit in the IXRS.
- Administer IMP (bimekizumab).

The following procedures of assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing.

#### Week 36 (+/-4 days) (Visit 13) 8.4.6

The following procedures of assessments will be completed prior to administration of IMP:

- ...octurnal spinal pain NRS.
  ...reculosis questionnaire.
  ...perature, pulse, and BP.
  ...re weight.

  Administer the PhGADA.

  Collect samples for hematology/biochemistry/urinalysis.

  Collect blood sample for bimekizumab plase body detection ation for rescue treatment elip?'

  1 visit in the IXRS.
  ...ster IMP (bimek;
  ...g procede)
  ...serulosis questionnaire.
  ...perature, pulse, and BP.
  ...re weight.

  Administer the PhGADA.

  Collect samples for hematology/biochemistry/urinalysis.

  Collect sample for bimekizumab plase body detection.

  1 visit in the IXRS.
  ...ster IMP (bimek;
  ...g procede)
  ...serulosis questionnaire.
  ...perature, pulse, and BP.
  ...re weight.

  Administer the PhGADA.

  Collect samples for hematology/biochemistry/urinalysis.

  Collect sample for bimekizumab plase body detection.

  1 visit in the IXRS.
  ...ster IMP (bimek;
  ...g procede)

The following procedures of assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing.

#### 8.4.7 Week 40 (+/-4 days) (Visit 14)

The following procedures of assessments will be completed prior to administration of IMP:

- Record concomitant medications.
- Record adverse events.

09 Mar 2018

AS0008

- eC-SSRS
- **HADS**
- Measure temperature, pulse, and BP.
- Collect samples for hematology/biochemistry/urinalysis.
- If there has been a delay in menses, perform a urine pregnancy test.
- Record visit in the IXRS.
- Administer IMP (bimekizumab).

The following procedures of assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing.

#### Week 44 (+/-4 days) (Visit 15) 8.4.8

The following procedures of assessments will be completed prior to administration of IMP:

Record concomitant medications.

Record adverse events.

eC-SSRS

HADS

Measure temperature, pulse, and BP.

Collect samples for hematology/biochemistry/urinalysis.

- If there has been a delay in menses, perform a urine pregnancy test.
- Perform the IGRA tuberculosis test.
- Record visit in the IXRS.
- Administer IMP (bimekizumab). This is the last dose of IMP.

The following procedures of assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing.

## Week 48 (+/-4 days) (Visit 16) 8.4.9

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- **HADS**
- Administer the AsQoL.
- Determine the BASDAI.
- Determine the BASFI.
- Administer the SF-36.

- Administer the MOS Short Sleep Scale.
- Perform the PGADA.
- Administer the total and nocturnal spinal pain NRS.
- Administer the tuberculosis questionnaire.
- Measure temperature, pulse, and BP.
- Measure weight.
- s of a splication and any extensions Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB.
- Determine the MASES.
- Determine the BASMI.
- Administer the PhGADA.
- Perform an ECG
- Collect samples for hematology/biochemistry/urinalysis.
- Collect a blood sample for CRP.
- Collect blood sample for hs-CRP.
- Perform a urine pregnancy test if the subject is a woman of childbearing potential. This requirement also applies to women of childbearing potential with infrequent or irregular menstrual cycles and women during menopause. Natural menopause is recognized to have occurred after 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause (International Menopause Society, 2015).
- Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.
- Collect blood samples for cytokines, complement, and biomarker analyses.
- For consenting subjects, collect blood samples for genomic and proteomic/metabolomic analyses.
- For participating centers, collect blood sample for flow cytometry.
- Obtain MRI of spine and the sacroiliac joint if the subject is participating in the MRI substudy and is MRI-positive at Baseline. Magnetic resonance imaging at Week 48 should be performed as close to the Week 48 Visit as possible.
- Record visit in the IXRS.

# **Early Termination Visit**

- Record concomitant medications.
- Record adverse events.
- eC-SSRS
- **HADS**

- Administer the AsOoL.
- Determine the BASDAI.

- and spinal pain NRS.

  Aculosis questionnaire.

  Actemperature, pulse, and BP.

  Measure weight.

  Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB.

  Determine the MASES.

  Determine the BASMI.

  dminister the PhGADA

  rform an ECG.

  llect samples for hematology/\*

  lect a blood same\*

- Collect blood sample for hs-CRP.
- Perform a urine pregnancy test of the subject is a woman of childbearing potential. This requirement also applies to women of childbearing potential with infrequent or irregular menstrual cycles and women during menopause. Natural menopause is recognized to have occurred after 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause (International Menopause Society, 2015).
- Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection.
- Collect blood samples for cytokines, complement, and biomarker analyses.
- For consenting subjects, collect blood samples for genomic and proteomic/metabolomic analyses.

For participating centers, collect blood sample for flow cytometry.

- Perform an IGRA tuberculosis test.
- Record visit in the IXRS.
- If subject is a PDILI case that results in immediate, permanent IMP discontinuation, conduct a thorough evaluation as described in Section 12.5.1.

## Safety Follow-Up Visit (20 weeks [-3 days/+7 days] after the final 8.6 dose)

- .cep Scale.

  .cep Scale.

  .ster the tuberculosis questionnaire.

  Measure temperature, pulse, and BP.

  Measure weight.

  Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB.

  Vetermine the BASMI.

  Iminister the PhGADA.

  Form an ECG.

  cet samples for hematology/biochemistry/urinalysis.

  1 a blood sample for CRP.

  blood sample for he-CRP.

  a urine pregnancy test if the subjection and active the result of the subjection of the subj Tomen during menopause. Natural menopause is recognized after 12 consecutive months of amenorrhea, for which there is no oth pathological or physiological cause (International Menopause Society, 2015).

  Collect a blood sample for bimekizumab plasma concentrations antibody detection.

  Perform
  - Collect a blood sample for bimekizumab plasma concentrations and anti-bimekizumab

  - Record visit in the IXRS.

#### 8.7 **Unscheduled Visit**

At the Investigator's discretion, an Unscheduled Visit may be completed at any time during the study but prior to the SFU Visit, if deemed necessary for the subject's safety and well-being.

reasons other than safety or efficacy concerns (eg, replacement of lost medication, repeated collection of a laboratory specimen due to collection or analysis issues) an eC-SSRS will not be required at these visits.

At this visit, any of the following assessments may be note that the visit:

- Record concomitant medication
- Record AEs
- eC-SSRS
- Vital signs
- Physical examination
- Record 12-lead ECG
- If medically indicated, obtain blood sample(s) for:
  - Standard safety laboratory tests (hematology, serum chemistry)
  - The blood sample may also be used for PK/PD assessments, if needed.
- Obtain urine sample for standard safety laboratory tests (including urine pregnancy test)

### 9 ASSESSMENT OF EFFICACY

The timing for all assessments described below is specified in the Schedule of Assessments, Table 5–1.

### ASAS20, 40, ASAS 5/6 response, and ASAS partial remission 9.1

The ASAS20 is defined as an improvement of at least 20% and absolute improvement of at least 1 unit on a 0 to 10 NRS in at least 3 of the 4 following domains:

- PGADA (see Section 9.2)
- Pain assessment (the total spinal pain NRS score; Section 9.3)
- Function (represented by BASFI, Section 9.4)
- Inflammation (the mean of the BASDAI questions 5 and 6, [see Section 9.5]

and absence of deterioration in the potential remaining domain [deterioration is defined as a relative worsening of at least 20% and an absolute worsening of at least 1 unit].

The ASAS criteria for 40% improvement are defined as relative improvements of at least 40%, and absolute improvement of at least 2 units on a 0 to 10 NRS in at least 3 of the 4 domains and no worsening at all in the remaining domain.

The ASAS 5/6 response is defined as at least 20% improvement in 5 of 6 domains, including spinal mobility (lateral spinal flexion) and hs-CRP as more objective measures (Brandt et al., 2004).

Patient global assessment
Subjects will score their global assessment of their disease activity in response to the question "How active was your spondylitis on average during the last week?" using a NRS where 0 "not active" and 10 is "very active" (van Tubergen et al, 2015).

9.3

Total and nocture.

The pain experienced by AS subjects is adequately measured by 2 separate questions: 1) total pain in the spine due to AS (ie, "How much pain of your spine due to spondylitis do you have?"); and 2) pain in the spine at night due to AS (ie, "How much pain of your spine due to spondylitis do you have at night?") (Sieper et al, 2009; van der Heijde et al, 2005; Committee for Proprietary Medicinal Product [CPMP]/EWP/556/95). When responding to each question, the subject is to consider the average amount of pain in the preceding week.

#### 9.4 Function – BASFI

The BASFI is a validated disease-specific instrument for assessing physical function (van der Heijde et al, 2005; Calin et al, 1994). The BASFI comprises 10 items relating to the past week. The NRS version will be used for the answering options of each item on a scale of 0 ("Easy") to 10 ("Impossible") (van Tubergen et al, 2015 and van Tubergen et al, 2002a). The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function. The MCID used to interpret scores is 7mm on a 0 to 100mm visual analog scale (VAS) or 17.5% of the Baseline score (Pavy et al, 2005); an MCID of 1 unit will be used for the NRS version.

## Inflammation BASDAI (mean of questions 5 and 6) 9.5

Question 5 of the BASDAI (described completely in Section 9.8) measures . The subject considers the previous week and responds to the question, "

The response is indicated on a 10-point NRS in which 0=None and 10=Very severe. Question 6 of the BASDAI measures . The subject considers the previous week and responds to the question, "

The response is indicated on a 10-point NRS in which 0=0 hours, 5=1 hour, and 10=2 or more hours. The ratings for each question are summed and divided by 2 to provide the mean of questions 5 and 6.

# CRP

This document Blood will be collected for measurement of CRP and hs-CRP. After Screening, the CRP data will not be sent to the Investigator to protect the blinded nature of the treatment assignments.


#### 9.7 ASDAS-CRP

The ASDAS is comprised of a number of assessments which are scored by the subject and ions of variations thereof. Investigator and multiplied by a validated formula (van der Heijde et al, 2009) as listed:

- (BASDAI Q2 result, Section 9.8) 0.121 x
- 0.058 x(BASDAI Q6 result, Section 9.8)
- 0.110 x PGADA (Section 9.2)
- 0.073 x(BASDAI Q3 result, Section 9.8)
- $0.579 \times (\text{natural logarithm of the CRP } [\text{mg/L}] + 1)$

, PGADA,

assessed on a numerical scale (0 to 10 units) (Lukas et al, 2009). The results of these calculations are summed to calculate the ASDAS.

#### 9.8 BASDAI

The most common instrument used to measure the disease activity of AS from the subject's perspective is the BASDAI (Garrett et al, 1994). The BASDAI is a validated self-reported instrument which consists of six 10-unit horizontal NRSs to

(van Tubergen et al., 2015). The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity. Question 2 of the BASDAI asks the subject to describe

factor in the calculation of ASDAS-CRP.

Question 3 of the BASDAI asks the subject to

factor in the calculation of ASDAS-CRP. Question 6 of the BASDAI asks the subject to describe

factor in the calculation of ASDAS-CRP.

The BASDAI is calculated as follows:

$$BASDAI = \frac{Q1+Q2+Q3+Q4+(\frac{Q5+Q6}{2})}{5}$$

Fatigue item of the BASDAI

Fatigue as a major symptom of AS can effectively be measured with single-item questions such as the BASDAI item (van Tubergen et al, 2002b). This item has shown moderate to good reliability and responsiveness (van Tubergen et al, 2002b). The same MCID will be used for the fatigue item of the BASDAI as for the total BASDAI score, ie, a change of 1 unit on the NRS.

## 9.9 BASMI

The BASMI characterizes the spinal mobility of subjects with AS. The BASMI is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral spinal flexion; modified Schober test; intermalleolar distance. Each of the 5 movements is scored according to the linear BASMI definition. The mean of the 5 scores provides the BASMI score. The higher the BASMI score the more severe the subject's limitation of movement due to their AS.


#### 9.10 **MASES**

Enthesitis is assessed with MASES. The MASES is an index that measures the severity (ie, Valiations the reof. intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) (Heuft-Dorenbosch et al, 2003) each scored as 0 or 1 and then summed for a possible score of 0 to 13.

#### 9.11 **PhGADA**

The Investigator will assess the overall status of the subject with respect to their AS signs and symptoms and functional capacity (considering both joint and skin components) using an NRS in which 0=very good, asymptomatic and no limitations of normal activities and 10=very poor, very severe symptoms which are intolerable and inability to carry out normal activities.

This assessment by the Investigator should be made blind to the PGADA.

The subject should be asked to consider both joint and skin components in their response to this question.

#### 9.12 **SF-36**

The SF-36 (Version 2, standard recall) is a 36-item generic health-related quality of life (HRQoL) instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and 1 item for perceived stability or change in health (Health Transition) during the last year. The concepts represented by these domains contribute to physical, mental, and social aspects of HROoL.

In addition to domain scores, the Physical Component Summary and Mental Component Summary scores are calculated from the 8 domains (excluding the Health Transition item). Component scores appreciate the impact of each domain on physical and mental health status (Maruish, 2011). Each of the 8 domain scores and the component summary scores range from 0 to 100, with a higher score indicating a better health status. The 2 component summary scores are standardized with a mean of 50 and a standard deviation (SD) of 10 in the general US population.

### **MOS-12** 9.13

The MOS Sleep Scale is a validated generic self-administered scale measuring specific aspects of sleep. The frequency with which each problem has been experienced during the previous 4 weeks is rated on a 6-point scale ranging from "none of the time" to "all of the time," except sleep quantity, which is reported in hours. All scores are transformed linearly to range from 0 to 100, again with the exception of the sleep quantity subscale, which is scored in hours. Higher scores indicate more of the attribute implied by the scale name (eg, more sleep disturbance, more adequate sleep, and greater sleep quantity). The psychometric properties of the MOS Sleep Scale have been found to be satisfactory by Hays and colleagues (Hays et al, 2005). The domains of interest for this study are the Sleep Disturbance and the Sleep Problems Index II domains.

**UCB** 

The ASQoL, a validated disease-specific 18-item questionnaire, has been developed specifically for measuring HROoL in subjects with AS (Doward et al. 2003). The ASOoL has been used and

while radiography can detect chronic bony changes (eg, sclerosis, erosions, bridging, and ankyloses), structural changes generally occur slowly and x-rays are insensitive; therefore, changes are difficult to detect in the relatively short duration of a randomized clinical trial. Unlike radiography, MRI can be used to visualize inflammation in the ST in expected that radiography amenable to treatment appreciately specifically amenable to treatment. expected that reduction in inflammation in the SI joints and spine can be detected using MRI within the 48-week Treatment Period of this study. Recently a Danish study demonstrated significant changes in in ASspiMRI-a (Berlin modification) and SPARCC MRI-assessed inflammation scores and in SPARCC MRI-assessed erosion scores within 12 weeks after initiation of adalimumab (see below for further description of these MRI scoring methods). The researchers concluded that MRI-assessed structural lesions change rapidly and may have value for assessing the effects of disease-modifying treatment in clinical trials (Pedersen SJ et al, 2016).

An MRI of the spine and sacroiliac joints will be performed in a substudy with approximately 20 subjects per treatment arm at Baseline. A central reader will assess Baseline MRIs to identify MRI-positive subjects as per the ASAS-Outcome Measures in Rheumatology Clinical Trials (OMERACT) criteria. An MRI at Week 12 and Week 48 will be performed for those subjects who were MRI-positive at Baseline. The Baseline MRI should be performed after confirmation of eligibility based on screening assessments for the study and before the first bimekizumab injection. Magnetic resonance imaging at Week 12 and Week 48 should be performed as close to the Week 12/Week 48 Visit as possible. Additional details for standardized performance and processing of MRIs will be provided in an MRI manual. The MRIs will be read centrally by readers who are blinded to treatment assignment and chronological order of the MRIs according to a charter for independent imaging assessment.

The following 2 different scoring systems will be utilized to determine changes from Screening (Lukas et al, 2007):

# ASspiMRI-a (Berlin modification) score

This method is a scoring system with a concentration on short-tau-inversion recovery (STIR) sequences which quantifies changes in 23 disco-vertebral units (DVU) of the spine. A DVU is defined as the region between 2 virtual lines through the middle of each vertebra. Active inflammation is scored by grading the degree of bone marrow edema from 0 to 3 in 1 dimension on 1 or more consecutive slices that represent the highest level of inflammation in a particular VU. There is no grading for erosion in the Berlin modification. The total spine ASspiMRI-a score in the Berlin modification can range from 0 to 69.


# SPARCC SI Joint score

This method is a scoring system for assessing the SI joint based on STIR sequences. An abnormal increased signal on the STIR sequence represents bone marrow edema. The SI joint is 1—Increased signal. The maximum score for abnormal signal in the 2 SI joints of 1 coronal slice is therefore 8. Joints that include a lesion exhibiting intense signal are each given an additional score of 1 per slice (that demonstrate this feature). Each SI joint that includes a lesion demonstrating continuous increase signal of depth  $\geq 1$  cm from the articular surface an additional score of 1. The maximum score for a score of 1 and of 6 according to the score of 1. in each of 6 consecutive coronal slices, so that the total SI joint SPARCC MRI score can range from 0 to 72.

### **Hospital Anxiety and Depression Scale** 9.16

The HADS was chosen for its well-established psychometric properties and its use in clinical research on biological therapy in subjects with chronic plaque psoriasis (Langley et al, 2010; Dauden et al, 2009). The HADS scores for anxiety and for depression range from 0 to 21 with higher scores indicating worse state. A score below 8 is considered to be normal whereas a score of 15 and above is considered severe (Snaith and Zigmond, 1994).

# ASSESSMENT OF PHARMACOKINETIC, 10 PHARMACODYNAMIC, PHARMACOGENOMIC, AND PROTEOMIC VARIABLES

Plasma concentrations of bimekizumab, population PK variables (CL/F, V/F) and dose-exposure responses (for ASAS40 response) are the PK variables.

The PD variables are the concentrations of cytokines of relevance to IL-17A/F signaling pathway and AS biology. Where local regulations permit, additional blood samples will be collected from consenting subjects at specific time points and stored at -80°C for up to 20 years to allow for potential exploratory analyses of genomic, genetic/epigenetic, proteomic, and metabolite biomarkers relevant to the disease biology, disease progression, response to therapy, and inflammatory and immune response processes

The Investigator or designee will obtain blood samples for these measurements at the time points specified in Table 3–1. When these samples are required at a visit during which the subject is dosed with IMP, the blood samples will be drawn prior to dosing. Samples should be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF. Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. Detailed information on sample analysis will be provided in a bioanalytical report.

# ASSESSMENT OF IMMUNOLOGICAL VARIABLES

This docurat The immunological variables comprise detection of anti-bimekizumab antibodies related to immunogenicity, serum complement concentrations, mononuclear cell subtypes (analyzed by flow cytometry/fluorescence-activated cell sorting), and other exploratory biomarkers.

> The Investigator or designee will obtain blood samples for these measurements at the time points specified in Table 5–1. When these samples are required at a visit during which the subject is

 dosed with IMP, the blood samples will be drawn prior to dosing. Samples should be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be 75 Of Variations thereof recorded in the eCRF. Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. The presence of antibodies to bimekizumab will be determined using a validated bioanalytical method. Detailed information on sample analysis will be provided in a bioanalytical report.

#### 12 ASSESSMENT OF SAFETY

#### 12.1 Adverse events

#### 12.1.1 Definition of adverse event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In order to ensure complete safety data collection, all AEs occurring during the study (ie, after the signing of the Informed Consent Form), including any pretreatment and posttreatment periods required by the protocol, must be reported in the eCRF even if no IMP was taken but specific study procedures were conducted. This includes all AEs not present prior to the initial visit and all AEs that recurred or worsened after the initial visit.

Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the Investigator from the subject's history or the Baseline Period.

### Adverse events of special interest 12.1.2

An AE of special interest (AESI) is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.

Potential Hy's Law, defined as ≥3xULN ALT or AST with coexisting ≥2xULN total bilirubin in the absence of >2xULN ALP, with no alternative explanation for the biochemical abnormality. must ALWAYS be reported to UCB as an AESI (ie, without waiting for any additional etiologic investigations to have been concluded). Follow-up information should then be reported if an alternative etiology is identified during investigation and monitoring of the subject.

# Adverse events for special monitoring

UCB has identified AEs for special monitoring (AESM). An AESM is an AE or safety topic for which special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB), are considered appropriate. Identified AESM can be of particular concern based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or comorbidities and risk factors prevalent in the study population.

Adverse events for special monitoring for this study include: serious infections (including opportunistic infections and TB, see Section 12.6.5), cytopenias, hypersensitivities, suicide

 ideation or behavior (assessed using the eC-SSRS), depression and anxiety (assessed using the HADS, see Section 9.16), major cardiovascular events and liver function test changes/enzyme elevations (ALT, AST, and bilirubin; see Section 12.5.1), malignancies, and inflammatory bowel diseases.

# 12.1.4 Procedures for reporting and recording adverse events

The subject will be given the opportunity to report AEs spontaneously. A general prompt will also be given at each study visit to detect AEs. For example:

"Did you notice anything unusual about your health (since your last visit)?"

In addition, the Investigator should review any self-assessment procedures (eg, diary cards) employed in the study.

# 12.1.5 Description of adverse events

When recording an AE, the Investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words on his/her own records (eg, diary card) and the corresponding medical terminology should be clarified in the source documentation.

When recording the intensity of an AE in the eCRF (ie, mild, moderate, or severe), the Investigator should use the following criteria:

- Mild: the subject is aware of the sign or symptom (syndrome), but it does not interfere with his/her usual activities and/or is of no clinical consequence
- Moderate: the AE interferes with the usual activities of the subject or it is of some clinical consequence
- Severe: the subject is unable to work normally or to carry out his/her usual activities, or the AE is of definite clinical consequency

Details for completion of the Adverse Event eCRF (including judgment of intensity and relationship to IMP) are described in the eCRF Completion Guidelines.

# 12.1.6 Follow-up of adverse events

An AE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, AESIs, and AESMs; further details regarding follow-up of PDILI events are provided in Section 12.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the Patient Safety (PS) database without limitation of time.

If an AE is ongoing at the end of the study for a subject, follow-up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems that it is clinically significant, or until the subject is lost to follow-up. If no follow-up is provided, the Investigator must provide a justification. The follow-up will usually be continued for 20 weeks after the subject has discontinued his/her IMP.
An increase in the intensity of an AE should lead to the repetition of the AE being reported with:

- Valiations thereof. The outcome date of the first AE that is not related to the natural course of the disease being the same as the start date of the repeated AE, and the outcome of "worsening"
- The AE verbatim term being the same for the first and repeated AE, so that the repeated AE can be easily identified as the worsening of the first one

#### 12.1.8 **Pregnancy**

**UCB** 

If an Investigator is notified that a subject has become pregnant after the first intake of any IMP, the Investigator must immediately notify UCB's PS department by providing the completed Pregnancy Report and Outcome Form (for contact details see SAE reporting information at the beginning of this protocol). The subject should be withdrawn from the study as soon as pregnancy is known (by positive pregnancy test), and the following should be completed:

- The subject should return for the ET Visit.
- The subject should immediately stop the intake of the IMP.
- An SFU Visit should be scheduled 20 weeks after the subject has discontinued her IMP.

The Investigator must inform the subject of information currently known about potential risks and about available treatment alternatives.

The pregnancy will be documented on the Pregnancy Report and Outcome Form provided to the Investigator. The progression of the pregnancy and the eventual birth (if applicable) must be followed up using the Pregnancy Report and Outcome Form in which the Investigator has to report on the health of the mother and of the child. Every reasonable attempt should be made to follow the health of the child for 30 days after birth for any significant medical issues. In certain circumstances, UCB may request that follow-up is continued for a period longer than 30 days. If the subject is lost to follow-up and/or refuses to give information, written documentation of attempts to contact the subject needs to be provided by the Investigator and filed at the site. UCB's Drug Safety department is the primary contact for any questions related to the data collection for the pregnancy, eventual birth, and follow-up.

In cases where the partner of a male subject enrolled in a clinical study becomes pregnant, the Investigator or designee is asked to contact the subject to request consent of the partner via the Partner Pregnancy Consent Form that has been approved by the responsible IRB/IEC and should be available in the Investigator site file. In case of questions about the consent process, the Investigator may contact the UCB/ CRO contract monitor for the study. The Investigator will complete the Pregnancy Report and Outcome Form and send it to UCB's PS department (for Partner Pregnancy Consent Form. UCB's PS department is also the primary contact for any questions related to the data collection for the partner pregnancy, eventual birth and the provided the signed.

A pregnancy becomes an SAE: contact details see SAE reporting information at the beginning of this protocol) only after the questions related to the data collection for the partner pregnancy, eventual birth, and follow-up.

A pregnancy becomes an SAE in the following circumstances: miscarriage, elective abortion when medically indicated (eg., when pregnancy is endangering life or health of woman or when fetus will be born with severe abnormalities), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal


09 Mar 2018 AS0008

demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report form.

# 12.1.9 Suspected transmission of an infectious agent via a medicinal product

For the purposes of reporting, any suspected transmission of an infectious agent via a medicinal product should be considered as an SAE; such cases must be reported immediately, recorded in the AE module of the eCRF, and followed as any other SAE. Any organism, virus, or infectious particle (eg, prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

# 12.1.10 Overdose of investigational medicinal product

Excessive dosing (beyond that prescribed in the protocol and including overdose) should be recorded in the eCRF. Any SAE or nonserious AE associated with excessive dosing must be followed as any other SAE or nonserious AE. These events are only considered AEs or SAEs if there are associated clinical signs and symptoms or if the act of taking the excess medicine itself is an AE or SAE (eg, suicide attempt).

# 12.1.11 Safety signal detection

Selected data from this study will be reviewed periodically to detect as early as possible any safety concern(s) related to the IMP so that Investigators, clinical study subjects, regulatory authorities, and IRBs/IECs will be informed appropriately and as early as possible.

The Study Physician or medically qualified designee/equivalent will conduct an ongoing review of SAEs and perform ongoing SAE reconciliations in collaboration with the PS representative.

As appropriate for the stage of development and accumulated experience with the IMP, medically qualified personnel at UCB may identify additional safety measures (eg, AEs, vital signs, laboratory or ECG results) for which data will be periodically reviewed during the course of the study.

In addition, an independent DMC will periodically review and monitor the safety data from this study and advise UCB. The DMC membership includes clinicians knowledgeable about the disease or the treatment. All members have experience and expertise in clinical trials. Board members may not participate in the study as principal or co-Investigators, or as study subject care physicians. The duration of membership for the DMC will be inclusive of planned analyses for AS0008. The DMC may also be asked to provide a review of final study results, as deemed appropriate. The DMC procedures will ensure that data remain blind to the study team and Investigators at all times throughout the conduct of the study. The detailed role, scope, responsibilities, and complete procedures, as well as the identity of the DMC members, will be described in a separate charter document. A cardiovascular adjudication committee will be in place for this study. Specific procedures will be outlined in the charter, which will be developed by the committee members.

#### 12.2 Serious adverse events

#### 12.2.1 Definition of serious adverse event

Once it is determined that a subject experienced an AE, the seriousness of the AE must be determined. An SAE must meet 1 or more of the following criteria:

- Death
- Life-threatening

itations thereof (Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.)

- Significant or persistent disability/incapacity
- Congenital anomaly/birth defect (including that occurring in a fetus)
- Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious.

(Important medical events may include, but are not limited to potential Hy's Law [see Section 12.1.2], allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.)

Initial inpatient hospitalization or prolongation of hospitalization

A patient admitted to a hospital, even if he/she is released on the same day, meets the criteria for the initial inpatient hospitalization. An emergency room visit that results in admission to the hospital would also qualify for the initial inpatient hospitalization criteria. However, emergency room visits that do not result in admission to the hospital would not qualify for this criteria and, instead, should be evaluated for 1 of the other criteria in the definition of serious (eg, life-threatening adverse experience, important medical event).

Hospitalizations for reasons not associated with the occurrence of an AE [eg, preplanned surgery or elective surgery for a pre-existing condition that has not worsened or manifested in an unusual or uncharacteristic manner] do not qualify for reporting. For example, if a subject has a condition recorded on his/her medical history and later has a preplanned surgery for this condition, it is not appropriate to record the surgery or hospitalization as an SAE, since there is no AE upon which to assess the serious criteria. Please note that, if the pre-existing condition has worsened or manifested in an unusual or uncharacteristic manner, this would then qualify as an AE and, if necessary, the seriousness of the event would need to

SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements.

12.2.2 Procedures for reporting serious adverse avantation of the SAE is not a serious adverse avantation.

If an SAE is reported, UCB must be informed within 24 hours of receipt of this information by the site (see contact information for SAE reporting listed in the SAE Reporting section at the front of the protocol). The Investigator must forward to UCB (or its representative) a duly completed "Investigator SAE Report Form for Development Drug" (SAE report Form) provided

 by UCB, even if the data are incomplete, or if it is obvious that more data will be needed in order to draw any conclusions. Information recorded on this form will be entered into the global PS database.

In is important for the Investigator, when completing the SAE report Form, to include the assessment as to a causal relationship between the SAE and the IMP administration. This insight from the Investigator is very important for UCB to consider in assessing the safety of the IMP and in determining whether the SAE requires reporting to the rocal expedited manner.

Additional information (eg., autopsy or laboratory reports) received by the Investigator must be provided within 24 hours. All documents in the local language must be accompanied by a translation in English, or the relevant information included in the same document must be summarized in the Investigator SAE report Form.

The Investigator is specifically requested to collect and report to UCB (or its representative) any SAEs (even if the Investigator is certain that they are in no way associated with the IMP), up to 30 days from the end of the study for each subject, and to also inform participating subjects of the need to inform the Investigator of any SAE within this period. Serious AEs that the Investigator thinks may be associated with the IMP must be reported to UCB regardless of the time between the event and the end of the study.

Upon receipt of the SAE report Form, UCB will perform an assessment of expectedness of the reported SAE. The assessment of the expectedness of the SAE is based on the IB.

## Follow-up of serious adverse events 12.2.3

An SAE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, AESIs, and AESMs; further details regarding follow-up of PDILI events are provided in Section 12.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the PS database without limitation of time.

# Immediate reporting of adverse events 12.3

The following AEs must be reported immediately:

- SAE: AE that the Investigator classifies as serious by the above definitions regardless of causality
- Suspected transmission of an infectious agent via a medicinal product
- AEs of special interest as defined in Section 12.1.2

# **Anticipated serious adverse events**

his document. The following list of Anticipated SAEs (Table 12–1) has been identified, as these events are anticipated to occur in the population studied in this protocol at some frequency that is independent of drug exposure. This original list will remain in effect for the duration of the protocol. Note that listed events will not be regarded as anticipated SAEs if they are life threatening or if they result in the death of the study subject.

This list does not change the Investigator's obligation to report <u>all</u> SAEs (including Anticipated SAEs) as detailed in Section 12.2.2.

Table 12–1: Anticipated serious adverse events for the population of subjects with ankylosing spondylitis

| MedDRA system organ class | MedDRA preferred term |
|---|---|
| Skin and subcutaneous tissue disorders | Psoriasis |
| Eye disorders | Uveitis |
| Musculoskeletal and connective tissue disorders | Dactylitis Tendonitis Atlantoaxial instability |
| Gastrointestinal disorders | Colitis ulcerative<br>Crohn's disease |
| Cardiac disorders | Aortic valve incompetence Atrial tachycardia Atrioventricular block Bundle branch block Cardiomyopathy |
| Vascular disorders | Aortitis |
| Respiratory, thoracic and mediastinal disorders | Pulmonary fibrosis |
| Nervous system disorders | Cauda equina syndrome |
| Injury, poisoning and procedural complications | Spinal cord injury Spinal fracture Cervical Vertebral fracture Lumbar Vertebral fracture Thoracic Vertebral fracture |
| Immune system disorders | Amyloidosis |
| Psychiatric disorders | Depression |

MedDRA=Medical Dictionary for Regulatory Activities

Note: Exception: Listed events will not be regarded as anticipated SAEs if they are life threatening or if they result in the death of the study subject.

# 12.5 Laboratory measurements

Clinical laboratory assessments consist of serum chemistry, hematology, and urinalysis, and pregnancy tests (serum or urine) (Table 12–2). A centralized laboratory will be used to supply all laboratory test supplies and analyze all blood and urine samples for hematology, biochemistry and urinalysis measurements. Any unscheduled laboratory testing should also be collected using the central laboratory. Testing to rule out hepatitis B, hepatitis C, and HIV (see Exclusion Criterion #9, Section 6.2) will be performed at Screening in addition to those measurements listed in Table 12–2.

Specific details regarding the handling and processing of serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.


# Table 12-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis |
|---|---|---|
| Basophils | Calcium | Albumin |
| Eosinophils | Chloride | Bacteria |
| Lymphocytes | Magnesium | Crystals |
| Atypical lymphocytes | Potassium | Glucose |
| Monocytes | Sodium | pH |
| Neutrophils | Glucose | RBC |
| Hematocrit | BUN | WBC |
| Hemoglobin | Creatinine | Urine dipstick for pregnancy testing <sup>a</sup> |
| MCH | AST | 0101 |
| MCHC | ALT | 7 2/1 |
| MCV | ALP | alle |
| Platelet count | GGT | diol |
| RBC count | Total bilirubin | dico |
| WBC count | LDH | , P |
| | Uric acid | |
| | Total cholesterol | |
| | Serum pregnancy testing <sup>a</sup> | |
| | CRPb | |
| | hs-CRP <sup>b</sup> | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CRP=C-reactive protein; GGT=gamma glutamyltransferase; hs-CRP=high sensitivity C-reactive protein; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; SFU=Safety Follow-up; WBC=white blood cell

# 12.5.1 Evaluation of PDILI

The PDILI IMP discontinuation criteria for this study are provided in Section 6.3.1, with the accompanying required follow-up investigation and monitoring detailed below. All PDILI events must be reported as an AE and reported to the study site and sponsor within 24 hours of learning of their occurrence. Any PDILI event that meets the criterion for potential Hy's Law must be

A serum pregnancy test will be performed at Screening for all women of childbearing potential. This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles and women during menopause. Natural menopause is recognized to have occurred after 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause (International Menopause Society [IMS], 2015). A urine pregnancy test is also required at the Baseline, Week 48, ET, and at SFU visits. A urine pregnancy test will also be performed at any study visit where there has been a delay in menses. This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles. Pregnancy test results must be negative prior to administering IMP.

b Both CRP and hs-CRP will be tested at specified visits per Table 5–1.

reported as an AE of special interest (see Section 12.1.2), and, if applicable, also reported as an SAE (see Section 12.2.1).

Evaluation of PDILI consists of the diagnostic testing and continued monitoring included in Table 12–3 (specific tests dependent on laboratory results and corresponding symptoms) and consultation with a local hepatologist (if applicable; discussed in Section 12.5.1.1). The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. Additional investigation and monitoring may be required and adapted based on the diagnosis after the cause of the liver injury/abnormality is confirmed (details in Section 12.5.1.5).

The results of all monitoring, including laboratory testing and other testing, should be made available to the study site and sponsor.

All initial tests resulting in abnormal hepatic laboratory values need to be repeated, but appropriate medical action must not be delayed waiting for the repeat result.

If tests are done locally for more rapid results, a concurrent sample should also be sent to the central laboratory whenever possible. Medical care decisions are to be made initially using the most rapidly available results and a conservative approach must be taken if the results from the 2 laboratory tests are significantly different. Data from the local and central laboratory are to be recorded on the applicable eCRF pages.

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. In these cases, the Investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, may be fatal, and must not occur.

the a the authority of the lised to support this document cannot be used to support the lised Table 12-3 summarizes the approach to investigate PDILI.

# Table 12-3: Required investigations and follow-up for PDILI

| Laboratory value | Table 12–3: Require | Required investigations | s and follow-up for PDILI | PDILI | | Mel4 |
|---|---|---|---|---|---|---|
| | value | | Immediate | diate | ************************************** | Follow-up |
| ALT or AST | Total<br>bilirubin | Symptoms <sup>a</sup> of hepatitis of hypersensitivity | Consultation requirements | Actions | Testing Charles | Evaluation |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult <sup>c</sup> | Immediate, permanent | Essential Must have | Monitoring of liver |
| ≥3xULN | NA | Yes | Medical Monitor must<br>be notified within<br>24 hours (eg, by<br>laboratory alert) and<br>subject discussed with<br>Medical Monitor ASAP. | IMP discontinuation | repeat ther chemistry values and additional testing completed ASAP (see Section 12.5.1.4); recommended to occur | chemistry values at least twice per week until values normalize, stabilize, or return to within baseline values <sup>d</sup> |
| ≥5xULN | NA | NA | Need for hepatology consult to be discussed.( required if ALT or AST >8xULN) Medical Monitor must be notified within 24 hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP. | Immediate, permanent IMP discontinuation | at the site with HCP. | |
| >3xULN (and >2x baseline) and <5xULN (and >2x baseline) and <5xULN (and >2x baseline) | <2xULN <2xULN | e) No | Discussion with Medical Monitor required. Consider need for hepatology consult if there is no evidence of resolution (see Follow-up requirements). | Further investigation – immediate IMP discontinuation not required (see Section 12.5.1.2). IMP discontinuation required if any of the following occur: Subject cannot comply with monitoring schedule. | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48 hours at the site with HCP (see Section 12.5.1.4). | Monitoring of liver chemistry values at least twice per week for 2 weeks. <sup>d</sup> • Immediate IMP discontinuation required if liver chemistry values continue to increase. |

| | | | | | | 00 Mar 2018 |
|---|---|---|---|---|---|---|
| Clinical Study Protocol | Protocol | | Birr | Bimekizumab | | AS0008 |
| le 12–3 | : Require | Table 12–3: Required investigations an | s and follow-up for PDILI | PDILI | | ORCHE |
| Laboratory value | y value | | Imme | Immediate | <b>₹</b> | Follow-up |
| ALT or AST | Total<br>bilirubin | Symptoms <sup>a</sup> of hepatitis of hypersensitivity | Consultation<br>requirements | Actions | Testing Testing | Evaluation |
| | | | | <ul> <li>Liver chemistry</li> </ul> | to | |
| | | | | values continue to | TC, | liver chemistry values: |
| | | | | increase | | <ul> <li>Discontinue IMP if</li> </ul> |
| | | | | <ul> <li>Liver chemistry</li> </ul> | DU <sub>K</sub> | |
| | | | | values remain | | |
| | | | | >3xULN (and | | without evidence of |
| | | | | ≥2x baseline) after 2 | | resolution <sup>d</sup> |
| | | | | weeks of monitoring | | Continue to monitor until |
| | | | | without evidence of | | values normalize, stabilize, |
| | | | | resolution | | or return to within baseline |
| | | | | | | values. <sup>d</sup> |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; ASAP=as soon as possible; AST=aspartate aminotransferase; HCP=healthcare practitioner;

<sup>a</sup> Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug induced liver injury; ULN=upper limit of normal rash, and fever (without clear alternative cause).

<sup>b</sup> If the subject also has ≥2xULN ALP, the possibility of an indication of biliary obstruction should be discussed with the Medical Monitor.

<sup>c</sup> Details provided in Section 12.5.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist but may be a gastroenterologist.

Unless an alternative monitoring schedule is agreed by the investigator and UCB responsible physician. Determination of stabilization is at the discretion of the investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed. Confidential Acumental Applications of the Confidential Applicatio

## 12.5.1.1 Consultation with Medical Monitor and local hepatologist

Potential drug-induced liver injury events require notification of the Medical Monitor within All PDILI events require immediate action, testing, and monitoring.

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.3.1 and Table 12.3 for dot.

When IMP is discontinued, all concomitant medications and herbore eduction for medically necessary should also be discontinued. The reduction for medically necessary concomiquired concomitant medications. 24 hours (eg. by laboratory alert), and the subject must be discussed with the Medical Monitor as

#### 12.5.1.3 IMP restart/rechallenge

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, maybe fatal, and must not occur.

# Testing: identification/exclusion of alternative etiology 12.5.1.4

The measurements and additional information required for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are included but not limited to those listed in Table 12–4 (laboratory measurements) and Table 12–5 (additional information). Results of the laboratory measurements and information collected are to be submitted to the sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other assessments not included below, these additional assessments should be completed and submitted, as applicable.

All blood samples should be stored, if possible. If tests are done locally for more rapid results, a concurrent sample must also be sent to the central laboratory.

The following measurements are to be assessed (Table 12–4): This document cannot

Table 12-4: PDILI laboratory measurements

| Virology- | Hepatitis A IgM antibody |
|---|---|
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophil antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| | ALT, AST |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| Additional | Prothrombin time/INR |
| | Serum pregnancy test |
| | PK sample |

ALT=alanine aminotransferase; AST=aspartate aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody.IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

<sup>a</sup> For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

b Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause)

09 Mar 2018 AS0008

The following additional information is to be collected (Table 12–5):

# Table 12-5: PDILI information to be collected

# New or updated information

Concomitant prescription and over-the-counter medications (eg., acetaminophen, herbal remedies, vitamins); dosages and dates should be included.

Pertinent medical history, including the following:

- History of liver disease (eg, autoimmune hepatitis, nonalcoholic steatohepatitis or other "fatty liver disease")

  Adverse reactions to drugs

  Allergies

  Relevant family history or inherital.

  leficiency) deficiency)
- Recent travel
- Progression of malignancy involving the liver (Note: Metastatic disease to the liver, by itself, should not be used as an explanation for significant AST and/or ALT elevations.)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity (eg., fatigue, nausea, vomiting, right upper quadrant pain or tenderness, decreased appetite, abdominal pain, jaundice, fever, or rash)

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Alcohol and illicit drug use

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Any postmortem/pathology reports

ALT=alanine aminotransferase; AST=aspartate aminotransferase; PDILI=potential drug-induced liver injury

# Follow-up evaluation 12.5.1.5

Potential drug-induced liver injury events require follow-up monitoring as described in Table 12–3. Monitoring should continue until liver chemistry values normalize, stabilize, or return to baseline. Determination of stabilization is at the discretion of the Investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

# Other safety measurements

# 12.6.1 Vital signs

The Investigator or designee should measure all vital signs (systolic and diastolic BP, temperature [oral, axillary, or otic], pulse rate) after the subject has been sitting for at least 5 minutes, and the subject should remain seated during the measurements. Body temperature should be obtained prior to dosing with IMP at study visits when IMP is administered. At Baseline/Day 1 and Week 12, collect pulse and BP prior to drug administration and then at

09 Mar 2018 AS0008

30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing.

# 12.6.2 Body weight and height

Height is collected at Screening only. The Investigator or designee will measure the height of the subject with shoes removed in meters and the weight of the subject in kilograms. The same scale should be utilized throughout the study where possible.

# 12.6.3 Physical examination

The physical examination should be conducted by the Investigator or designee at the time points listed in Table 5–1 and will include general appearance; ear, nose, and throat; eyes, hair, and skin; respiratory; cardiovascular; GI; musculoskeletal; hepatic; neurological (including limb reflexes); and mental status. Findings considered clinically significant changes since the physical examination at the Screening Visit will be recorded as AEs.

# 12.6.4 12-lead electrocardiogram

The Investigator or designee will perform the ECG. The ECGs will be read locally.

# 12.6.5 Tuberculosis and TB risk factor assessment and management

All subjects will be assessed for TB at Screening and at the time points specified in the Schedule of Assessments (Table 5–1) through physical examination for signs and symptoms of TB, chest x-ray (Section 12.6.5.2), laboratory testing (Section 12.6.5.1), and subject questionnaire (Section 12.6.5.3).

At Screening, all subjects will have an IGRA test (QuantiFERON TB GOLD is recommended), a chest x-ray (unless already performed within 3 months of screening) and examination for signs and symptoms of TB. In addition, each subject will complete a TB questionnaire with questions directed at symptoms of TB and potential exposure to TB.

# **Exclusion Criteria at Screening**

Subjects with known TB infection, at high risk of acquiring TB infection, with LTBI\*, or current or history of NTMB infection.

- \*Subjects with LTBI may enter the study only after they have completed at least 8 weeks of appropriate prophylactic therapy and thereafter, will continue and complete the entire regimen. Following consultation with the Medical Monitor, subjects may be rescreened after completion of at least 8 weeks of LTBI prophylactic therapy.
- a. Known TB infection whether present or past is defined as:
  - Active TB infection or clinical signs and symptoms suspicious for TB (pulmonary or extra-pulmonary)
  - History of active TB infection involving any organ system or findings in other organ systems consistent with TB infection, unless adequately treated and proven to be fully recovered upon consult with a TB specialist.
  - Any evidence by radiography or other imaging modalities consistent with previously active TB infection that is not reported in the subject's medical history

- b. High risk of acquiring TB infection is defined as:
  - Known exposure to another person with active TB infection within the 3 months prior to Screening
- Latent TB infection (unless appropriate prophylaxis is initiated at least 8 weeks prior to study treatment and continued to completion of prophylaxis) is defined as:

   The absence of signs, symptoms (ie evidence of findings suggest): test results) and a chest x-ray (or other imaging) without evidence of TB infection. If the result of the IGRA test is indeterminate, the particular IGRA test previously performed may be repeated once; if positive or indeterminate on retest, the subject may not be randomized to IMP without further evaluation, treatment and discussion with Study Physician, if Latent TB infection is identified. The retest must be done during the protocol-defined Screening window.

Note: If available, respiratory or other specimens must also be smear and culture negative for TB (Centers for Disease Control [CDC] diagnosis of LTB infection) http://www.cdc.gov/TB/topic/testing/default.htm)

d. Current or history of NTMB infection despite prior or current therapy.

# Signs and Symptoms

The Investigator should consider all potential sites of infection when assessing for TB during the physical examination, and other evaluations, and based on the subject's medical or social history.

The most common primary focus of TB is the lung. Other sites may include gastrointestinal system, bone/joints, lymph glands and meninges, etc. However, in immune compromised patients and/or patients treated with TNF inhibitors, extra-pulmonary manifestations of TB are common compared to normal population.

Some common symptoms that the subject may present are dependent on the primary focus of infection and may include cough, blood in sputum, night sweats, lymphadenitis, joint pain/swelling, spinal deformity, headache/confusion, abdominal pain (mimicking inflammatory bowel disease), etc. Unusual presentations should always be considered.

Latent tuberculosis infection is defined in the "Exclusion Criteria" above. If the result of the IGRA is indeterminate, the particular IGRA previously performed may be repeated once; if positive or indeterminate on retest, the subject may not be randomized to IMP without further evaluation by a TB specialist. If LTBI or active TB is identified, subject must undergo appropriate study specified withdrawal procedures. The retest must be done during the protocoldefined Screening window. Laboratory diagnosis should be undertaken via mycobacteria culture media (or if available by preferred nucleic acid amplification test such as the Xpert mycobacterium tuberculosis [MTB] rifampin [RIF] test) and result must be negative for TB inducing pathogens.

# Test Conversion

Tuberculosis test conversion is defined as a positive IGRA result for the current test, when previous IGRA test results were negative. All subjects with TB test conversion must immediately stop IMP administration. In case of a TB test conversion, the subject must be considered as having either a suspected new latent or an active TB infection and be promptly referred to an appropriate specialist (eg. pulmonologist, infectious disease specialist) for further evaluation. If test conversion indicates LTBI, active TB, or NTMB then, per UCB TB working instructions, TB test conversion (confirmed) should be classified adequately, either as due to LTBI, active TB infection, or NTMB, respectively. Additional assessments (eg, blood tests or IGRA, chest x-rays, or other imaging) should be performed where medically relevant and documented. Such conversions should be reported to the UCB PS function.

# Latent TB

In case the evaluation by the appropriate specialist indicates a new LTBI during the study, a prophylactic TB treatment should be initiated and the IMP can be continued no sooner than 4 weeks after start of prophylactic TB treatment, if it is deemed likely by the Investigator that prophylactic TB treatment is continued to completion.

If prophylaxis is not initiated, the subject must be withdrawn,

Every related action should be discussed in advance with the Medical Monitor.

Once withdrawn from study treatment, subjects should return for the ET Visit, complete all ET Visit assessments, and complete a SFU Visit (20 weeks after the last dose of IMP).

# Active TB or NTMB infection

Subjects who develop active TB or NTMB infection during the study must be withdrawn from the study. The subject must be immediately discontinued from IMP and an ET Visit must be scheduled as soon as possible, but no later than the next scheduled visit. The subject should be encouraged to keep the SFU Visit as specified by the protocol. Treatment should be started immediately.

Note that subjects with history of NTMB or active NTMB infection are excluded from the study regardless of prior or current therapy for this condition.

# Tuberculosis assessment by IGRA 12.6.5.1

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLD is recommended) will be performed at Screening and should be repeated at Week 44, ET, and SFU Visits for all subjects. The test results will be reported as positive, negative, or indeterminate. UCB also recommends that a TB specialist be consulted where TB (latent or doubts regarding test results. If latent or active doubts regarding test results. If latent or active during Screening must be done during the protocol-defined Screening window.

12.6.5.2 Chest x-ray for tuberculosis

A plain post. active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures. The retest

A plain posteroanterior chest x-ray must be performed in the Screening Period unless one has been performed within 3 months prior to the Screening Visit. The chest x-ray (or, if done, Computed Axial Tomography of the Chest) must be clear of signs of TB infection (previous or

current) before first IMP administration. All chest imaging (particularly x-rays) should be available for review by the Investigator before randomization of the subject. The chest x-ray The chest imaging must be negative for any old or recent TB infection as determined by a qualified radiologist and/or pulmonary physician. Any new clinically significant findings must be documented in the source documents and of the questionnairs.

The questionnairs are the properties of the propert should be repeated only if the TB test was confirmed positive or any further evidence is

The questionnaire "Evaluation of signs and symptoms of tuberculosis" should be used as a source document. The questionnaire will be completed at Screening, Baseline, and at the Week 12, Week 24, Week 36, Week 48, ET, and SFU Visits. The questionnaire will assist with the identification of subjects who may require therapy for TB. A subject who answers "Yes" to the question

" at Screening is excluded. A "Yes" response to any of the other questions within the questionnaire at Screening should trigger further careful assessment to determine if subject has LTB or active TB (see Exclusion Criterion 16, Section 6.2). A "Yes" response to any of the questions during the study should trigger further assessments to determine if the subject has either LTB or active TB infection.

Subjects with a latent or active TB infection must be withdrawn from the study.

#### 12.6.5.4 **Tuberculosis management**

# LTB infection and active TB identified during study

During the study, subjects who develop evidence of LTB infection or active TB must immediately stop further administration of IMP and will be referred to an appropriate TB specialist (pulmonologist or infectious disease specialist) for further evaluation. Evidence of LTB infection is defined as subject's IGRA test converts to positive or indeterminate (and confirmed indeterminate on repeat), or the subject's questionnaire or history and physical indicates that TB infection or exposure may have occurred. Evidence of active TB includes, in addition to the aforementioned tests, signs and symptoms of organ involvement. In either situation, the subject should be carefully assessed by a TB specialist for active TB. Subjects diagnosed with active TB or LTB infection should be withdrawn from the study and receive appropriate TB or prophylaxis therapy.

If TB specialist excludes an active TB infection the subject can proceed with the IMP no earlier than 4 weeks after the start of an appropriate prophylactic therapy.

Any presumptive diagnosis or diagnosis of a TB infection is a reportable event. Confirmed active TB must be reported as an SAE. The Investigator is to complete and submit the TB follow-up Form provided.

The subject should be transferred to the care of his/her physician and managed according to the best available standard of care. Subjects identified as having converted to active TB during the

study must be withdrawn and scheduled to return for the ET Visit as soon as possible but no later than the next scheduled study visit and complete all ET Visit assessments.

lations thereof The subject should be encouraged to complete a SFU Visit (20 weeks after the last dose of IMP).

If infection with NTMB is identified during the study, the same procedure as for active TB acquired during the study must be followed.

#### 12.6.6 **Pregnancy testing**

A serum pregnancy test will be performed at Screening for all women of childbearing potential This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles and women during menopause. Natural menopause is recognized to have occurred after 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause (International Menopause Society, 2015).

A urine pregnancy test is also required at the Baseline, Week 48, ET, and at SFU visits.

A urine pregnancy test will also be performed at any study visit where there has been a delay in menses. This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles.

Pregnancy test results (serum and urine) must be negative prior to administering IMP.

## Assessment of suicidal ideation and behavior 12.6.7

Suicidal ideation and behavior will be assessed by trained study personnel using the eC-SSRS. This scale will be used to assess suicidal ideation and behavior that may occur during the study. The visits at which the eC-SSRS assessments will be performed are specified in the schedule of study assessments (Section 5.2).

The eC-SSRS is a standardized and validated instrument developed for the assessment of the severity and frequency of suicidal ideation and behavior (Posner et al., 2011; Mundt et al., 2010). Subjects respond to standardized clinical questions that are presented in a uniform fashion. The eC-SSRS defines 5 subtypes of suicidal ideation and behavior in addition to self-injurious behavior with no suicidal intent. The eC-SSRS takes approximately 3 to 10 minutes to complete.

Refer to Section 6.3 for eC-SSRS-related withdrawal criteria.

## OTHER STUDY MEASUREMENTS 13

# 13.1 Demography

The Investigator or designee will collect demographic information for all subjects according to local rules and regulations. This will include age, gender, race and ethnicity. Information on demographics will be collected according to local rules and regulations. Demographic information will be recorded in the eCRF.

# **Medical history**

nis documan. The Investigator or designee will obtain a complete medical history of AS as part of the screening assessment and include all clinically relevant past or coexisting medical conditions, responses to AS treatment as available, and surgeries. Findings will be recorded in the eCRF.

## 13.3 **Ankylosing spondylitis history**

The Investigator or designee will obtain a detailed history of AS, including the date of onset and past treatments for AS. Specific information related to AS history will be recorded in the eCRF.

As part of the medical history, the Investigator or designee will determine prior and concomitant medications and record these in the eCRF.

14 STUDY MANAGEMENT AND ADMINISTRATION

14.1 Adherence to protocol

The Investigator should not deviate from the protocol. However the Investigator in deviation for the Investigator f measure necessary in deviation from or not defined by the protocol in order to protect clinical study subjects from any immediate hazard to their health and safety. In this case, this action should be taken immediately, without prior notification of the regulatory authority, IRB/IEC, or Sponsor.

After implementation of such measure, the Investigator must notify the CPM of the Sponsor within 24 hours and follow any local regulatory requirements.

## 14.2 **Monitoring**

UCB (or designee) will monitor the study to meet the CRO's monitoring Standard Operating Procedures (SOPs), ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. Monitoring of the study may be delegated by UCB to a CRO or a contract monitor.

The Investigator and his/her staff are expected to cooperate with UCB (or designee) and to be available during the monitoring visits to answer questions sufficiently and to provide any missing information. The Investigator(s)/institution(s) will permit direct access to source data/documents for study-related monitoring, audits, IRB/IEC review, and regulatory inspection(s).

The Investigator will allow UCB (or designee) to periodically review all eCRFs and corresponding source documents (eg., hospital and laboratory records for each study participant). Monitoring visits will provide UCB (or designee) with the opportunity to evaluate the progress of the study, verify the accuracy and completeness of eCRFs, ensure that all protocol requirements, applicable authorities regulations, and Investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records.

# **Definition of source data**

All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. They should be made using some permanent form of recording (ink, typing, printing, optical disc). They should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Photocopies of CRFs are not considered acceptable source documents. Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records, ECG or other printouts, completed scales, or quality of


life questionnaires, for example. Source documents should be kept in a secure, limited access area.

Sponsor or designee will review to ensure that computerized source documents produced by the site are compliant with Food and Drug Administration (FDA) Part 11 requirements and document appropriately. Source documents that are computer generated and stored electronically must be printed for review by the monitor (eg, ECG reports). Once printed, these copies should be signed and dated by the Investigator and become a permanent part of the subject's source documents. The Investigator will facilitate the process for enabling the monitor to compare the content of the printout and the data stored in the computer to ensure all data are consistent.

Electronic data records must be saved and stored as instructed by UCB (or designee).

# 14.2.2 Source data verification

Source data verification ensures accuracy and credibility of the data obtained. During monitoring visits, reported data are reviewed with regard to being accurate, complete, and verifiable from source documents (eg, subject files, recordings from automated instruments, tracings [ECG], x-ray films, laboratory notes). All data reported on the eCRF should be supported by source documents, unless otherwise specified in Section 14.2.1.

# 14.3 Data handling

# 14.3.1 Case Report Form completion

This study will use electronic data capture (EDC); the investigator is responsible for prompt reporting of accurate, complete, and legible data in the eCRF and in all required reports.

This study will also use an electronic device (Site Tablet) to capture patient reported outcomes.

Serious AE reporting will be done using the SAE Report Form (see Section 12.2.2) while also entering the event in the appropriate eCRF section. The safety database and the clinical database will be reconciled during the study and discrepancies will be corrected as needed.

The Investigator should maintain a list of personnel authorized to enter data into the eCRF. Access to the EDC will be given after training has been received. A training certificate will be provided and filed.

Detailed instructions on the use of the EDC will be provided in the eCRF Completion Guidelines.

Corrections made after the Investigator's review and approval (by means of a password/electronic signature) will be re-approved by the Investigator. Any change or correction to the eCRF after saving must be accompanied by a reason for the change.

# 14.3.2 Database entry and reconciliation

Case Report Forms/external electronic data will be entered/loaded into a validated electronic database using a clinical data management system (CDMS). Computerized data cleaning checks will be used in addition to manual review to check for discrepancies and to ensure consistency of the data. This study is performed using EDC. The data are entered into the eCRFs once and are subsequently verified.

An electronic audit trail system will be maintained within the CDMS to track all data changes in the database once the data have been saved initially into the system or electronically loaded. Regular backups of the electronic data will be performed.

## 14.3.3 Subject Screening and Enrollment log/Subject Identification Code list

Variations thereof. The subject's screening and enrollment will be recorded in a Subject Screening and Enrollment

The Investigator will keep a Subject Identification Code list. This list remains with the Investigator and is used for unambiguous identification of each subject.

The subject's consent and enrollment in the study must be recorded in the subject's medical record. These data should identify the study and document the dates of the subject's participation.

## 14.4 Termination of the study

UCB reserves the right to temporarily suspend or prematurely discontinue this study either at a single site, multiple sites, or at all sites at any time for reasons including, but not limited to, safety or ethical issues, inaccurate or incomplete data recording, noncompliance, or unsatisfactory enrollment with respect to quality or quantity.

If the study is prematurely terminated or suspended, UCB (or its representative) will inform the investigators/institutions and the regulatory authority(ies) of the termination or suspension and the reason(s) for the termination or suspension, in accordance with applicable regulatory requirement(s). The IRB/IEC should also be informed and provided with reason(s) for the termination or suspension by the Sponsor or by the Investigator/institution, as specified by the applicable regulatory requirement(s). In addition, arrangements will be made for the return of all unused IMP and other material in accordance with UCB procedures for the study.

# 14.5 Archiving and data retention

The Investigator will maintain adequate records for the study, including eCRFs, medical records, laboratory results, Informed Consent documents, drug dispensing and disposition records, safety reports, information regarding participants who discontinued, and other pertinent data.

All essential documents are to be retained by the Investigator until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the IMP. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or by an agreement with UCB (CPMP/ICH/135/95, 2002 [Section 4.9.5]). The Investigator will contact UCB for authorization prior to the destruction of any study records or in the event of accidental loss or destruction of any study records. The Investigator will also notify UCB should he/she relocate or move the study-related files to a location other than that specified in the Sponsor's study master file.

# 14.6 **Audit and inspection**

The Investigator will permit study-related audits mandated by UCB, after reasonable notice, and inspections by domestic or foreign regulatory authorities.

The main purposes of an audit or inspection are to confirm that the rights and well-being of the subjects enrolled have been protected, that enrolled subjects (ie, signing consent and undergoing study procedures) are appropriate for the study, and that all data relevant for the evaluation of the Ine Investigator will provide direct access to all study documents, source records, and source data. If an inspection by a regulatory authority is announced, the Investigator will immediately inform UCB (or designee).

14.7 Good Clinical Practice

Noncompliance with the

Investigator, institution, institution staff, or designees of the Sponsor will lead to prompt action by UCB to secure compliance. Continued noncompliance may result in the termination of the site's involvement in the study.

#### 15 **STATISTICS**

A description of statistical methods follows and will be described in more detail in the Statistical Analysis Plan (SAP).

# Definition of analysis sets 15.1

The following analysis sets were defined:

The Enrolled Set (ES) will consist of all subjects who have given informed consent.

The Randomized Set (RS) will consist of all randomized subjects.

The Safety Set (SS) will consist of all randomized subjects who received at least 1 dose of IMP.

The Full Analysis Set (FAS) will consist of all randomized subjects who received at least 1 dose of IMP and have a valid measurement of the primary efficacy variable at Baseline.

The Per-Protocol Set (PPS) will consist of all subjects in the FAS who had no important protocol deviation affecting the primary efficacy variable. The subjects with important protocol deviations will be predefined and evaluated during a data evaluation meeting prior to unblinding of the data.

The Pharmacokinetic Per Protocol Set (PK-PPS) is a subset of the FAS, consisting of those subjects who had no important protocol deviations affecting the pharmacokinetic variables, as confirmed during ongoing data cleaning meetings prior to database lock.

The Pharmacodynamic Per Protocol Set (PD-PPS) will consist of all randomized subjects who took at least 1 dose of IMP and provide at least 1 PD measurement postdose that is without

The Dose-Blind Set (DBS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period in 1981. received at least 1 dose of the IMP during the Dose-Blind Period including the dose at Week 12.

The Escape Subject Set (ESS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period and who have not achieved an at least 10% reduction from Baseline in PGADA and total and nocturnal spinal pain at either Week 16, Week 24, or Week 36.

The Dose-Blind Responder Set (DBRS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period and who have achieved an at least 10% reduction from Baseline in PGADA and total and nocturnal spinal pain

Summary statistics will consist of frequency tables for categorical variables. For continuous variables, summary statistics will consist of number of available observations, arithmetic means SD, median, minimum, and maximum unless stated otherwise.

All statistical tests will be performed 2-sided at a 5% level.

All statistical tests will be performed 2-sided at a 5% level of significance unless stated otherwise.

Analysis of the primary efficacy variable

The primary efficacy variable will be analyzed for all subjects in the FAS.

The dose-response relationship between treatment and ASASAO an ordered categorical analysis using a non-Haenszel (Mantel and IT The dose-response relationship between treatment and ASAS40 response will be assessed with an ordered categorical analysis using a non-parametric correlation statistic of Mantel and Haenszel (Mantel and Haenszel, 1959) and modified ridit scores with the corresponding p-value. The analysis will include region and prior TNF inhibitor exposure as stratification factors. Prior TNF inhibitor exposure will be used as stratification factor as it may have an impact on efficacy. The use of region as stratification factor is intended to combine study centers in similar geographic regions. The geographic regions to be used will be defined in the IXRS and in the SAP. The correlation between dose and ASAS40 response will be evaluated at a significance level of  $\alpha$ =0.05. This evaluation of dose-response will constitute the primary efficacy analysis.

As a supportive analysis for the primary efficacy variable, a logistic regression model will be used to assess the effect of each individual dose versus placebo on ASAS40 response. The model will include fixed effects for treatment, region, and prior TNF inhibitor exposure (yes/no). If the logistic regression model is unable to converge, then region may be dropped from the model to facilitate convergence. Comparisons will be made for each dose vs placebo at a 2-sided significance level of  $\alpha$ =0.05. For each dose, the odds ratio vs placebo, the 95% confidence interval, and the corresponding p-value will be calculated.

The pairwise comparisons of bimekizumab versus placebo will be formally evaluated for statistical significance only if the primary dose response efficacy analysis is statistically significant. Once the dose response has been established, pairwise testing of each bimekizumab dose versus placebo will account for multiplicity by using a fixed sequence testing procedure with each bimekizumab dose being tested sequentially from the highest dose to the lowest dose. Each test will only be conducted if the previous test reaches significance at a 2-sided significance level of  $\alpha$ =0.05. This procedure will control the overall Type I error rate. If the dose response relationship fails to reach significance at a significance level of  $\alpha$ =0.05, then no further testing will be conducted and the pairwise comparisons are seen as nonsignificant.

Nonresponder imputation will be used to account for missing data in the primary analysis. That is, subjects with a missing ASAS40 score at Week 12 or who discontinued study treatment prior to the Week 12 visit will be considered nonresponders for the primary analysis.

## 15.3.1.1 Supportive analyses

The following supportive analyses for the primary endpoint are planned:

- 1. The primary dose-response analysis and pairwise comparisons will be repeated for all
- subjects in the RS to evaluate the consistency of the FAS with the intent-to-treat (ITT) principle. Subjects with no valid measurement of the primary efficacy variable at Baseline will be included as nonresponders.

  The primary dose response analysis and pairwise comparindividual components of the ASAGAC symptoms of the 2. The primary dose response analysis and pairwise comparisons will be repeated for all
- 3. The primary dose response analysis and pairwise comparisons will also be repeated for all symptoms of the individual components on the composite endpoint. Since all ASAS components are continuous variables (eg. change from Baseline in PGADA), and analysis of covariance (ANCOVA) with treatment, region, and prior TNF inhibitor exposure as fixed effects and the Baseline values as covariate will be used for the analysis.

Additional sensitivity analyses to evaluate the assumptions related to the handling of missing data for the primary efficacy variable will be performed and are described in Section 15.7.

#### 15.3.2 Other efficacy analyses

# Analysis of the secondary efficacy variables 15.3.2.1

The secondary efficacy variables will be analyzed for all subjects in the FAS.

All categorical variables (ie, ASAS20 response and ASAS5/6) will be analyzed for treatment effects using pairwise comparisons based on the same method as that for the primary efficacy variable.

All continuous variables (ie, ASDAS-CRP, ASDAS, BASDAI, and BASFI) will be analyzed for treatment effects using pairwise comparisons based on an analysis of covariance (ANCOVA) model with treatment, region, and biologic prior treatment as fixed effects and the Baseline value as covariate.

Pairwise testing of each bimekizumab dose versus placebo will account for multiplicity by using a fixed sequence testing procedure with each bimekizumab dose being tested sequentially from the highest dose to the lowest dose as described in Section 15.3.1.

Dose and exposure response will be assessed using a nonlinear mixed effects modeling to characterize the relationship between dose, exposure and ASAS response. The model will be partitioned into structural and stochastic models. The structural model describes the main trends and dependencies in the data, for example how drug concentrations depend on dose and time, or how ASAS response depend on drug exposure. The stochastic part of the model is further divided into the interindividual variability (IIV) and the residual unexplained variability (RUV). The IIV describes how individual specific parameters differ from the typical individual. The RUV describes the differences between the observations and the predictions from the model. Further details will be given in a separate data analysis plan and reported in a separate document.


## 15.3.2.2 Analysis of the other efficacy variables

All other efficacy variables in the Double-Blind Period will be analyzed for all subjects in the FAS. For the Dose-Blind Period, other efficacy variables will be analyzed for all subjects in the DBRS and ESS.

All categorical variables will be summarized using frequency tables by each visit.

All continuous variables will be summarized using descriptive statistics by each visit.

Time to onset of ASAS20 response and ASAS40 response will be estimated and presented using the Kaplan-Meier product-limit method for each treatment. Time to a given response will be defined as the length in days from Baseline until the first date when the response is achieved. Subjects who discontinue study treatment prior to achieving a response will be censored at the date of study treatment discontinuation. Subjects who reach the Week 12 visit without achieving a response will be censored at the date of the Week 12 visit.

The median time to response including the 2-sided 95% confidence interval will be calculated for each treatment. Between group differences (each bimekizumab dose vs placebo will be analyzed with the log-rank statistic.

All other efficacy variables will be analyzed using observed cases as treated and imputed with NRI for binary variables and multiple imputation (MI) for continuous variables (see Section 15.7).

Subjects in the ESS who discontinue with bimekizumab treatment during the Dose-Blind Period will be treated as missing and categorical/continuous variables will be imputed.

# Subgroup analyses 15.4

Subgroup analyses will be performed on the primary and secondary efficacy variables. The following variables for subgroup analyses will be defined:

- Age
- Gender
- Region
- Anti-bimekizumab antibody status
- TNF inhibitor exposure
- Concomitant synthetic DMARDs vs no concomitant synthetic DMARDs
- BASDAI (<4 [mild disease];  $\ge 4$  to  $\le 7$  [moderate disease]; >7 to  $\le 10$  [severe disease])

All subgroup analyses are based on imputed data and will be summarized using descriptive statistics only.

# This docul 15.5 Planned safety and other analyses

## 15.5.1 Safety analyses

All safety variables will be analyzed for all subjects in the SS. In addition, safety analyses during the Dose-Blind Period will be conducted on all subjects in the DBS.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA<sup>®</sup>). Adverse events will be summarized descriptively by treatment group, primary system organ class, high level term, and preferred term. Additional tables will summarize AEs

Incomment-emergent AEs will be defined as events that have a start date on or following the first administration of study treatment through the final administration of study treatment +140 days (covering the 20-week SFU Period).

Laboratory values, urinary values, ECGs. vital signal descriptively by treatment.

descriptively by treatment group.

#### 15.5.2 Other analyses

Pharmacokinetic variables will be analyzed for all subjects in the PK-PPS. Pharmacodynamic variables will be analyzed for all subjects in the PD-PPS.

Pharmacokinetic and PD analyses including the calculation of population estimates for total body clearance (CL/F) and volume of distribution (V/F) will be detailed in a separate data analysis plan and reported in a separate document. Plasma concentration-time data of bimekizumab and ASAS40 responder rates will be used as the PK and PD response. If data merits, a further PK/PD analysis on other PD variables may be performed.

Bimekizumab plasma concentrations will be summarized for each treatment at each scheduled visit.

Anti-bimekizumab antibody status will be summarized for each treatment at each scheduled

The biomarker data including IL-17A, IL-17F, IL-6, and IL-23 concentrations will be summarized for each treatment at each scheduled visit.

In addition to the PD variables, whole blood will be stored to isolate deoxyribonucleic acid (DNA) which may be used to examine genetic and epigenetic changes. Analysis will include, but not be limited to genotyping of HLA alleles (HLA Cw6, HLAB27, etc).

# Handling of protocol deviations 15.6

Important protocol deviations are deviations from the protocol which potentially could have a meaningful impact on study conduct, or on the primary efficacy, key safety, or PK/PD outcomes for an individual subject. The criteria for identifying important protocol deviations will be defined within the appropriate protocol-specific document. Important protocol deviations will be reviewed as part of the ongoing data cleaning process and all important deviations will be identified and documented prior to unblinding to confirm exclusion from analysis sets

# **15.7** Handling of dropouts or missing data

The analysis for the binary primary and secondary efficacy variables will use NRI for handling missing data. In NRI, each subject with missing data or who has discontinued double-blind study treatment prior to Week 12 will be counted as a nonresponder. Continuous secondary efficacy variables will be imputed using MI assuming that missingness is missing at random (MAR).

Two sensitivity analyses will be performed for the primary dose response analysis and for the supportive analysis (3) (Section 15.3.1.1):

1. An analysis will be performed in which all available data at Week 12 will be considered. This analysis will be based on the ordered categorical analysis to evaluate dose-response as specified in the primary analysis. However, in this case, subjects will be analyzed according to their randomized treatment, even if they discontinued prior to Week 12 and were no longer on the randomized study treatment when the assessment was performed at Week 12. Even though efforts will be made to collect the primary outcome data for all subjects at Week 12, there may still be some subjects for whom Week 12 efficacy data cannot be obtained. In this case, the subjects will be assumed to be nonresponders. The estimand here is the difference in outcome improvement at the planned endpoint for all randomized participants (Mallinckrodt, 2012). This is an estimand of effectiveness to evaluate the de facto hypothesis. It should be noted that this measures something different from the primary analysis and could be confounded by placebo subjects who withdraw and are subsequently on another active medication at the time of the Week 12 assessment. Therefore, the results of this analysis should be interpreted in the appropriate context.

An additional sensitivity analysis will be based on observed data only for subjects who are still on the initially randomized treatment at Week 12. Subjects with missing data or who have prematurely discontinued study treatment will be excluded from the analysis. The same procedure described for the primary efficacy analysis of dose response will be used.

Sensitivity analyses will also be performed for the pairwise comparisons of bimekizumab doses versus placebo based on ASAS40 response at Week 12. The following analyses will be conducted:

- 1. Missing data will be imputed using MI In MI, the missing value is replaced by a set of plausible values, where each value is a Bayesian draw from the conditional distribution of the missing data given the observed data. Intermittent missing data will be imputed using the Markov-Chain Monte Carlo [MCMC] method, followed by monotone regression for monotone missing data to evaluate the effect of the method for handling missing data on the analysis. The ASAS components will be imputed individually and then the ASAS response will be calculated using the complete datasets. The multiply imputed data sets will be analyzed using a logistic regression model with fixed effects fixed effects for treatment, region, and prior TNF inhibitor exposure. Finally, the results will be combined into a single inference using Rubin's rule (Carpenter and Kenward, 2013). This procedure assumes a MAR pattern of missingness and corresponds to an estimand of what has been called the difference in outcome improvement if all subjects tolerated or adhered to treatment (Mallinckrodt et al, 2012).
- 2. The logistic regression model will be applied where all available data at Week 12 will be considered, as described in sensitivity analysis (1) for the primary dose-response efficacy analysis.
- 3. The logistic regression model will be applied where only observed data for subjects still on the initially randomized treatment at Week 12 will be considered, as described in sensitivity analysis (2) for the primary dose-response efficacy analysis.

**UCB** 09 Mar 2018 Bimekizumab AS0008

For the dose/exposure response model, missing data will not be imputed. If a subject drops out, this will be used as a covariate in the model.

Other binary efficacy variables will be imputed using NRI and other continuous efficacy

runned interim analysis and data monitoring

There is 1 interim analysis planned for this study. The interim analysis will be performed after all enrolled subjects have completed the 12 weeks Double-Blind Period.

The objectives of this interim analysis are (i) to analysis are (i) to analysis. ASAS response criteria to determine the optimal therapeutic dose(s) for subsequent studies, and (ii) to perform a comprehensive evaluation of all double-blind data of the study.

For the interim analysis, the database will be locked and the treatment codes will be made available to UCB personnel with exception of operational staff working on the study. An interim report will be written. The investigators and subjects will remain blind to the assigned bimekizumab dosing regimen until the subject completes the Dose-Blind Period at Week 48.

Safety data will be provided to an independent DMC. The DMC will review those safety data periodically. It is not planned for the DMC to review efficacy data, and no formal stopping rules will be applied.

# Determination of sample size 15.9

A total of 285 subjects (57 in each treatment group) are planned to be randomized in this study. The primary efficacy analysis will be based on the FAS. While some randomized subjects may not be in the FAS, it is expected that this number will not impact the following calculations.

The sample size is calculated based on the ASAS40 response data from the Phase 3 studies in subjects with AS treated with secukinumab (MEASURE 1 and 2; Baeten et al, 2015). The ASAS40 response rates at Week 12 were reported to be 40% in both studies for the secukinumab 150mg dose while placebo response rates were 18% (MEASURE 1) and 9% (MEASURE 2).

Based on those ASAS40 response rates and preliminary information on the bimekizumab dose-response profile, ASAS40 response rates of 40.0%, 36.0%, 20.0%, 15.0%, and 12.0% at the end of a 12-week Treatment Period for bimekizumab 320mg, bimekizumab 160mg, bimekizumab 64mg, bimekizumab 16mg, and placebo have been assumed, respectively. Since the loading dose regimen of MEASURE 1 (iv) was different from MEASURE 2 (sc), the assumption for placebo response was based primarily on MEASURE 2, but with a weighting towards the higher placebo response rate of MEASURE 1.

2-sided test for detecting a linear trend across proportions (Nam, 1987) at a 2-sided significance level of 0.05. Assuming 57 subjects in each treatment group, the test for detecting the overall dose response based on ASAS40 response is powered at 2000/ 6 subjects with diagnosis of AS (ie. 57 subjects.) calculated using a 2-sided test for detecting a linear trend across proportions (Nam, 1987) at a

The sample size calculations were performed using the software nQuery Advisor® 7.0.

#### ETHICS AND REGULATORY REQUIREMENTS 16

#### 16.1 Informed consent

Prior to obtaining informed consent, information should be given in a language and at a level of complexity understandable to the subject in both oral and written form by the Investigator (or the Investigator).

Prior to participation in the study, the written Informed Consent Form should be signed and personally dated by the subject, or his/her legal representative, and by the person who conducted the informed consent discussion (Investigator or designee). The subject or his/her legal representative must receive a copy of the signed and dated Informed Consent Form. As part of the consent process, each subject must consent to direct access to his/her medical records for study-related monitoring, auditing, IRB/IEC review, and regulatory inspection.

If the Informed Consent Form is amended during the study, the Investigator (or the Sponsor, if applicable) must follow all applicable regulatory requirements pertaining to the approval of the amended Informed Consent Form by the IRB/IEC and use of the amended form.

All studies conducted at centers in the United States must include the use of a Health Insurance Portability and Accountability Act Authorization Form.

The subject may withdraw his/her consent to participate in the study at any time. A subject is considered as enrolled in the study when he/she has signed the Informed Consent Form. An eCRF must not be started, nor may any study specific procedure be performed for a given subject, without having obtained his/her written consent to participate in the study.

# 16.2 Subject identification cards

Upon signing the Informed Consent, the subject or legal representative will be provided with a subject identification card in the language of the subject. The Investigator will fill in the subject identifying information and medical emergency contact information. The Investigator will instruct the subject to keep the card with him/her at all times.

# 16.3 Institutional Review Boards and Independent Ethics Committees

The study will be conducted under the auspices of an IRB/IEC, as defined in local regulations, ICH-GCP, and in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

The Investigator/UCB will ensure that an appropriately constituted IRB/IEC that complies with the requirements of the current ICH-GCP version or applicable country-specific regulations will be responsible for the initial and continuing review and approval of the clinical study. Prior to initiation of the study, the Investigator/UCB will forward copies of the protocol, Informed Consent Form, IB, Investigator's curriculum vitae (if applicable), advertisement (if applicable),

and all other subject-related documents to be used for the study to the IRB/IEC for its review and approval.

Before initiating a study, the Investigator will have written and dated full approval from the

Inc investigator will also promptly report to the IRB/IEC all changes in the study, all unanticipated problems involving risks to human subjects or others, and any protocol deviations to eliminate immediate hazards to subjects.

The Investigator will not make any changes in 41 approval.

approval, except where necessary to eliminate apparent immediate hazards to the subjects. For minor changes to a previously approved protocol during the period covered by the original approval, it may be possible for the Investigator to obtain an expedited review by the IRB/IEC as allowed.

As part of the IRB/IEC requirements for continuing review of approved studies, the Investigator will be responsible for submitting periodic progress reports to the IRB/IEC (based on IRB/IEC requirements), at intervals appropriate to the degree of subject risk involved, but no less than once per year. The Investigator should provide a final report to the IRB/IEC following study completion.

UCB (or its representative) will communicate safety information to the appropriate regulatory authorities and all active investigators in accordance with applicable regulatory requirements. The appropriate IRB/IEC will also be informed by the Investigator or the Sponsor, as specified by the applicable regulatory requirements in each concerned country. Where applicable, investigators are to provide the Sponsor (or its representative) with evidence of such IRB/IEC notification.

# 16.4 Subject privacy

UCB staff (or designee) will affirm and uphold the subject's confidentiality. Throughout this study, all data forwarded to UCB (or designee) will be identified only by the subject number assigned at Screening.

The Investigator agrees that representatives of UCB, its designee, representatives of the relevant IRB/IEC, or representatives of regulatory authorities will be allowed to review that portion of the subject's primary medical records that directly concerns this study (including, but not limited to, laboratory test result reports, ECG reports, admission/discharge summaries for hospital admissions occurring during a subject's study participation, and autopsy reports for deaths occurring during the study).

# **Protocol amendments** 16.5

Protocol changes may affect the legal and ethical status of the study and may also affect the statistical evaluations of sample size and the likelihood of the study fulfilling its primary objective.

Significant changes to the protocol will only be made as an amendment to the protocol and must be approved by UCB, the IRB/IEC, and the regulatory authorities (if required), prior to being implemented.

## 17 FINANCE, INSURANCE, AND PUBLICATION

Insurance coverage will be handled according to local requirements.

Finance, insurance, and publication rights are addressed in the Investigator and/or CRO agreements, as applicable.

#### 18 REFERENCES

Baeten D, Sieper J, Braun J, Baraliakos X, Dougados M, Emery P, et al. Secukinumab, an Interleukin-17A Inhibitor, in Ankylosing Spondylitis. N Engl J Med. 2015;373:2534-48.

Variations thereof. Barkham N, Keen HI, Coates LC, O'Connor P, Hensor E, Fraser AD, et al. Clinical and imaging efficacy of infliximab in HLA-B27-Positive patients with magnetic resonance imagingdetermined early sacroiliitis. Arthritis Rheum. 2009;60:946-54.

Braun J. Axial spondyloarthritis: thoughts about nomenclature and treatment targets. Clin Exp Rheumatol. 2012;30:S132-5.

Braun J, Sieper J. Ankylosing spondylitis. Lancet. 2007;369:1379-90.

Braun J, Baraliakos X. Imaging of axial spondyloarthritis including ankylosing spondylitis. Ann Rheum Dis. 2011;70(Suppl 1):i97-103.

Braun J, Baraliakos X, Golder W, Brandt J, Rudwaleit M, Listing J, et al. Magnetic resonance imaging examinations of the spine in patients with ankylosing spondylitis, before and after successful therapy with infliximab: evaluation of a new scoring system. Arthritis Rheum. 2003;48:1126-36.

Braun J, van den Berg R, Baraliakos X, Boehm H, Burgos-Vargas R, Collantes-Estevez E, et al. 2010 update of the ASAS/EULAR recommendations for the management of ankylosing spondylitis. Ann Rheum Dis. 2011;70:896-904.

Braun J, van der Heijde D. Imaging and scoring in ankylosing spondylitis. Best Pract Res Clin Rheumatol. 2002;16:573-604.

Braun J, Zochling J, Baraliakos X, Alten R, Burmester G, Grasedyck K, et al. Efficacy of sulfasalazine in patients with inflammatory back pain due to undifferentiated spondyloarthritis and early ankylosing spondylitis: a multicentre randomised controlled trial. Ann Rheum Dis. 2006;65:1147-53.

Calin A, Garrett S, Whitelock H, Kennedy LG, O'Hea J, Mallorie P, et al. A new approach to defining functional ability in ankylosing spondylitis: the development of the Bath Ankylosing Spondylitis Functional Index. J Rheumatol. 1994:2:2281-5.

Carpenter JR, Kenward MG. Multiple imputation and its application. Chichester: John Wiley & Sons Ltd; 2013.CPMP/EWP/556/95. Points to consider on the clinical investigation of medicinal products other than NSAIDS for the treatment of RA. June 2004.

CPMP/ICH/135/95. Note for guidance on good clinical practice. July 2002.

Dauden E, Griffiths CE, Ortonne JP, Kragballe K, Molta CT, Robertson D, et al. Improvements in patient-reported outcomes in moderate-to-severe psoriasis patients receiving continuous or paused etanercept treatment over 54 weeks: the CRYSTEL study. J Eur Acad Dermatol Venereol. 2009;23(12):1374-82.

Diderichsen PM, Cox E (Quantitative Solutions BV, Breda, NL). Comparative effectiveness modeling of treatment in ankylosing spondylitis. Final Report. UCB Celltech; 2016 Feb. Project report No.: UCB-MBMA-AS-164.

Bimekizumab

Food and Drug Administration. Guidance for Industry. Drug-induced liver injury: premarketing clinical evaluation. US Dept of Health and Human Services, Center for Drug Evaluation and Research, Center for Biologics Evaluation and Research, 07/2000

Garrett S, Jenkinson T. Kenneda T C.

defining disease status in ankylosing spondylitis: the Bath Ankylosing Spondylitis Disease Activity Index. J Rheumatol. 1994;21:2286-91.

Haibel H, Brandt HC, Song IH, Brandt A, Listing J, Rudwaleit M, et al. No efficacy of subcutaneous methotrexate in active ankylosing spondylitis: a 16-week open-label trial. Ann Rheum Dis. 2007;66:419-21.

Haibel H, Rudwaleit M, Braun J, Sieper J. Six months open label trial of leflunomide in active ankylosing spondylitis. Ann Rheum Dis. 2005;64:124-6.

Haibel H. Rudwaleit M. Listing J. Heldmann F. Wong RL Kupper H. et al. Efficacy of adalimumab in the treatment of axial spondyloarthritis without radiographically defined sacroiliitis: results of a twelve-week randomized, double-blind, placebo-controlled trial by an open-label extension up to week fifty-two. Arthritis Rheum. 2008;58:1981-91.

Hays RD, Martin SA, Sesti AM, Spritzer KL Psychometric properties of the Medical Outcomes study sleep measure. Sleep Med. 2005;6:41-4.

Helmick CG, Felson DT, Lawrence RC, Gabriel S, Hirsch R, Kwoh KC, et al. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part I. Arthritis Rheum. 2008;58:15-25.

Heuft-Dorenbosch L, Spoorenberg A, van Tubergen A, Landewé R, van der Tempel H, Mielants H, et al. Assessment of enthesitis in ankylosing spondylitis. Ann Rheum Dis. 2003;62:127-32.

International Menopause Society. Cornwall, UK: Menopause Terminology; c2015. http://www.imsociety.org/menopause\_terminology.php. Accessed 25 Jan 2016.

Ivanov II, Frutos Rde L, Manel N, Yoshinaga K, Rifkin DB, Sartor RB, et al. Specific microbiota direct the differentiation of IL-17-producing T-helper cells in the mucosa of the small intestine. Cell Host Microbe. 2008;4:337–49.

Langley RG, Feldman SR, Han C, Schenkel B, Szapary P, Hsu MC, et al. Ustekinumab significantly improves symptoms of anxiety, depression, and skin-related quality of life in patients with moderate-to-severe psoriasis: Results from a randomized, double-blind, placebocontrolled phase III trial. J Am Acad Dermatol. 2010;63(3):457-65.

Lukas C, Braun J, van der Heijde D, Hermann K-G A, Rudwaleit M, Ostergaard M, et al. Scoring inflammatory activity of the spine by magnetic resonance imaging in ankylosing spondylitis: a multireader experiment. J of Rheum. 2007;34:862-70.

Lukas C, Landewé R, Sieper J, Dougados M, Davis J, Braun J, et al. Development of an ASAS-endorsed disease activity score (ASDAS) in patients with ankylosing spondylitis. Ann Rheum Dis. 2009;68:18-24.

riations thereof. Mantel N, Haenszel W. Statistical aspects of the Analysis of Data From Retrospective Studies of Disease. J Natl Cancer Inst. 1959; 22:719-48.

Maruish ME, editor. User's manual for the SF-36v2 Health Survey. 3rd ed. Lincoln, RI: QualityMetric Incorporated; 2011.

Mundt JC, Greist JH, Gelenberg AJ, Katzelnick DJ, Jefferson JW, Modell JG. Feasibility and Validation of a Computer-Automated Columbia-Suicide severity Rating Scale Using Interactive Voice Response Technology. J Psychiatr Res. 2010;44(16):1224-8.

Myasoedova E, Crowson CS, Kremers HM, Therneau TM, Gabriel SE. Is the incidence of rheumatoid arthritis rising?: results from Olmsted County, Minnesota, 1955-2007. Arthritis Rheum. 2010;62:1576-82.

Nam, JM. A simple approximation for calculating sample sizes for detecting linear trend in proportions. Biometrics. 1987;43(3):701-5.

National Research Council Panel on Handling Missing Data in Clinical Trials. The prevention and treatment of missing data in clinical trials. Washington DC: National Academies Press. 2010. Ogdie A, Weiss P. The Epidemiology of Psoriatic Arthritis. Rheum Dis Clin North Am. 2015;41(4):545-68.

Pavy S, Brophy S, Calin A. Establishment of the minimum clinically important difference for the bath ankylosing spondylitis indices: a prospective study. J Rheumatol. 2005;32:80-5.

Pedersen SJ, Poddubmyy D, Sorensen IJ, Loft A-G, Hindrup JS, Thamsborg G, et al. Course of Magnetic Resonance Imaging-Detected Inflammation and Structural Lesions in the Sacroiliac Joints of Patients in the Randomized, Double-Blind, Placebo-Controlled Danish Multicenter Study of Adalimumab in Spondyloarthritis, as Assessed by the Berlin and Spondyloarthritis Research Consortium of Canada Methods. Arthritis and Rheumatology. 2016;68:418-29.

Poddubnyy D. Axial spondyloarthritis: is there a treatment of choice? Ther Adv Musculoskelet Dis. 2013;5:45-54.

Poddubnyv D, Rudwaleit M, Haibel H, Listing J, Märker-Hermann E, Zeidler H, et al. Effect of non-steroidal anti-inflammatory drugs on radiographic spinal progression in patients with axial spondyloarthritis: results from the German Spondyloarthritis Inception Cohort. Ann Rheum Dis. 2012;71:1616-22.

Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oguendo MA, et al. The Columbia-Suicide Severity Rating Scale: Initial Validity and Internal Consistency Findings From Three Multisite Studies With Adolescents and Adults. Am J Psychiatry. 2011;168(12):1266-77.

Reveille JD, Witter JP, Weisman MH. Prevalence of axial spondyloarthritis in the United States: estimates from a cross-sectional survey. Arthritis Care Res (Hoboken). 2012;64:905-10.

Rudwaleit M. New approaches to diagnosis and classification of axial and peripheral spondyloarthritis. Curr Opin Rheumatol. 2010;22:375-80.

Rudwaleit M, Haibel H, Baraliakos X, Listing J, Märker-Hermann E, Zeidler H, et al. The early disease stage in axial spondylarthritis: results from the German Spondyloarthritis Inception Cohort. Arthritis Rheum. 2009a;60:717-27.

Bimekizumab

Rudwaleit M, van der Heijde D, Landewe R, Akkoc N, Brandt J, Chou CT, et al. The Assessment of SpondyloArthritis International Society classification criteria for peripheral spondyloarthritis and for spondyloarthritis in general. Ann Rheum Dis. 2011:70:25-31.

Rudwaleit M, Landewé R, van der Heijde D, Listing J, Brandt J, Braun J, et al. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part I): classification of paper patients by expert opinion including uncertainty appraisal. Ann Rheum Dis. 2009b;68:770-6.

Sieper J, Rudwaleit M, Baraliakos X, Brandt J, Braun J, Burgos-Vargas R, et al. The Assessment of SpondyloArthritis International Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009;68(Supple 2):ii1-44.

Snaith RP, Zigmond AS. The hospital anxiety and depression scale, with the irritabilitydepression-anxiety scale and the Leeds situational anxiety scale manual. 1994.

Woodworth T, Furst DE, Alten R, Bingham C, Yocum D, Sloan V, et al. Standardizing assessment and reporting of adverse effects in rheumatology clinical trials II: the Rheumatology Common Toxicity Criteria v.2.0. J Rheumatol. 2007;34:1401-14.

van der Heijde D, Dougados M, Davis J, Weisman MH, Maksymowych W, Braun J, et al. Assessment in Ankylosing Spondylitis International Working Group/Spondylitis Association of America recommendations for conducting clinical trials in ankylosing spondylitis. Arthritis Rheum. 2005;52:386-94.

van der Heijde D, Schiff MH, Sieper J, Kivitz AJ, Wong RL, Kupper H, et al. Adalimumab effectiveness for the treatment of ankylosing spondylitis is maintained for up to 2 years: long-term results from the ATLAS trial. Ann Rheum Dis. 2009;68:922-9.

van Tubergen A, Black PM, Coteur G. Are patient-reported outcome instruments for ankylosing spondylitis fit-for-purpose for the axial spondyloarthritis patient? A Qualitative and Psychometric Analysis. Rheum. 2015;54:1842-51.

van Tubergen A, Debats I, Ryser L, Londoño J, Burgos-Vargas R, Cardiel MH, et al. Use of a numerical rating scale as an answer modality in ankylosing spondylitis-specific questionnaires. Arthritis Rheum, 2002a;47:242-8.

van Tubergen A, Coenen J, Landewé R, Spoorenberg A, Chorus A, Boonen A, et al. Assessment of fatigue in patients with ankylosing spondylitis: a psychometric analysis. Arthritis Rheum. 2002b;47:8-16.

Ware JE, Kosinski M, Keller SD. SF-36 Physical and Mental Health Summary scales: a user's

ware JE, Kosi manual; 1994. Wells Wells G, Li T, Maxwell L, MacLean R, Tugwell P. Determining the minimal clinically important differences in activity, fatigue, and sleep quality in patients with rheumatoid arthritis. J Rheumatol. 2007;34:280-9.

#### 19 **APPENDICES**

## 19.1 Modified New York (mNY) Classification Criteria for AS

# Table 19–1: Modified New York (mNY) Classification Criteria for AS

# **Diagnosis**

Clinical criteria:

- a. Low back pain and stiffness for more than 3 months which improves with exercise, but is not relieved by rest
- b. Limitation of motion of the lumbar spine in both the sagittal and frontal planes.
- Limitation of chest expansion relative to normal values corrected for age and

Radiologic criterion:

Sacroiliitis grade ≥2 bilaterally or grade 3 to 4 unilaterally

# Grading

Definite ankylosing spondylitis if the radiologic criterion is associated with at least 1 clinical criterion

AS=ankylosing spondylitis; mNY=modified New York Criteria

w York Consing spondylitis Note: A second grading of "probable ankylosing spondylitis" is part of the modified NY criteria, but it is not

# Markedly abnormal laboratory values 19.2

Table 19-2: Definitions of markedly abnormal hematology values

| | Markedly Abno | ormal Definition |
|---|---|---|
| Parameter (RCTC units) | Low | High |
| Hemoglobin (g/dL) | <lln< td=""><td>N/A valialio</td></lln<> | N/A valialio |
| | AND | iarito |
| | >2.0 decrease from baseline | oi 7° |
| Hemoglobin (g/dL) | <8.0 | N/A |
| Leukocytes (total x 1000) | <2.0 | NA |
| Lymphocytes (x 1000) | <0.5 | et N/A |
| Neutrophils (x 1000) | <1.0 | N/A |
| Platelets (x 1000) | <50 | N/A |

LLN=lower limit of normal; N/A = Not Applicable; RCTC=Rheumatology Common Toxicity Criteria Data source: modified from Appendix Rheumatology Common Toxicity Criteria v.2.0 presented in Woodworth et al, 2007

Table 19–3: Definitions of markedly apnormal biochemistry values

| Parameter (RCTC units) | Low | High |
|---|---|---|
| Alkaline Phosphatase | N/A | >3 x ULN |
| ALT | N/A | >3 x ULN |
| AST | N/A | >3 x ULN |
| Calcium (mg/dL) | <7.0 | >12.5 |
| Creatinine (mg/dL) | N/A | >1.8 x ULN |
| Glucose (mg/dL) | <40 | >250 |
| Potassium (mmol/L) | <3.0 | >6.4 |
| Sodium (mmol/L) | <125 | N/A |
| Total bilirubin | N/A | ≥2 x ULN |
| Uric acid | N/A | ≥3 x ULN |
| ALT=alanine aminotransferase; AST=aspa<br>Common Toxicity Criteria; ULN=upper | | plicable; RCTC=Rheumatolo |

<sup>&</sup>lt;sup>a</sup> Withdrawal criteria for neutrophils is <0.5 (Section 6.3).

#### 19.3 **Protocol Amendment 1**

# Rationale for the amendment

The purpose of this protocol amendment is the following:

- The extra-articular manifestations variable was removed from the other efficacy variables, as these will be assessed as AEs. In addition, the other objective regarding extra-articular manifestations was updated to be specific to enthesition.
- The number of subjects to be included in the imaging evaluation was increased from 10 subjects to 20 subjects at Baseline. The MRIs at Weeks 12 and 48 will be performed only for subjects who were classified as MRI-positive as per ASAS-OMERACT Criteria at Baseline. An MRI can be used to visualize inflammation in the SI joints and spine in addition to structural lesions. Inflammation of the SI joints and spine is a key feature of AS that is potentially amenable to treatment with bimekizumab. It is expected that reduction in inflammation in the SI joints and spine in MRI-positive subjects at Baseline can be detected within the 48-week Treatment Period. This effect can not be demonstrated for subjects who are MRI-negative at Baseline. Thus, MRI-negative subjects are excluded from the substudy.
- A clarification that MRI assessments will occur at the Baseline Visit was added to all relevant sections.
- Criteria for the definition of AE intensity were added in response to a regulatory agency
- All study variables have been rearranged for clarification reasons.

In addition, minor typographical errors were corrected.

# Modifications and changes

# Global change #1

Abbreviations within the protocol and in the list of abbreviations have been adjusted as needed.

# Global change #2

The following global change was made for all visits from Week 4 (Section 8.3.3) through Week 44 (Section 8.4.8).

Collect pulse and BP once after dosing (any time).

# Has been changed to:

Collect pulse and BP once after dosing (any time).
# Global change #3

**UCB** 

The following appendices and respective in-text references have been removed from the protocol.

- Section 19.3: PGADA (NRS)
- Section 19.4: Total spinal pain NRS and nocturnal spinal pain NRS
- Section 19.5: Bath Ankylosing Spondylitis Functional Index (BASFI)
- Section 19.6: Bath Ankylosing Disease Activity Index (BASDAI)
- Section 19.7: Lateral spinal flexion
- Section 19.8: BASMI linear function
- Section 19.9: ShortForm (SF36) Questionnaire
- Section 19.10: MOS Sleep Scale Questionnaire
- Section 19.11: ASQoL
- Section 19.12: Tuberculosis Questionnaire

### **Specific changes**

### Change #1

### **Original text:**

Serious adverse event reporting

| bal change a | <del>*</del> #3 |
|---|---|
| following appearance. | ollowing appendices and respective in-text references have been removed from the col. |
| ection 19.3: PC | GADA (NRS) |
| Section 19.4: To | otal spinal pain NRS and nocturnal spinal pain NRS |
| Section 19.5: Ba | nth Ankylosing Spondylitis Functional Index (BASFI) |
| ection 19.6: Ba | ath Ankylosing Disease Activity Index (BASDAI) |
| ection 19.7: La | iteral spinal flexion |
| Section 19.8: BA | ASMI – linear function |
| ection 19.9: Sh | nortForm (SF36) Questionnaire |
| Section 19.10: N | MOS Sleep Scale Questionnaire |
| Section 19.11: A | ASQoL |
| Section 19.12: T | Suberculosis Questionnaire |
| following appendices and respective in-text references have been removed from the col. ection 19.3: PGADA (NRS) ection 19.4: Total spinal pain NRS and nocturnal spinal pain NRS ection 19.5: Bath Ankylosing Spondylitis Functional Index (BASFI) ection 19.6: Bath Ankylosing Disease Activity Index (BASDAI) ection 19.7: Lateral spinal flexion ection 19.8: BASMI – linear function ection 19.9: ShortForm (SF36) Questionnaire ection 19.10: MOS Sleep Scale Questionnaire ection 19.11: ASQoL ection 19.12: Tuberculosis Questionnaire cific changes nge #1 inal text: bus adverse event reporting Serious adverse event reporting (24h) | |
| | Serious adverse event reporting (24h) |
| Fax | Europe and Rest of the World: +32 2 386 2421 |
| | USA: +1 800 880 6949<br>or +1 866 890 3175 |
| δ | Canada: +1 877 582 8842 |
| Email | Global: DS_ICT@ucb.com |
| X T | |

# Has been changed to:

| паѕ | been changed to: | |
|---|---|---|
| agric's | | Serious adverse event reporting (24h) |
| 40CUMI | Fax | Europe and Rest of the World: +32 2 386 2421 |
| Nis | | USA and Canada: +1 800 880 6949 or +1 866 890 3175 |
| \'\'\' | Email | Global: DS_ICT@ucb.com |



### Change #2

### **Section 1 Summary**

### Original text:

The secondary objectives of the study are to assess the efficacy of the individual dose regimens of bimekizumab compared to placebo, safety and tolerability, PK, PD, immunogenicity, and the exposure:response relationship of bimekizumab as it relates to efficacy and safety. The secondary efficacy variables include: Change from Baseline in Ankylosing Spondylitis Disease Activity Score C reactive protein (ASDAS-CRP), Assessment in Axial SpondyloArthritis International Society 20% response criteria (ASAS20) response, Assessment in Axial SpondyloArthritis International Society 5 out of 6 response criteria (ASAS5/6) response, Change from Baseline in BASDAI, and Change from Baseline in BASFI, all at Week 12, Safety variables include incidence of adverse events (AEs) and serious adverse events (SAEs), withdrawal due to AEs, change from Baseline in vital signs, body weight, physical examination, ECG, and clinical laboratory variables.

Other objectives are to assess the impact on patient-reported quality of life (fatigue, sleep, and pain), extra-articular disease manifestations (uveitis, inflammatory bowel disease [IBD], and psoriasis), the impact of administration of bimekizumab on biological pathways relating to disease biology and response to therapy via candidate biomarker analysis and to enable genomic and proteomic analysis of subject samples and evaluation of the potential for subject stratification approaches, and to assess the impact of bimekizumab on inflammatory changes in the spine and sacroiliac (SI) joint using magnetic resonance imaging (MRI) in a subset of subjects (approximately 10 subjects per treatment arm).

# Has been changed to:

The secondary objectives of the study are to assess the efficacy of the individual dose regimens of bimekizumab compared to placebo, safety and tolerability, PK, PD, immunogenicity, and the exposure:response relationship of bimekizumab as it relates to efficacy and safety. The secondary efficacy variables include: Change from Baseline in Ankylosing Spondylitis Disease Activity Score C-reactive protein (ASDAS-CRP), Assessment in Axial SpondyloArthritis International Society 20% response criteria (ASAS20) response, Assessment in Axial SpondyloArthritis International Society 5 out of 6 response criteria (ASAS5/6) response, Change from Baseline in BASDAI, and Change from Baseline in BASFI, all at Week 12. Safety variables include incidence of adverse events (AEs), serious adverse events (SAEs), and withdrawal due to AEs as secondary safety variables and change from Baseline in vital signs, body weight, physical examination, ECG, and clinical laboratory variables as other safety variables.

Other objectives are to assess the impact on patient-reported quality of life (fatigue, sleep, and pain), extra articular disease manifestations (uveitis, inflammatory bowel disease [IBD], and psoriasis), the impact of administration of bimekizumab on biological pathways relating to disease biology and response to therapy via candidate biomarker analysis, and to enable genomic and proteomic analysis of subject samples and evaluation of the potential for subject stratification approaches, and to assess the impact of bimekizumab on inflammatory changes in the spine and sacroiliac (SI) joint using magnetic resonance imaging (MRI) in a subset of subjects (approximately 10 subjects per treatment arm at Baseline).

### Change #3

### Section 2.1.1 Clinical studies

### **Original text:**

Three clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque psoriasis, RA0124 in 30 healthy volunteers, and PA0007 in 53 subjects with PsA.

### Has been changed to:

**Four** clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque psoriasis, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, and UP0031 in 12 healthy volunteers.

### Change #4

### **Section 2.1.1 Clinical studies**

# The following text has been added:

UP0031 was a Phase 1, open-label, parallel-group, randomized, single-dose study to evaluate the BA, PK, and tolerability of 2 different formulations of bimekizumab in healthy subjects. There were no treatment-emergent adverse events (TEAEs) leading to discontinuation, and no SAEs or fatalities were reported.

### Change #5

### Section 2.1.1 Clinical studies

### Original text:

Two additional studies of bimekizumab are ongoing. RA0123 is a Phase 2a, double-blind, randomized, placebo-controlled, multiple dose study to evaluate the safety, PK, PD, and efficacy of multiple doses of bimekizumab administered as add-on therapy to stable certolizumab pegol (CZP; Cimzia®) therapy in subjects with moderate to severe RA. UP0031 is an open-label, parallel-group, single-dose study designed to evaluate the relative bioavailability and tolerability of 2 dose levels of UCB4940 (bimekizumab) given as 2 x80mg or 1x 160mg given via sc injection in healthy subjects.

### Has been changed to:

One additional study of bimekizumab is ongoing. RA0123 is a Phase 2a, double-blind, Aty ons there of variations there of or variations of variations. randomized, placebo-controlled, multiple dose study to evaluate the safety, PK, PD, and efficacy of multiple doses of bimekizumab administered as add-on therapy to stable certolizumab pegol (CZP; Cimzia<sup>®</sup>) therapy in subjects with moderate to severe RA. <del>UP0031 is an open label,</del> parallel group, single dose study designed to evaluate the relative bioavailability and tolerability of 2 dose levels of UCB4940 (bimekizumab) given as 2 x80mg or 1x 160mg given via sc injection in healthy subjects.

### Change #6

### Section 3.3 Other objectives

### Original text:

To assess extra-articular disease manifestations (enthesitis, uveitis, inflammatory bowel disease, and psoriasis)

### Has been changed to:

To assess the impact on extra articular disease manifestations (enthesitis, uveitis, inflammatory bowel disease, and psoriasis) enthesitis

### Change #7

**Section 4 Study Variables** 

### **Original text:**

- 4 STUDY VARIABLES
- 4.1 Efficacy variable(s)

### 4.1.1 Primary efficacy variable

The primary efficacy variable for this study is as follows:

• ASAS40 response at Week 12

# 4.1.2 Secondary efficacy variables

The secondary efficacy variables for this study are as follows:

- Change from Baseline in ASDAS-CRP at Week 12
- ASAS20 response at Week 12
- ASAS5/6 response at Week 12
- Change from Baseline in BASDAI at Week 12
- Change from Baseline in BASFI at Week 12

### 4.1.3 Other efficacy variables

extensions of Variations thereof. Other efficacy variables will be assessed as specified in Table 5–1 (analyses at all time points not specified in Section 4.1.1 or Section 4.2.1 are exploratory):

- ASAS40 response
- Time to ASAS40 response
- Change from Baseline in ASDAS-CRP
- ASDAS status (eg, inactive disease, moderate, high and very high disease activity)
- ASAS20 response
- Time to ASAS20 response
- ASAS5/6 response
- Ankylosing Spondylitis Disease Activity Score major improvement (ASDAS-MI)
- ASAS partial remission
- Change from Baseline in BASDAI
- Change from Baseline in BASFI
- Change from Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
- Occurrence of extra-articular manifestations
  - Uveitis flares (as determined by an ophthalmologist or other eye specialist, as appropriate)
  - Inflammatory bowel disease flares (as determined by a gastroenterologist, as appropriate)
  - Psoriasis disease activity
- Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index
- Physician's Global Assessment of Disease Activity (PhGADA)
- Change from Baseline in Patient's Global Assessment of Disease Activity (PGADA)
- Change from Baseline in total and nocturnal spinal pain (NRS)
- Change from Baseline in the average of Questions 5 and 6 of the BASDAI



Change from Baseline in Sleep quality (Medical Outcomes Study [MOS]-12 item scale)

Change from Baseline in Ankylosing Spondylitis Quality of Life (ASQoL)

- Change from Baseline in:
  - Spondyloarthritis Research Consortium of Canada (SPARCC) MRI index for Assessment of Spinal Inflammation in AS, and
- Change from Baseline in Hospital Anxiety and Depression Scale Anxiety (HADS-A) and Hospital Anxiety and Depression (HADS-D) scores

  Percentage of subjects with scores below 8 in HADSscores)

### 4.2 PK and PD variables

### 4.2.1 PK variables

The PK variables are plasma concentrations of bimekizumab, total body clearance (CL/F), and volume of distribution (V/F)

### 4.2.2 PD variables

The PD variables are concentrations of cytokines of relevance to the IL-17A/F signaling pathway and AS biology, and include but are not limited to IL-17A, IL-17F, IL-23, IL-6, and TNFα

### 4.3 Pharmacogenomic variables

### 4.3.1 Genomic, proteomic, and metabolite variables

Where local regulations permit, additional blood samples will be collected from consenting subjects at specific time points and stored at -80°C for up to 20 years to allow for potential, exploratory analyses of genomic, genetic, proteomic, and metabolomic biomarkers relevant to disease biology and progression, response to therapy, and the inflammatory and immune response processes.

# 4.4 Immunological variables

Immunological variables allow evaluation of immunogenicity as well as immunological biomarkers.

- Anti-bimekizumab antibody detection prior to and following study treatment
- Serum complement concentrations.
- Flow cytometry analysis of key immune cell populations, including but not limited to CD3, CD19, CD4, CD8, and CD69 (using fluorescence activated cell sorting).
- Cytokines and other exploratory markers

### 4.5 Safety variables

Safety variables to be assessed as specified in Table 5–1 are as follows:

- Standard 12-lead electrocardiogram (ECG) intervals (RR, PR, QRS, QT, and QT intervals corrected for heart rate using Bazett's and Fridericia's formulas [QTcB and QTcF]). including changes from Baseline Electrocardiogram (ECG) variables.

  Change from Baseline in clinical labor urinalysis)
- 4.1.1 Primary efficacy variable
  The primary efficacy variable for this study is as follows:
  ASAS40 response at Week 12
  4.2 Secondary variables
  1.2.1 Secondary efficacy variables
  Change from Baseline in ASD

  ASAS20 response ASAS20 response ASAS20 response at Meek 12

- ASAS20 response at Week 12
- ASAS5/6 response at Week 12
- Change from Baseline in BASDAI at Week 12
- In Bi Change from Baseline in BASFI at Week 12

### 4.2.2 Secondary safety variables

Assessment time points for safety variables are specified in Table 5–1. Variables are as follows:

- Incidence of AEs and SAEs
- Withdrawal due to AEs

### 4.3 Other variables

### 4.3.1 Other efficacy variables

Assessment time points for the other efficacy variables are specified in Table 5–1 (analyses at all time points not specified in Section 4.1.1 or Section 4.2.1 are exploratory). Variables are as follows:

- ASAS40 response
- Time to ASAS40 response
- Change from Baseline in ASDAS-CRP
- ASDAS status (eg, inactive disease, moderate, high and very high disease activity)

- ASAS20 response
  Time to ASAS20 response
  ASAS5/6 response
  Ankylosing Spondylitis Disease Activity Score major improvement (ASDAS-MI)
- ASAS partial remission
- Change from Baseline in BASD
- Change from Baseline in BASEI
- Change from Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
- Occurrence of extra articular manifestations
  - Uveitis flares (as determined by an ophthalmologist or other eye specialist, as appropriate)
  - Inflammatory bowel disease flares (as determined by a gastroenterologist, as appropriate)
  - Psoriasis disease activity
- Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index
- Physician's Global Assessment of Disease Activity (PhGADA)
- Change from Baseline in Patient's Global Assessment of Disease Activity (PGADA)
- Change from Baseline in total and nocturnal spinal pain (NRS)
- Change from Baseline in the average of Questions 5 and 6 of the BASDAI

- Change from Baseline in Physical Component Summary (PCS) and Mental Component Summary (MCS) of the SF-36 (Short-Form 36-Item Health Survey)
- Change from Baseline in Sleep quality (Medical Outcomes Study [MOS]-12 item scale)
- Change from Baseline in Ankylosing Spondylitis Quality of Life (ASQoL)
- Change from Baseline in:
- Spondyloarthritis Research Consortium of Canada (SPARCC) MRI index for Assessment of Spinal Inflammation in AS, and

  Ankylosing Spondylitis spine MRI- activity (ASeria Prosecute)
  - Ankylosing Spondylitis spine MRI- activity (ASspiMRI-a) in the Berlin modification
- Change from Baseline in Hospital Anxiety and Depression Scale Anxiety (HADS-A) and Hospital Anxiety and Depression Scale - Depression (HADS-D) scores
- Percentage of subjects with scores below 8 in HADS-A and HADS-D subjects with normal scores)

### 4.3.2 Other safety variables

Assessment time points for other safety variables are specified in Table 5–1. Variables are as follows:

- Change from Baseline in vital signs (blood pressure, pulse rate) and body weight
- Standard 12-lead electrocardiogram (ECG) intervals (RR, PR, QRS, QT, and QT intervals corrected for heart rate using Bazett's and Fridericia's formulas [OTcB and OTcF]). including changes from Baseline Electrocardiogram (ECG) variables
- Change from Baseline in clinical laboratory variables (hematology, biochemistry, and urinalysis)

### 4.3.3 Other PK and PD variables

- The PK variables are plasma concentrations of bimekizumab, total body clearance (CL/F), and volume of distribution (V/F).
- The PD variables are concentrations of cytokines of relevance to the IL-17A/F signaling pathway and AS biology, and include but are not limited to IL-17A, IL-17F, IL-23, IL-6, and TNFα.

# 4.3.4 Other immunological variables

Immunological variables allow evaluation of immunogenicity as well as immunological biomarkers.

Anti-bimekizumab antibody detection prior to and following study treatment

- Serum complement concentrations.
- Flow cytometry analysis of key immune cell populations, including but not limited to CD3, CD19, CD4, CD8, and CD69 (using fluorescence activated cell sorting).
- Cytokines and other exploratory markers

### 4.3.5 Other pharmacogenomic, proteomic, and metabolite variables

Where local regulations permit, additional blood samples will be collected from consenting isions or variations thereof subjects at specific time points and stored at -80°C for up to 20 years to allow for potential, exploratory analyses of genomic, genetic, proteomic, and metabolomic biomarkers relevant to disease biology and progression, response to therapy, and the inflammatory and immune response processes.

### Change #8

### Section 5.1.2 Double-Blind Period

### Original text:

At Baseline/Day 1, subjects will be randomized 1:1:1:1:1 (stratified by region and prior TNF) inhibitor exposure) to receive the following blinded IMP treatment regimens at the clinical site. The enrollment of TNF inhibitor-experienced subjects will be limited to approximately 30% of the total study population. Therefore, each arm will have approximately 8 TNF inhibitor experienced subjects in a total of 57 subjects per arm.

### Has been changed to:

At Baseline/Day 1, subjects will be randomized 1:1:1.1:1 (stratified by region and prior TNF inhibitor exposure) to receive the following blinded IMP treatment regimens at the clinical site. The enrollment of TNF inhibitor-experienced subjects will be limited to approximately 30% of the total study population. Therefore, each arm will have approximately 18 TNF inhibitor experienced subjects in a total of 57 subjects per arm.

### Change #9

# Section 5.1.7 Radiographic evaluation

# **Original text:**

# 5.1.7 Radiographic evaluation

In a subpopulation of A\$0008, MRIs of the spine and SI joints will be performed in approximately 10 subjects per treatment arm at Baseline, Week 12, and Week 48. Analyses will be exploratory in nature and will be performed at selected sites.

# Has been changed to:

# 5.1.7 Imaging evaluation

In a subpopulation of AS0008, MRIs of the spine and SI joints will be performed in approximately 20 subjects per treatment arm at Baseline. Magnetic resonance imaging at Week 12 and Week 48 will be performed only for subjects who are MRI-positive at Baseline based on an ASAS-Outcome Measures in Rheumatology Clinical Trials (OMERACT) assessment. The Baseline MRI should be performed after confirmation of eligibility for the study based on screening assessments and before the first bimekizumab injection. Magnetic resonance imaging at Week 12 and Week 48 should be performed as close to the Week 12/Week 48 Visit as possible. Further details are provided in Section 9.15. Analyses will be exploratory in nature and will be performed at selected sites.

### Change #10

### Section 5.2 Table 5-1, footnote d

### **Original text:**

<sup>d</sup> At Baseline/Day 1 and Week 1, collect pulse and BP prior to drug administration and then at 30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing (any time). All other procedures are done prior to dosing.

### Has been changed to:

d At Baseline/Day 1 and Week **12**, collect pulse and BP prior to drug administration and then at 30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing (any time). All other procedures are done prior to dosing.

### Change #11

### Section 5.2 Table 5-1, footnote n and p

### **Original text:**

- <sup>n</sup> An MRI of the spine and sacroiliac joints will be performed in a subpopulation of approximately 10 subjects per treatment arm for exploratory purposes at Screening, Week 12, and Week 48. The MRI will be read centrally.
- <sup>p</sup> The minimum time between doses during the Double-Blind Period should be no less than 26 days and no more than 30 days and during the Dose-Blind Period should be no less than 24 days and no more than 32 days.

### Has been changed to:

- An MRI of the spine and sacroiliac joints will be performed in a substudy with approximately 20 subjects per treatment arm at Screening Baseline. A central reader will assess Baseline MRIs to identify MRI-positive subjects as per the ASAS-Outcome Measures in Rheumatology Clinical Trials (OMERACT) criteria. An MRI at Week 12 and Week 48 will be performed for those subjects who were MRI-positive at Baseline. The Baseline MRI should be performed after confirmation of eligibility based on screening assessments for the study and before the first bimekizumab injection. Magnetic resonance imaging at Week 12 and Week 48 should be performed as close to the Week 12/Week 48 Visit as possible. For logistical reasons, it may not be possible to schedule the MRIs at the actual visit date and an additional visit for the MRI may be required.
- P The minimum time between closes during the Double-Blind Period should be no less than 25 days and no more than 31 days and during the Dose-Blind Period should be no less than 24 days and no more than 32 days.

### Change #12

### Section 6.2 Inclusion criterion 11

### **Original text:**

11. Subjects taking sulfasalazine (up to 3mg/day) or hydroxychloroquine (up to 400mg per day total) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomization. Dose and dosing schedule should remain stable up to Week 16.

### Has been changed to:

11. Subjects taking sulfasalazine (up to 3mg/day) or hydroxychloroquine (up to 400mg per day total) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomization. Dose and dosing schedule should remain stable up to Week 16

### Change #13

### Section 6.2, Inclusion criterion 12

### **Original text:**

- 12. Subjects may be TNF inhibitor-naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:
  - experienced an inadequate response to previous treatment given for at least 3 months
  - been intolerant to administration (eg, had a side effect/AE that led to discontinuation)
  - lost access to TNF inhibitor for other reasons

# Has been changed to:

- 12. Subjects may be TNF inhibitor-naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:
  - experienced an inadequate response to previous treatment given for at least 3 months
     12 weeks
  - been intolerant to administration (eg, had a side effect/AE that led to discontinuation)
  - lost access to TNF inhibitor for other reasons

# Change #14

### Section 6.2 Exclusion criterion 3

# Original text:

3. Subjects participating in another study of a medication or a medical device under investigation within the last 3 months or at least 5 half-lives whichever is greater.

### Has been changed to:

3. Subjects participating in another study of a medication or a medical device under variations thereof investigation within the last 3 months 12 weeks or at least 5 half-lives whichever is greater.

### Change #15

### Section 6.2 Exclusion criterion 10

### Original text:

10. Subjects with known history of or current clinically active infection with Histoplasma. Coccidiodes, Paracoccidioides, Pneumocystis, nontuberculous mycobacteria (NTMB), Blastomyces, or Aspergillus or current active Candidiasis (local or systemic).

### Has been changed to:

12. Subjects with known history of or current clinically active infection with Histoplasma, Coccidioides, Paracoccidioides, Pneumocystis, nontuberculous mycobacteria (NTMB), COPT application Blastomyces, or Aspergillus or current active Candidiasis (local or systemic).

### Change #16

### Section 6.3 Withdrawal criterion 8

### **Original text:**

8. Subject develops laboratory abnormalities (with or without clinical symptoms) of ALT or AST as defined in Section 6.3.1; neutropenia <0.5x10<sup>9</sup>/mL; lymphopenia <0.5x10<sup>9</sup>/mL. Any laboratory value or change judged to be clinically significant by the Investigator, and/or any lab values meeting the Rheumatology Common Toxicity Criteria (RCTC) Grade 4 criteria (with the exception of neutrophils which will be permitted with the above withdrawal criterion [neutropenia <0.5x10\mathcal{fmL}]; Table 19-2 and Table 19-3) must be discussed with the medical monitor before the subject is dosed again. (Refer to Section 6.3.1 for withdrawal criteria in relation to potential drug-induced liver injury [PDILI].)

# Has been changed to

8. Subject develops laboratory abnormalities (with or without clinical symptoms) of ALT or AST as defined in Section 6.3.1; neutropenia <0.5x10<sup>9</sup>/mL; lymphopenia <0.5x10<sup>9</sup>/mL. Any laboratory value or change judged to be clinically significant by the Investigator should prompt consideration of whether the subject should continue on IMP. For clarification, laboratory values that are markedly abnormal as per Table 19-2 and Table 19–3 will be flagged to the Investigator and to the medical monitor but do not trigger mandatory withdrawal unless listed above and/or any lab values meeting the Rheumatology Common Toxicity Criteria (RCTC) Grade 4 criteria (with the exception of neutrophils, which will be permitted with the above withdraw criterion [neutropenia < 0.5x109/mL]; Table 19 2 and Table 19 3) must be discussed with the medical monitor before the subject is dosed again (Refer to Section 6.3.1 for withdrawal criteria in relation to potential drug induced liver injury [PDILI].)

### Change #17

### **Section 7.3 Packaging**

win be packaged and labeled according to Good Manufacturing ractice (GMP) guidelines and applicable laws or regulations. They will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual. rejone of Vi

### Change #18

# Section 7.8.2 Prohibited concomitant treatments (medications and therapies), Table 7-1 Original text:

| Drug class | Dose | Exclusion criteria |
|---|---|---|
| Analgesics, including opioid analgesics (acetaminophen/paracetamol, etc) | Any dose | Any ad hoc use in the 24 hours prior to any study visit. Stable doses of analgesics permitted. |
| NSAIDs/COX-2 inhibitors | Any dose regimen | Any change in dose/dose regimen in the 14 days prior to the Baseline Visit |
| Oral corticosteroids | Any dose regimen | Any change in dose/dose regimen in the 28 days prior to the Baseline Visit |
| Intramuscular (im)/intravenous (iv)/<br>intra-articular (ia) corticosteroids/bursal<br>corticosteroids | Any dose | Use in the 28 days prior to the Baseline Visit. |
| Intra-articular hyaluronic acid | Any dose | Any use in the 6 months prior to the Baseline Visit. |
| DMARDs: -azathioprine -cyclosporine, -cyclophosphamide, -mycophenolic acid, -mycophenylate mofetil -any other small molecule DMARDs (eg tofacitinib, apremilast) | Any dose | Use within 12 weeks prior to the Baseline Visit. |
| MTX | Any dose regimen | Use within 12 weeks prior to the Baseline Visit unless Inclusion Criterion #10 is met |
| SSZ | Any dose | Use within 12 weeks prior to the Baseline Visit unless Inclusion Criterion #11 is met |
| HCQ | Any dose | Use within 12 weeks prior to the Baseline Visit unless Inclusion Criterion #11 is met |

| Drug class | Dose | Exclusion criteria |
|---|---|---|
| DMARDs:<br>-leflunomide | Any dose | Use in the 6 months prior to the Baseline Visit unless a cholestyramine washout has been performed; in which case, use up to 28 days prior to the Baseline Visit is acceptable. |
| TNF inhibitors -infliximab (IFX) -adalimumab (ADA) -etanercept (ETN) -golimumab (GOL) -certolizumab pegol (CZP) | Any dose | For IFX, ADA, GOL, and CZP, any use within the 3 months prior to the Baseline Visit For ETN, use within the 28 days prior to the Baseline Visit. This applies to biosimilar versions of any TNF inhibitors. |

# Has been changed to:

| Drug class | Dose | Exclusion criteria |
|---|---|---|
| Analgesics, including opioid analgesics (acetaminophen/paracetamol, etc) | Any dose | Any ad hoc use in the 24 hours prior to any study visit. |
| | .c.D. 18tile | Stable doses of analgesics permitted. |
| NSAIDs/COX-2 inhibitors | Any dose regimen | Any change in dose/dose regimen in the 14 days prior to the Baseline Visit |
| Oral corticosteroids | Any dose regimen | Any change in dose/dose regimen in the 28 14 days prior to the Baseline Visit |
| Intramuscular (im)/intravenous (iv)/<br>intra-articular (ia) corticosteroids/bursal<br>corticosteroids | Any dose | Use in the 28 days prior to the Baseline Visit. |
| Intra-articular hyaluronic acid | Any dose | Any use in the 6 months prior to the Baseline Visit. |
| DMARDs: -azathioprine -cyclosporine, -cyclophosphamide, -mycophenolic acid, -mycophenylate mofetil -any other small molecule DMARDs (eg tofacitinib, apremilast) | Any dose | Use within 12 weeks prior to the Baseline Visit. |
| MTX | Any dose regimen | Use within 12 weeks prior to the Baseline Visit unless Inclusion Criterion #10 is met |
| SSZ | Any dose | Use within 12 weeks prior to the Baseline Visit unless Inclusion Criterion #11 is met |

| Drug class | Dose | Exclusion criteria |
|---|---|---|
| HCQ | Any dose | Use within 12 weeks prior to the Baseline<br>Visit unless Inclusion Criterion #11 is met |
| DMARDs:<br>-leflunomide | Any dose | Use in the 6 months prior to the Baseline Visit unless a cholestyramine washout has been performed; in which case, use up to 28 days prior to the Baseline Visit is acceptable. |
| TNF inhibitors -infliximab (IFX) -adalimumab (ADA) -etanercept (ETN) -golimumab (GOL) -certolizumab pegol (CZP) | Any dose | For IFX, ADA, GOL, and CZP, any use within the 3 months 12 weeks prior to the Baseline Visit For ETN, use within the 28 days prior to the Baseline Visit. This applies to biosimilar versions of any TNF inhibitors. |

The following paragraphs have been added:

Subjects who initially fail to meet selected altricular documented completion of LTPT could not be complete.

Medical \*\*\* Subjects who initially fail to meet selected eligibility criteria (including but not limited to documented completion of LTBI prophylactic therapy) or for whom eligibility assessments could not be completed as planned may be rescreened once after discussion with the **Medical Monitor.** 

The MRI (done at selected sites) can be performed prior to the Baseline (Day 1, first dose of IMP, Visit 2) if eligibility is confirmed based on screening assessments, and before the first dose of IMP.

### Change #20

### Section 8.2 Baseline (Day 1, first dose of IMP) (Visit 2)

# Original text:

Obtain MRI of spine and the SI joint if the subject is participating in the MRI substudy.

# Has been changed to:

Obtain MRI of spine and the SI joint if the subject is participating in the MRI substudy. **The** Baseline MRI should be performed after confirmation of eligibility based on screening assessments for the study and before the first bimekizumab injection.

### Change #21

### Section 8.3.5 Week 12 (+/-3 days) (Visit 7)

### **Original text:**

The following procedures of assessments will be completed prior to administration of IMP:

. . .

 Obtain MRI of spine and the sacroiliac joint if the subject is participating in the MRI substudy.

. . .

The following procedures of assessments will be completed following administration of IMP:

• Collect pulse and BP once after dosing (any time).

### Has been changed to:

The following procedures of assessments will be completed prior to administration of IMP:

. . .

Obtain MRI of spine and the sacroiliac joint if the subject is participating in the MRI substudy and is MRI-positive at Baseline. Magnetic resonance imaging at Week 12 should be performed as close to the Week 12 Visit as possible.

. . .

The following procedures of assessments will be completed following administration of IMP:

• Collect pulse and BP once after dosing (any time pulse and BP to be collected 30 minutes and 1 hour after dosing).

# Change #22

# Section 8.4.9 Week 48 (+/-4 days) (Visit 16)

# Original text:

• Obtain MRI of spine and the sacroiliac joint if the subject is participating in the MRI substudy.

### Has been changed to:

Obtain MRI of spine and the sacroiliac joint if the subject is participating in the MRI Valiations the reof. substudy and is MRI-positive at Baseline. Magnetic resonance imaging at Week 48 should be performed as close to the Week 48 Visit as possible.

### Change #23

# Section 9.1 ASAS20, 40, ASAS 5/6 response, and ASAS partial remission **Original text:**

The ASAS 5/6 response is defined as at least 20% improvement in 5 of 6 domains, including spinal mobility (lateral spinal flexion) and CRP as more objective measures (Brandt et al., 2004).

### Has been changed to:

The ASAS 5/6 response is defined as at least 20% improvement in 5 of 6 domains, including ctive COPT application spinal mobility (lateral spinal flexion) and hs-CRP as more objective measures (Brandt et al, 2004).

### Change #24

### **Section 9.7 Spinal mobility**

### **Original text:**

Lateral spinal flexion is measured with the subject's heels and back resting against the wall with no flexion in the knees and no bending forward. The subject lets the arm hang normally with the palm of the hand resting against the outer thigh and the fingers extended. A mark is drawn on the thigh at the tip of the middle finger. The subject is then asked to bend sideways without bending the knees or lifting the heels, while sliding the hand down the thigh. At the point of furthest reach, another mark is drawn at the tip of the middle finger. The distance between the first and second mark is measured to the nearest 0.1cm. An alternative method is to measure the distances to the 2 lines from the floor and record the difference. The better of 2 tries is recorded for left and right separately. The mean of the left and right is reported for lateral spine flexion (in cm to the nearest 0.1cm) (Sieper et al, 2009) (Appendix Section 19.7).

Has been deleted.

Change #25

Original text:

The BASFI is described in Section 9.4 above.

Has been deleted.

### Change #26

### Section 9.12 Extra-articular manifestations

### Original sections and text:

Information regarding uveitis, enthesitis, inflammatory bowel disease, and psoriasis disease activity will be captured. Enthesitis is assessed via MASES.

### **Section 9.13 MASES**

The MASES is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) (Heuft-Dorenbosch et al, 2003) each scored as 0 or 1 and then summed for a possible score of 0 to 13.

### Have been merged and changed to:

### Section 9.12 Extra artucilar manifestations

Information regarding uveitis, enthesitis, inflammatory bowel disease, and psoriasis disease activity will be captured. Enthesitis is assessed via MASES.

### **Section 9.10 MASES**

Enthesitis is assessed with MASES. The MASES is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) (Heuft-Dorenbosch et al, 2003) each scored as 0 or 1 and then summed for a possible score of 0 to 13.

### Change #27

**Section 9.12 PhGADA** 

### Original text:

### 9.14 PhGADA

The Investigator will assess the overall status of the subject with respect to their AS signs and symptoms and functional capacity (considering both joint and skin components) using an NRS in which 0=very good, asymptomatic and no limitations of normal activities and 100=very poor, very severe symptoms which are intolerable and inability to carry out normal activities.

### Has been changed to:

### 9.11 PhGADA

Section 9.15 Total and nocturnal spinal pain
Assessment of total and nocturnal spinal pain was described above in Section 9.15 MRI Assessment (SP\*\*
riginal text:

19 MP\*\*

### 9.19 MRI Assessment (SPARCC and ASspiMRI)

An MRI of the spine and sacroiliac joints will be performed in a substudy with approximately 10 subjects per treatment arm at Screening Week 12, and Week 48. Additional details for standardized performance and processing of MRIs will be provided in an MRI manual. The MRIs will be read centrally by readers who are blinded to treatment assignment and chronological order of the MRIs according to a charter for independent imaging assessment.

# Has been changed to:

### 9.15 MRI Assessment (SPARCC and ASspiMRI)

An MRI of the spine and sacroiliac joints will be performed in a substudy with approximately 20 subjects per treatment arm at Screening Baseline. A central reader will assess Baseline MRIs to identify MRI-positive subjects as per the ASAS-Outcome Measures in Rheumatology Clinical Trials (OMERACT) criteria. An MRI at Week 12 and Week 48 will be performed for those subjects who were MRI-positive at Baseline. The Baseline MRI should be performed after confirmation of eligibility based on screening assessments for the study and before the first bimekizumab injection. Magnetic resonance imaging at Week 12 and Week 48 should be performed as close to the Week 12/Week 48 Visit as possible. Additional details for standardized performance and processing of MRIs will be provided in an MRI manual. The MRIs will be read centrally by readers who are blinded to treatment assignment and chronological order of the MRIs according to a charter for independent imaging assessment.

### Change #30

### Section 12.1.5 Description of adverse events

### Original text:

When recording an AE, the Investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words on his/her own records (eg, diary card) and the corresponding medical terminology should be clarified in the source documentation.

Details for completion of the Adverse Event eCRF (including judgment of relationship to IMP) are described in the eCRF Completion Guidelines.

### Has been changed to:

When recording an AE, the Investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words on his/her own records (eg, diary card) and the corresponding medical terminology should be clarified in the source documentation.

When recording the intensity of an AE in the eCRF (ie, mild, moderate, or severe), the Investigator should use the following criteria:

- Mild: the subject is aware of the sign or symptom (syndrome), but it does not interfere with his/her usual activities and/or is of no clinical consequence
- Moderate: the AE interferes with the usual activities of the subject or it is of some clinical consequence
- Severe: the subject is unable to work normally or to carry out his/her usual activities, or the AE is of definite clinical consequency

Details for completion of the Adverse Event eCRF (including judgment of intensity and relationship to IMP) are described in the eCRF Completion Guidelines.

AS0008

### Change #31

### Section 12.5 Laboratory measurements, Table 12-2

### Original text:

| Hematology | Chemistry | Urinalysis |
|---|---|---|
| Basophils | Calcium | Albumin |
| Eosinophils | Chloride | Bacteria |
| Lymphocytes | Magnesium | Crystals |
| Atypical lymphocytes | Potassium | Glucose |
| Monocytes | Sodium | pH |
| Neutrophils | Glucose | RBC |
| Hematocrit | BUN | WBC SO' |
| Hemoglobin | Creatinine | Urine dipstick for pregnancy testing <sup>a</sup> |
| MCH | AST | alle |
| MCHC | ALT | dio |
| MCV | ALP | Silco |
| Platelet count | GGT R | 54 |
| RBC count | Total bilirubin | |
| WBC count | LDH | |
| | Total cholesterol | |
| | Serum pregnancy testing <sup>a</sup> | |
| | CRP <sup>b</sup> | |
| | hs-CRP <sup>b</sup> | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CRP=C-reactive protein; GGT=gamma glutamyltransferase; hs-CRP=high sensitivity C-reactive protein; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; SFU=Safety Follow-up; WBC=white blood

# Has been changed to:

| Hematology | Chemistry | Urinalysis |
|---|---|---|
| Basophils | Calcium | Albumin |
| Eosinophils | Chloride | Bacteria |
| Lymphocytes | Magnesium | Crystals |
| Atypical lymphocytes | Potassium | Glucose |
| Monocytes | Sodium | рН |
| Neutrophils | Glucose | RBC |
| Hematocrit | BUN | WBC |
| Hemoglobin | Creatinine | Urine dipstick for pregnancy testing <sup>a</sup> |

| Hematology | Chemistry | Urinalysis |
|----------------|--------------------------------------|------------|
| MCH | AST | |
| MCHC | ALT | |
| MCV | ALP | |
| Platelet count | GGT | |
| RBC count | Total bilirubin | igilo |
| WBC count | LDH | Valle |
| | Uric acid | e o's |
| | Total cholesterol | ions |
| | Serum pregnancy testing <sup>a</sup> | |
| | CRPb | et |
| | hs-CRP <sup>b</sup> | 303 |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CRP=C-reactive protein; GGT=gamma glutamyltransferase; hs-CRP=high sensitivity C-reactive protein; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; SFU=Safety Follow-up; WBC=white blood cell

### Change #32

### Section 12.6.1 Vital signs

### **Original text:**

The Investigator or designee should measure all vital signs (systolic and diastolic BP, temperature [oral, axillary, or otic], pulse rate) after the subject has been sitting for at least 5 minutes, and the subject should remain seated during the measurements. Body temperature should be obtained prior to dosing with IMP at study visits when IMP is administered. At Baseline/Day 1 and Week 1, collect pulse and BP prior to drug administration and then at 30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing (any time).

# Has been changed to:

The Investigator or designee should measure all vital signs (systolic and diastolic BP, temperature [oral, axillary, or otic], pulse rate) after the subject has been sitting for at least 5 minutes, and the subject should remain seated during the measurements. Body temperature should be obtained prior to dosing with IMP at study visits when IMP is administered. At Baseline/Day 1 and Week 12, collect pulse and BP prior to drug administration and then at 30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing (any time).

### Change #33

### Section 12.6.5 Tuberculosis and TB risk factor assessment and management, **Exclusion criteria at Screening**

Subjects with known TB infection, at high risk of acquiring TB infection, with LTBI\*, or current or history of NTMB infection.

\*Subjects with LTBI may enter the study only after the appropriate prophylactic 41.

### Has been changed to:

**Exclusion Criteria at Screening** 

Subjects with known TB infection, at high risk of acquiring TB infection, with LTBI\*, or current or history of NTMB infection.

\*Subjects with LTBI may enter the study only after they have completed at least 8 weeks of appropriate prophylactic therapy and thereafter, will continue and complete the entire regimen. Following consultation with the Medical Monitor, subjects may be rescreened after completion at least 8 weeks of LTBI prophylactic therapy.

### Change #34

# Section 15.1 Definition of analysis sets

### **Original text:**

The PK-PPS will consist of all randomized subjects who took at least 1 dose of IMP and provide at least 1 quantifiable plasma concentration postdose.

The PD-PPS will consist of all randomized subjects who took at least 1 dose of IMP and provide at least 1 PD measurement postdose that is without important protocol deviation affecting that time point.

The Dose-Blind Set (DBS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period.

The Escape Subject Set (ESS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period and who have not achieved an at least 10% reduction from Baseline in PGADA and total and nocturnal spinal pain at either Week 16, Week 24, or Week 36.

The Dose-Blind Responder Set (DBRS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period and who have achieved an at least 10% reduction from Baseline in PGADA and total and nocturnal spinal pain at Week 16, Week 24, and Week 36. Subjects who are eligible for the ESS, but do not receive rescue medication, remain in the DBRS.

### Has been changed to:

The Pharmacokinetic Per Protocol Set (PK-PPS) is a subset of the FAS, consisting of those subjects who had no important protocol deviations affecting the pharmacokinetic

The Dose-Blind Set (DBS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period including the dose at Week 12.

The Escape Subject Set (ESS) consists of all subjects starting the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the dose at the second at least 1 dose of the IMP during the Dose-Blind Period including the Dose-Blind Period including the Dose-Blind Period including the Dose-B

at least 10% reduction from Baseline in PGADA and total and nocturnal spinal pain at either Week 16, Week 24, or Week 36.

The Dose-Blind Responder Set (DBRS) consists of all subjects starting the Dose-Blind Period and who received at least 1 dose of the IMP during the Dose-Blind Period and who have achieved an at least 10% reduction from Baseline in PGADA and total and nocturnal spinal pain at Week 16, Week 24, and Week 36. Subjects who are eligible for the ESS, but do not receive rescue medication, remain in the DBRS.

### Change #35

Section 15.4 Subgroup analyses

### **Original text:**

• BASDAI ( $\geq 4$  to  $\leq 7$  [moderate disease];  $\geq 7$  to  $\leq 10$  [severe disease])

# Has been changed to:

BASDAI (<4 [mild disease];  $\ge 4$  to  $\le 7$  [moderate disease]; >7 to  $\le 10$  [severe disease])

### Change #36

Section 15.5.1 Safety analyses

### The following paragraph has been added:

Treatment-emergent AEs will be defined as events that have a start date on or following the first administration of study treatment through the final administration of study treatment +140 days (covering the 20 week SFU Period).

### Change #37

### Section 15.5.2 Other analyses

analysis plan and reported in a separate data analysis plan and reported in a separate document. Plasma concentration-time data of bimekizumab and ASAS40 responder rates will be used as the PK and PD response. If data merits, a further PK/PD analysis on other PD variables may be performed.

Has been changed to:

Pharmacokinetic and PD analyses including the calculation of population estimates for total body clearance (CL/F) and volume of distribution (V/F) will be detailed in a separate of the bimeking of the population analysis plan and reported in a separate of the bimeking of the population in the population of population estimates for total bimeking of the population estimates for total bimeking of the population of population estimates for total bimeking of the population

bimekizumab and ASAS40 responder rates will be used as the PK and PD response. If data merits, a further PK/PD analysis on other PD variables may be performed.

### Change #38

### **Table 19-1 Table footnote**

### **Original text:**

Note: A second grading of "probably ankylosing spondylitis" is part of the modified NY criteria, but it is not applicable for this study. It is included here for completeness. The grading will be probable ankylosing spondylitis if 3 clinical criteria are present and the radiologic criterion is present without any signs or symptoms satisfying the clinical criteria (other causes of sacroiliitis should be considered).

# Has been changed to:

AS=ankylosing spondylitis; mNY=modified New York Criteria

Note: A second grading of "probable ankylosing spondylitis" is part of the modified NY criteria, but it is not applicable for this study. It is included here for completeness. The grading will be probable ankylosing spondylitis if 3 clinical criteria are present and the radiologic criterion is present without any signs or symptoms satisfying the clinical criteria (other causes of sacroiliitis should be considered).

### 19.4 Protocol Amendment 2

### Rationale for the amendment

The purpose of this substantial protocol amendment is the following:

- To update the study contact details for the sponsor study physician and clinical trial biostatistician
- To revise the withdrawal criteria section to provide instructions for the management of subjects with newly diagnosed IBD or with IBD flares during the study.
- Amend the time window between doses during the Double-Blind Period of the study.
- To revise and clarify the SAE criteria for pregnancy for consistency.
- Amend the table for identification/exclusion of alternative etiology to include ALT and AST.

### Modifications and changes

### Global changes

No global changes have been made. Specific changes are listed below.

### **Specific changes**

### Change #1

### LIST OF ABBREVIATIONS

The following abbreviation and definition was added:

**RCTC** 

Rheumatology Common Toxicity Criteria

### Change #2

### STUDY CONTACT INFORMATION

### **Original text:**

### Sponsor Study Physician

| Name: S | , MD |
|----------|---------------------------|
| Address: | UCB BIOSCIENCES Inc. |
| arot | 8010 Arco Corporate Drive |
| | Raleigh, NC 27617 |
| | UNITED STATES |
| Phone: | |

### Has been changed to:

| Name: | , MD, MSc, PhD |
|----------|-----------------------------------------|
| Address: | UCB Pharma Ltd. UCB BIOSCIENCES Inc. |
| | 208 Bath Road 8010 Arco Corporate Drive |
| | Slough, SL1 3WE Raleigh, NC 27617 |
| | UNITED KINGDOM UNITED STATES |
| Phone: | |

Change #3

STUDY CONTACT INFORMATION

**Original text:** 

### **Clinical Trial Biostatistician**

| Name: | Dr. , Senior Biostatistician |
|---|---|
| Address: | UCB BIOSCIENCES GmbH Alfred-Nobel-Str.10 40789 Monheim am Rhein GERMANY |
| Phone: | |

# Has been changed to:

# Clinical Trial Biostatistician

| Name: | , MSDr. , Senior |
|---|---|
| Address: | UCB BIOSCIENCES Inc.GmbH |
| 8010 Arco Corporate Drive Alfred Nobel Str.10 | |
| 11500 | Raleigh, NC 2761740789 Monheim am Rhein |
| , pe | UNITED STATESGERMANY |
| Phone: | |

# Change #4 Section

### **Section 6.3 Withdrawal Criteria**

The following was added to the withdrawal criteria:

11. Subjects with newly diagnosed IBD or with IBD flares during the study must:

- Be referred, as appropriate, to a health care professional treating IBD, such as a gastroenterologist
- Discontinue IMP and be followed-up until resolution of active IBD symptoms

extensions or variations thereof. If IBD flares increase in severity or frequency during the study, the Investigator should use clinical judgment in deciding whether the subject should continue in the study and contact the Medical Monitor and UCB study physician to confirm the subject's suitability for continued participation in the study.

### Change #5

### Section 7.2 Treatments to be administered, paragraph 2

### Original text:

The IMP (bimekizumab and placebo) will be administered at the times indicated in Table 5–1. The minimum time between doses during the Double-Blind Period should be no less than 26 days and no more than 30 days and during the Dose-Blind Period should be no less than 24 days and no more than 32 days.

### Has been changed to:

The IMP (bimekizumab and placebo) will be administered at the times indicated in Table 5–1. The minimum time between doses during the Double-Blind Period should be no less than 256 days and no more than 310 days and during the Dose-Blind Period should be no less than 24 days and no more than 32 days.

### Change #6

### Section 7.3 Packaging

### **Original text:**

Bimekizumab and placebo will be packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. They will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

# Has been changed to:

Bimekizumab and placebo will be **manufactured**, packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. They will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

### Change #7

### Section 12.1.8 Pregnancy, paragraph 5

mue normonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report Form.

Has been changed to:

A pregnancy becomes an SAE in the following circumstances: miscarriage, elective abortion when medically indicated (e.g. when pregnancy is endangering life or health of woman or when fetus will be born with severe abnormalities), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report form.

### Change #8

### Testing: identification/exclusion of alternative etiology, Table **Section 12.5.1.4** 12-4

### Original table:

| Original table. | |
|---|---|
| Virology- | Hepatitis A IgM antibody |
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM AND |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| rmmunology | Anti-smooth muscle antibody (qualitative and quantitative) |
| A Co | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |

| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
|---|---|
| Additional | ditional Prothrombin time/INR <sup>b</sup> |
| | Serum pregnancy test |
| | PK sample |

ALT=alanine aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

<sup>a</sup> For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

b Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

### Has been changed to:

| | 1 dic |
|---|---|
| Virology- | Hepatitis A IgM antibody |
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | Hepatitis A IgM antibody HBsAg Hepatitis E IgM antibody HBcAb-IgM Hapatitis C RNA |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| nent | ALT, AST |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |

| Additional | Prothrombin time/INR <sup>b</sup> |
|------------|-----------------------------------|
| | Serum pregnancy test |
| | PK sample |

ALT=alanine aminotransferase; AST=aspartate aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

<sup>a</sup> For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

b Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

### Change #9

Markedly abnormal laboratory values, Tables 17-10 Definitions of markedly Section 17.1 abnormal hematology values) and 17-2 (Definitions of markedly abnormal biochemistry values)

Amended units in both table headers:

| | Markedly Abnormal Definition | |
|--------------------------|------------------------------|------|
| Parameter (SI units) | Low | High |
| Has been changed to: | akDA auti | |
| | Markedly Abnormal Definition | |
| Parameter (SIRCTC units) | Low | High |

# Change #10

Markedly abnormal laboratory values, Table 17-1 (Definitions of markedly Section 17.1 abnormal hematology values), abbreviations in table footer:

LLN=lower limit of normal; N/A = Not Applicable; SI = standard international

# Has been changed to:

LLN=lower limit of normal; N/A = Not Applicable; SI = standard international RCTC= Rheumatology Common Toxicity Criteria

# Change #11

Markedly abnormal laboratory values, Table 17-2 (Definitions of markedly Section 17.1 abnormal biochemistry values), abbreviations in table footer:

The document control be used to support any materials altered the support of the


### 20 DECLARATION AND SIGNATURE OF INVESTIGATOR

I confirm that I have carefully read and understood this protocol and agree to conduct this clinical study as outlined in this protocol, according to current Good Clinical Practice and local laws and requirements.

I will ensure that all subinvestigators and other staff members read and understand all aspects of this protocol.

I have received and read all study-related information provided to me.

The objectives and content of this protocol as well as the results deriving from it will be treated confidentially, and will not be made available to third parties without prior authorization by UCB.

All rights of publication of the results reside with UCB, unless other agreements were made in a separate contract.

| Investigator: | and of the |
|---|---|
| | - J -dication |
| Printed name | Date/Signature |
| se used to support any me | |
| Printed name Printed name Printed name This document common to be used to support any marketing the support and the s | |

The document control be used to support any materials about the control of the co

